## Phase III, Single-arm, Open-label, International, Multicentre Study to Evaluate the Efficacy and Safety of Lomitapide in Paediatric Patients with Homozygous Familial Hypercholesterolaemia (HoFH) on Stable Lipidlowering Therapy

Amryt Pharma Study No: APH-19 SQN Clinical Study No: OCH19003

## **Table, Figure and Listing Shells**

Version: Final 5.0 Date: 28 June 2024



### **Approved By Amryt Pharma**



## Associate Director Clinical Operations



Zsuzsanna Tamas Senior Director / Project Physician Leader Global Rare Diseases

## TABLE/FIGURE/LISTING CONTENTS

| Table 14.1.1.1 Subject Disposition | |
|---|---|
| Table 14.1.1.2 Subject Study Visits | . 13 |
| Table 14.1.2.1 Demography | . 14 |
| Table 14.1.2.2 Baseline Lipids | . 18 |
| Table 14.1.2.3 Diagnosis of HoFH | . 22 |
| Table 14.1.3.1 Medical History | . 24 |
| Table 14.1.3.2 Cardiovascular History | . 25 |
| Table 14.1.3.3 Cardiovascular Disease History at Screening | . 26 |
| Table 14.1.4.1 Prior and 'Run-in Medications' Medications | |
| Table 14.1.4.2 Concomitant Medications | |
| Table 14.1.4.3 Lipid-Lowering-Therapy Medications | |
| Table 14.1.4.5 Procedures | |
| Table 14.1.4.6 Days from most recent apheresis to the corresponding LDL-C primary efficac | СУ |
| assessment | . 32 |
| Table 14.1.5.1 Study Drug Exposure and Dosing | . 34 |
| Table 14.1.5.2 Summary of Compliance to IMP | . 43 |
| Table 14.1.5.3 Time to Dose Reduction and Interruption | . 44 |
| Table 14.1.5.4 Distribution of Achieved Doses | . 45 |
| Table 14.2.1.1 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | . 46 |
| Table 14.2.1.2 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Supplementary analysis - per protocol set) | . 51 |
| Table 14.2.1.3 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Supplementary analysis - completer analysis set) | . 52 |
| Table 14.2.1.4 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 1 - Age groups) | . 53 |
| Table 14.2.1.5 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 2 - Documented cardiovascular disease history) | . 57 |
| Table 14.2.1.6 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve | |
| disease and/or coronary atherosclerosis)) | . 61 |
| Table 14.2.1.7 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 4 - Concomitant LLT medications/procedures) | . 66 |
| Table 14.2.1.8 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 5 - Dose reductions / dose interruptions) | . 70 |
| Table 14.2.1.9 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group) | . 74 |
| Table 14.2.1.10 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks | |
| | . 78 |
| Table 14.2.1.11 Lipid parameter: LDL-C (mg/dL) Responder Analysis (Supplementary | |
| analysis) | |
| Table 14.2.2.1 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Secondary analysis) | . 83 |
| Table 14.2.2.2 Lipid parameter: Non-HDL-C (mg/dL)and change from baseline at 24 weeks | |
| (Supplementary analysis - per protocol set) | |
| Table 14.2.2.3 Lipid parameter: Non-HDL-C value (mg/dL) change from baseline at 24 week | |
| (Supplementary analysis - completer analysis set) | |
| Table 14.2.2.4 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 1 - Age groups) | . გნ |
| Table 14.2.2.5 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 2 - Documented cardiovascular disease history) | |
| Table 14.2.2.6 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks | ; |
| (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve | 0.0 |
| disease and/or coronary atherosclerosis)) | . გგ |
| Table 14.2.2.7 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 4 - Concomitant LLT medications/procedures) | . გ |

| Table 14.2.2.8 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks | |
|---|---|
| | . 90 |
| Table 14.2.2.9 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group) | |
| Table 14.2.2.10 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 week | |
| | . 92 |
| Table 14.2.2.11 Lipid parameter: Non-HDL-C (mg/dL) Responder Analysis (Supplementary | 00 |
| analysis)<br>Table 14.2.3.1 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks | 93 |
| | 04 |
| (Secondary analysis)<br>Table 14.2.3.2 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks | 94 |
| (Supplementary analysis - per protocol set) | 05 |
| Table 14.2.3.3 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks | . 90 |
| (Supplementary analysis - completer analysis set) | 96 |
| Table 14.2.3.4 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgrou | |
| analysis 1 - Age groups) | |
| Table 14.2.3.5 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgrou | |
| analysis 2 - Documented cardiovascular disease history) | |
| Table 14.2.3.6 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgrou | |
| analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and | |
| coronary atherosclerosis)) | |
| Table 14.2.3.7 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subground | up |
| analysis 4 - Concomitant LLT medications/procedures) | 100 |
| Table 14.2.3.8 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subground) | up |
| analysis 5 - Dose reductions / dose interruptions) 1 | |
| Table 14.2.3.9 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subground | |
| analysis 6 - Reached MTD for age group/ did not reach MTD for age group)1 | 102 |
| Table 14.2.3.10 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 7 - Sex)1 | 103 |
| Table 14.2.3.11 Lipid parameter: TC (mg/dL) Responder Analysis (Supplementary | |
| | 104 |
| Table 14.2.4.1 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | 405 |
| | 105 |
| Table 14.2.4.2 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | 106 |
| (Supplementary analysis - per protocol set) | 100 |
| Table 14.2.4.3 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | 107 |
| (Supplementary analysis - completer analysis set) | 107 |
| (Subgroup analysis 1 - Age groups) | 108 |
| Table 14.2.4.5 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | 100 |
| (Subgroup analysis 2 - Documented cardiovascular disease history) | 100 |
| Table 14.2.4.6 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | 100 |
| (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve | |
| disease and/or coronary atherosclerosis)) | 110 |
| Table 14.2.4.7 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 4 - Concomitant LLT medications/procedures) | 111 |
| Table 14.2.4.8 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 5 - Dose reductions / dose interruptions) | 112 |
| Table 14.2.4.9 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group) 1 | 113 |
| Table 14.2.4.10 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 7 - Sex)1 | 114 |
| Table 14.2.4.11 Lipid parameter: VLDL-C (mg/dL) Responder Analysis (Supplementary | |
| analysis)1 | 115 |
| Table 14.2.5.1 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | |
| (Secondary analysis)1 | 116 |
| Table 14.2.5.2 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | |
| (Supplementary analysis - per protocol set) | 117 |
| Table 14.2.5.3 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | |
| (Supplementary analysis - completer analysis set)1 | 118 |

| Table 14.2.5.4 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | |
|---|---|
| (Subgroup analysis 1 - Age groups) | 119 |
| Table 14.2.5.5 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 2 - Documented cardiovascular disease history) | 120 |
| Table 14.2.5.6 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve | |
| disease and/or coronary atherosclerosis)) | 121 |
| Table 14.2.5.7 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 4 - Concomitant LLT medications/procedures) | 122 |
| Table 14.2.5.8 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 5 - Dose reductions / dose interruptions) | 123 |
| Table 14.2.5.9 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | 120 |
| (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group) | 12/ |
| Table 14.2.5.10 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks | 127 |
| (Subgroup analysis 7 - Sex) | 125 |
| Table 14.2.5.11 Lipid parameter: Apo B (mg/dL) Responder Analysis (Supplementary | 120 |
| | 400 |
| analysis) | 120 |
| Table 14.2.6.1 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks | 407 |
| (Secondary analysis) | 127 |
| Table 14.2.6.2 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks | |
| (Supplementary analysis - per protocol set) | 128 |
| Table 14.2.6.3 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks | |
| (Supplementary analysis - completer analysis set) | |
| Table 14.2.6.4 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgro | oup |
| analysis 1 - Age groups) | 130 |
| Table 14.2.6.5 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgro | oup |
| analysis 2 - Documented cardiovascular disease history) | 131 |
| Table 14.2.6.6 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgro | |
| analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and | d/or |
| coronary atherosclerosis)) | |
| Table 14.2.6.7 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgro | |
| analysis 4 - Concomitant LLT medications/procedures) | |
| Table 14.2.6.8 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgro | |
| analysis 5 - Dose reductions / dose interruptions) | |
| Table 14.2.6.9 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgro | |
| analysis 6 - Reached MTD for age group/ did not reach MTD for age group) | |
| Table 14.2.6.10 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks | 100 |
| (Subgroup analysis 7 - Sex) | 136 |
| Table 14.2.6.11 Lipid parameter: TG (mg/dL) Responder Analysis (Supplementary | 130 |
| | 127 |
| analysis) | 137 |
| Table 14.2.7.1 Lipid parameter: Lp(a) and change from baseline at 24 weeks (Secondary | 420 |
| analysis) | 130 |
| Table 14.2.7.2 Lipid parameter: LP(a) and change from baseline at 24 weeks (Supplemental Parameters and Paramet | |
| analysis - per protocol set) | |
| Table 14.2.7.3 Lipid parameter: LP(a) and change from baseline at 24 weeks (Supplemental | |
| analysis - completer analysis set) | 140 |
| Table 14.2.7.4 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 1 - Age groups) | 141 |
| Table 14.2.7.5 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 2 - Documented cardiovascular disease history) | 142 |
| Table 14.2.7.6 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve | |
| disease and/or coronary atherosclerosis)) | |
| Table 14.2.7.7 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 4 - Concomitant LLT medications/procedures) | 144 |
| Table 14.2.7.8 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 5 - Dose reductions / dose interruptions) | 145 |
| Table 14.2.7.9 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks | |
| (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group) | 146 |
| Table 14.2.7.10 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks | 1-10 |
| | 117 |
| (Subgroup analysis 7 - Sex) | 14/ |

Date: 28JUN2024

Version: Final 5.0

| Table 14.2.7.11 Lipid parameter: LP(a) (mg/dL) Responder Analysis (Supplementary |
|---|
| analysis) |
| Table 14.2.8.1 Lipid parameter: LDL-C (mg/dL) and change from Baseline to EOT / Week 104 |
| by age group (Summary Measures) |
| Table 14.2.8.2 Lipid parameter: Non-HDL-C (mg/dL) and change from Baseline to EOT / Week |
| 104 by age group (Summary Measures) |
| Table 14.2.8.3 Lipid parameter: TC (mg/dL) and change from Baseline to EOT / Week 104 by |
| age group (Summary Measures) |
| Table 14.2.8.4 Lipid parameter: VLDL-C (mg/dL) and change from Baseline to EOT / Week |
| 104 by age group (Summary Measures) |
| Table 14.2.8.5 Lipid parameter: Apo B (g/L) and change from Baseline to EOT / Week 104 by |
| age group (Summary Measures) |
| Table 14.2.8.6 Lipid parameter: TG (mg/dL) and change from Baseline to EOT / Week 104 by |
| age group (Summary Measures) |
| Table 14.2.8.7 Lipid parameter: Lp(a) and change from Baseline to EOT / Week 104 by age |
| group (Summary Measures)157 |
| Table 14.2.8.8 Lipid parameter: TC/HDL-C ratio and change from Baseline to EOT / Week 104 |
| by age group (Summary Measures) |
| Table 14.2.0.1 Linid parameters LDL C (mar/dL) and sharps from Decaling to FOT (Week 104. |
| Table 14.2.9.1 Lipid parameter: LDL-C (mg/dL) and change from Baseline to EOT / Week 104 |
| (Mixed Model Repeated Measures analysis) |
| Table 14.2.9.2 Lipid parameter: Non-HDL-C (mg/dL) and change from Baseline to EOT / Week |
| 104 (Mixed Model Repeated Measures analysis) |
| Table 14.2.9.3 Lipid parameter: TC (mmol/L) and change from Baseline to EOT / Week 104 |
| (Mixed Model Repeated Measures analysis) |
| Table 14.2.9.4 Lipid parameter: VLDL-C (mg/dL) and change from Baseline to EOT / Week |
| 104 (Mixed Model Repeated Measures analysis) |
| Table 14.2.9.5 Lipid parameter: Apo B (g/L) and change from Baseline to EOT / Week 104 |
| (Mixed Model Repeated Measures analysis) |
| Table 14.2.9.6 Lipid parameter: TG (mg/dL) and change from Baseline to EOT / Week 104 |
| (Mixed Model Repeated Measures analysis) |
| Table 14.2.9.7 Lipid parameter: LP(a) and change from Baseline to EOT / Week 104 (Mixed |
| Model Repeated Measures analysis) |
| Table 14.2.9.8 Lipid parameter: TC/HDL-C ratio and change from Baseline to EOT / Week 104 |
| (Mixed Model Repeated Measures analysis) |
| Table 14.2.10.1 Treated with standard Lipid Lowering Therapy (LLT) (including Lipoprotein |
| Apheresis (LA) |
| Table 14.2.10.2 Reduction in dose of standard Lipid Lowering Therapy (LLT) / Reduced need |
| for Lipoprotein Apheresis (LA) compared to Week 24 (end of Efficacy Phase) |
| Table 14.2.10.3 Discontinue standard Lipid Lowering Therapy (LLT) / Discontinue need for |
| Lipoprotein Apheresis (LA) compared to Week 24 (end of Efficacy Phase) |
| Table 14.2.10.4 Increase dose of standard Lipid Lowering Therapy (LLT) / Increased need for |
| Lipoprotein Apheresis (LA) compared to Week 24 (end of Efficacy Phase) |
| Table 14.2.11.1 Recommended target of LDL-C of <135 mg/dL (i.e. 3.5 mmol/L) - EAS |
| recommendation |
| Table 14.2.11.2 Recommended target of LDL-C of <135 mg/dL (i.e. 3.5 mmol/L) by age group |
| and Lomitapide dose - EAS recommendation |
| Table 14.2.11.3 Recommended targets of LDL-C - Exploratory endpoints |
| Table 14.2.11.4 Recommended targets of LDL-C by age group and Lomitapide dose - |
| Exploratory endpoints |
| Table 14.2.12.1 Lipid parameter: HDL-C (mg/dL) and change from Baseline to EOT / Week |
| 104 by age group (Summary Measures) |
| Table 14.2.12.2 Lipid parameter: HDL-C (mg/dL) and change from Baseline to EOT / Week |
| 104 (Mixed Model Repeated Measures analysis) |
| Table 14.3.1.1 Summary of Treatment-Emergent Adverse Events |
| Table 14.3.1.2 Summary of Treatment-Emergent Adverse Events by MedDRA System Organ |
| Class and Preferred Term |
| Table 14.3.1.3 Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Class |
| and Preferred Term |
| Table 14.3.1.4 Summary of Treatment-Emergent Adverse Events by MedDRA Preferred |
| Term 182 |
| Table 14.3.1.5 Summary of Serious Adverse Events (SAEs) by MedDRA Preferred Term 183 |

Date: 28JUN2024 Version: Final 5.0 

| Table 14.3.1.6 Summary of Treatment-Emergent Adverse Events by MedDRA System Orga | ın |
|---|---|
| Class, Preferred Term and Severity<br>Table 14.3.1.7 Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Cla | 184 |
| Table 14.3.1.7 Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Cla | ıss, |
| Preferred Term and Severity | 185 |
| Table 14.3.1.8 Summary of Treatment-Emergent Adverse Events by MedDRA System Orga | |
| Class, Preferred Term and Relationship to Study Treatment | 186 |
| Table 14.3.1.9 Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Cla | ISS, |
| Preferred Term and Relationship to Study Treatment | 187 |
| Table 14.3.1.10 Summary of Adverse Events of Special Interest (AESI) by AESI Category, | |
| MedDRA System Organ Class and Preferred Term | 188 |
| Table 14.3.1.11 Summary of Gastrointestinal (GI) Adverse Events by MedDRA System Organization | an |
| Class and Preferred Term | 189 |
| Table 14.3.1.12 Summary of Most Frequent Treatment-Emergent Adverse Events by MedD | RA |
| System Organ Class and Preferred Term | 190 |
| Table 14.3.1.13 Time to First Gastrointestinal Treatment-Emergent Adverse Events | 191 |
| Table 14.3.1.14 Time to First Hepatic Treatment-Emergent Adverse Events | |
| Table 14.3.1.15 Summary of Treatment-Emergent Adverse Events, by Sex | |
| Table 14.3.1.16 Summary of Adverse Events of Special Interest (AESI) by AESI Category, | |
| MedDRA System Organ Class and Preferred Term, by Sex | 194 |
| Table 14.3.1.17 Summary of Elevation in Serum Transaminases Related Treatment-Emerge | |
| Adverse Events by MedDRA System Organ Class and Preferred Term, by Country | |
| Table 14.3.2.1 Haematology Values and Change from Baseline over Time | |
| Table 14.3.2.2 Clinical Significance of Haematology Values over Time | |
| Table 14.3.2.3 Shift in Haematology Values over Time | |
| Table 14.3.3.1 Serum Clinical Chemistry Values and Change from Baseline over Time | |
| Table 14.3.3.2 Clinical Significance of Serum Clinical Chemistry Values over Time | |
| Table 14.3.3.3 Shift in Clinical Chemistry Values over Time | |
| Table 14.3.3.4 Summary of Maximum Clinical Chemistry Values | |
| Table 14.3.3.5 Summary of Subjects Exceeding Hepatotoxicity Thresholds over Time | |
| Table 14.3.3.6 Time to Onset of Liver Function Test Abnormality | |
| Table 14.3.4.1 Urinalysis Values and Change from Baseline over Time | |
| Table 14.3.4.1 Official Significance of Urinalysis Values over Time | |
| Table 14.3.4.3 Shift in Urinalysis Values over Time | |
| Table 14.3.6.1 Summary of Overall ECG Interpretation over Time | |
| Table 14.3.6.2 Shift in Overall ECG Interpretation over Time | |
| Table 14.3.5.1 Summary of Echocardiography (Standard of Care) over Time | |
| Table 14.3.7.2 Summary of Subjects with Worsening in Echocardiography over Time | |
| Table 14.3.8.1.1 Summary of Lipid Accumulation in the Liver over Time | |
| Table 14.3.8.1.2 Summary of Lipid Accumulation in the Liver over Time (Sensitivity Analysis | |
| Excluding Site 12) Table 14.3.8.2.1 Shift in Lipid Accumulation in the Liver over Time | |
| | <b>ZZZ</b> |
| Table 14.3.8.2.2 Shift in Lipid Accumulation in the Liver over Time (Sensitivity Analysis - | ഹഹ |
| Excluding Site 12) | |
| Table 14.3.8.3.1 Summary of Lipid Accumulation in the Liver over Time | |
| Table 14.3.8.3.2 Summary of Lipid Accumulation in the Liver over Time | |
| Table 14.3.8.4.1 Summary of Lipid Accumulation Increase over Time | |
| Table 14.3.8.4.2 Summary of Lipid Accumulation Increase over Time | |
| Table 14.3.9.1 Summary of Tanner Staging over Time | |
| Table 14.3.9.2 Summary of Sex Hormones in patients with Tanner Stage ≥ 2 over Time | |
| Table 14.3.9.3 Shift in Tanner Staging Over Time | |
| Table 14.3.10.1 Summary of Pulmonary Function Test (PFT) Parameters and Change from | |
| Baseline over Time | |
| Table 14.3.11.1 Summary of Xanthoma Assessment over Time | |
| Table 14.3.11.2 Changes to pre-existing Xanthoma over Time | |
| Table 14.3.11.3 Summary of new xanthomas over Time | |
| Table 14.3.11.4 Cumulative changes to pre-existing Xanthoma over Time | |
| Table 14.3.12.1 Carotid Intima-Media Thickness and Flow-mediated Dilation Summary and | |
| Percentage Change from Baseline over Time | |
| Table 14.3.13.1 Summary of Palatability over Time | |
| Table 14.3.14.1 Summary of Diet Compliance over Time | 249 |

Date: 28JUN2024

Version: Final 5.0

| Listing 16.2.1.1 Subject Completions and Withdrawals | 251 |
|---|---|
| Listing 16.2.2.1 Eligibility | |
| Listing 16.2.2.2 Protocol Deviations | 252 |
| Listing 16.2.2.3 COVID-19 Protocol Deviations | |
| Listing 16.2.3.1 Analysis Sets | |
| Listing 16.2.4.1 Demography | |
| Listing 16.2.4.2 Diagnosis of HoFH | |
| Listing 16.2.4.3 Medical History | |
| Listing 16.2.4.4 Cardiovascular Medical History | |
| Listing 16.2.4.5 Prior/Run-in/Concomitant Medications | 261 |
| Listing 16.2.4.6 Lipid-lowering-therapy (LLT) Medications | |
| Listing 16.2.4.7 Prior/Run-in/Concomitant Procedures | |
| Listing 16.2.5.1 IMP Administration | |
| Listing 16.2.6.1 Lipoprotein Apheresis (LA) History | |
| Listing 16.2.6.2 Lipoprotein Apheresis (LA) Treatment | |
| Listing 16.2.7.1 Adverse Events | |
| Listing 16.2.7.2 Serious Adverse Events | 2/3 |
| Listing 16.2.8.1 Serum Clinical Chemistry (Fasting Lipid Panel) Values | 274 |
| Listing 16.2.8.2 Serum Clinical Chemistry (Metabolic Panel) Values | |
| Listing 16.2.8.3 Serum Clinical Chemistry (Liver Function Tests) Values | 279 |
| Listing 16.2.8.4 Serum Clinical Chemistry (Essential Fatty Acids) Values | 280 |
| Listing 16.2.8.5 Serum Clinical Chemistry (Fat Soluble Vitamin Levels) Values | 282 |
| Listing 16.2.8.6 Serum Clinical Chemistry (Hormones) Values | |
| Listing 16.2.8.7 Serum Clinical Chemistry (Sex Hormones) Values | |
| Listing 16.2.8.8 Serum Clinical Chemistry (Serum Lipase) Values | |
| Listing 16.2.8.9 Serum Haematology Values | |
| Listing 16.2.8.10 Urinalysis Values | |
| Listing 16.2.9.1 Vital Signs | |
| Listing 16.2.10.1 ECG Results | |
| Listing 16.2.11.1 Echocardiography Results | |
| Listing 16.2.12.1 Lipid Accumulation in the Liver Results | 293 |
| Listing 16.2.13.1 Physical Examination | 294 |
| Listing 16.2.13.2 Tanner Staging | |
| Listing 16.2.14.1 Pulmonary Function Test | |
| Listing 16.2.15.1 Pregnancy Test | |
| Listing 16.2.16.1 Visit Dates | |
| Listing 16.2.17.1 Xanthoma Examination | |
| Listing 16.2.17.2 Carotid Intima-Media Thickness (CIMT) | |
| Listing 16.2.17.3 Flow-mediated Dilation (FMD) | |
| Listing 16.2.17.4 Palatability | |
| Listing 16.2.19.1 Diet and Dietary Supplement Compliance | |
| Figure 14.1.5.1 Kaplan-Meier Plot of Time to Dose Reduction | 308 |
| Figure 14.1.5.2 Kaplan-Meier Plot of Time to Dose Interruption | 309 |
| Figure 14.2.1.1 Waterfall Plot of Percentage Change (%) from Baseline in Fasting Lipid Par | nel |
| at Week 24 by age group | |
| Figure 14.2.1.2 Forest Plot of Sub-group analysis for primary end point (percentage change | |
| week 24) | |
| Figure 14.2.1.3 Profile Plot of LSMeans percentage change from baseline over time in Fast | |
| , | _ |
| Lipid Panel | 312 |
| Figure 14.2.1.4 Forest Plot of Sub-group analysis for key secondary endpoint: Non-HDL-C | |
| (percentage change at week 24) | |
| Figure 14.2.1.5 Forest Plot of Sub-group analysis for key secondary endpoint: TC (percenta | |
| change at week 24) | 314 |
| Figure 14.2.1.6 Forest Plot of Sub-group analysis for key secondary endpoint: VLDL-C | |
| (percentage change at week 24) | 315 |
| Figure 14.2.1.7 Forest Plot of Sub-group analysis for key secondary endpoint: Apo B | |
| (percentage change at week 24) | 316 |
| Figure 14.2.1.8 Forest Plot of Sub-group analysis for key secondary endpoint: TG (percenta | |
| change at week 24) | |
| Figure 14.2.1.9 Forest Plot of Sub-group analysis for key secondary endpoint: Lp(a) | 517 |
| | 240 |
| (percentage change at week 24) | 318 |

| Figure 14.2.1.10 Profile Plot of percentage change from baseline over time in Fasting Lipid | J |
|---|---|
| Panel 319 Figure 44.3.3.4 Computative distribution function (CDF) plot of LDL C at Week 34 | 220 |
| Figure 14.3.2.1 Cumulative distribution function (CDF) plot of LDL-C at Week 24 | |
| Figure 14.3.2.2 Cumulative distribution function (CDF) plot of LDL-C over time | |
| Figure 14.3.2.3 Cumulative distribution function (CDF) plot of percentage change in LDL-C | |
| Week 24 | . 322 |
| Figure 14.3.2.4 Cumulative distribution function (CDF) plot of lowest percentage change in | |
| LDL-C from Week 8Figure 14.3.1.1 Subject profile for distribution of Treatment-Emergent adverse events and of the subject profile for the subject | |
| at time of event | |
| Figure 14.3.1.2 Age profile for distribution of Treatment-Emergent adverse events and | . 324 |
| MTD 325 | |
| Figure 14.3.1.3 Histogram of Time to First Gastrointestinal Treatment-Emergent Adverse | |
| Event 326 | |
| Figure 14.3.1.4 Histogram of Time to First Hepatic Treatment-Emergent Adverse Event | 327 |
| Figure 14.3.3.1 Individual subject profiles of liver function data | . 328 |
| Figure 14.3.3.2 AST profiles over time, by subject age | |
| Figure 14.3.3.3 ALT profiles over time, by subject age | |
| Figure 14.3.3.4 AST profiles over time, by subject MTD | |
| Figure 14.3.3.5 ALT profiles over time, by subject MTD | . 332 |
| Figure 14.3.3.6 Individual subject profiles of LDL-C data | |
| Figure 14.3.3.7 LDL-C profiles over time, by subject age | . 334 |
| Figure 14.3.3.8 LDL-C profiles over time, by subject MTD | |
| Figure 14.3.3.9 Spaghetti plot of lipid profiles over time | |
| Figure 14.3.3.10 eDISH plot of Maximum Post-Baseline ALT by Maximum Post-Baseline T | |
| Bilirubin | . 337 |
| Figure 14.3.3.11 eDISH plot of Maximum Post-Baseline AST by Maximum Post-Baseline T | |
| Bilirubin | |
| Figure 14.3.3.12 Subject profile for distribution of Liver Function Test Abnormalities and do | |
| at time of event | |
| Figure 14.3.5.1 Boxplot of Observed Vital Signs over Time | |
| Figure 14.3.5.2 Boxplot of Change from Baseline Vital Signs over Time | |
| Figure 14.3.5.3 Waterfall plot of change in BMI at Week 24, 56 and 104, by patient sex | |
| Figure 14.3.8.1 Scatter plot of change in hepatic fat up with change in BMI Z score up to we | |
| 56 and 104, by subject age | |
| and 104, by subject MTD | |
| Figure 14.3.8.3 Scatter plot of change in hepatic fat up to week 56 and 104 and time fom | . 344 |
| Lomitapide administration, by subject age | 3/15 |
| Figure 14.3.8.4 Scatter plot of change in hepatic fat up to week 56 and 104 and time from | . 040 |
| Lomitapide administration, by subject MTD | 346 |
| Figure 14.3.8.5 Cumulative distribution function (CDF) plot of percentage change in hepatic | c fat |
| over time | |
| Figure 14.3.8.6 Scatter plot of ALT vs hepatic fat over time | |
| Figure 14.3.8.7 Scatter plot of AST vs hepatic fat over time | |
| Figure 14.3.9.1 Waterfall plot of change in BMI Z score at Week 24, 56 and 104, by patient | |
| age 350 | |
| Figure 14.3.9.2 Waterfall plot of change in BMI Z score at Week 24, 56 and 104, by patient | |
| sex 351 | |
| Figure 14.3.9.3 Spaghetti plot of BMI Z score over time, by patient age and sex | . 352 |
| Figure 14.3.9.4 Spaghetti plot of BMI absolute value over time, by patient age and sex | . 353 |
| Figure 14.3.9.5 Spaghetti plot of weight absolute value over time, by patient age and sex | |
| Figure 14.3.9.6 Spaghetti plot of sexual maturation development over time | |
| Figure 14.3.9.7 Spaghetti plot of growth development over time | |
| Figure 14.3.9.8 Waterfall plot of change in BMI Z-score at Week 24, 56 and 104, by baseling | |
| BMI for Age Z-score | |
| Figure 14.3.9.9 Spaghetti plot of BMI Z-score over time, by baseline BMI for Age Z-score | |
| Figure 14.3.9.10 Individual spaghetti plot of weight and Z scores over time | |
| Figure 14.3.9.11 Waterfall plot of change from baseline to maximum weight loss | |
| Figure 14.3.9.12 Waterfall plot of change from baseline to minimum BMI z-score change | . 361 |

### 1 PROGRAMMING NOTES

"Summary statistics" for quantitative data will be recorded as n, mean, standard deviation, minimum, median and maximum, 25th & 75th percentile (as specified in shell). For categorical data, a frequency table (showing n and %) will replace this summary.

Data manipulations will be detailed as appropriate in the SAS code. Derived database (DDB) specifications will be created and maintained by Veristat.

All tables, listings and figures will use recommended ICH numbering.

Complex manipulations should be detailed in the body of the SAP text or as "programming notes" on the table shells.

Decimal places will be as follows (where applicable), where x is the precision of the raw data:

- x +2 (standard errors, standard deviations, CV%).
- x +1 (means, medians, confidence intervals).
- x (min and max).
- 1 decimal place (percentages). Percentages will not be displayed where n=0.

Percentages will be based on the number of subjects in the analysis set/population, for the relevant treatment group (regardless of time point), unless otherwise stated.

The 'missing' category, where used, will not include subjects who have withdrawn at earlier visits. Subjects with missing results or assessment not done at visit x will be included in the missing category only if they have a visit x or a visit greater than x in the visit date listing.

Page set-up specifications for the SAS output TFLs:

- Word document landscape
- Word document margins set to:
  - $\circ$  top = 2.54 cm
  - o bottom = 1.5 cm
  - left = 2 cm
  - o right = 2 cm
  - o gutter = 0 cm
  - o header = 1.25 cm
  - o footer = 1.25 cm
- Word document font: Courier New, 8pt
- SAS output options Is=141 ps=52

All output will be provided as individual and collated .rtf files.

The sponsor study number and sponsor name will be displayed in the top left hand side of the TFLs and page numbers will be displayed in the top right hand side of the TFLs.

Date: 28JUN2024  Version: Final 5.0 For each listing, only the visits/time points where the data was collected will be listed, including unscheduled assessments where applicable. Tables will show results for all visits and time points where data was collected, unless specified otherwise within the shell (see programming notes).

Other standards and conventions:

### General:

- o UK spelling used in all tables, listings and figures.
- Output spans entire width of page (where possible).
- Top line spanning output but no line at bottom.
- Numeric results aligned by decimal place.

### Listings only:

- Ordered by age group (5-10,11-15 and 16-<=17), visit and subject number (as applicable).
- All dates will be displayed as DDMONYYYY. Missing days will be displayed in the listings as 'UK', missing months as 'UNK' and missing years as 'UKUK'. Add footnote 'UK/UNK = Unknown.' where required.
- o Data will be presented in date order.
- Leave all footnote decodes such as L = ..., H = .... even if not actually within data listed.
- Where adding a footnote for decodes such as Route/Frequency, add all possible values from CRF rather than just those in the data.
- Where one row per subject no break lines. Where more than one row per subject – break after subject/visit/time point as applicable.

### Tables only:

- o Remove percentages when count is zero.
- All results should be aligned. For example, numbers from summary statistics should align with results from frequency counts.


Table 14.1.1.1 Subject Disposition (Enrolled Set)

| | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) | 1 1 |
|---|---|---|---|---|
| Screen Failures, n | XX | XX | XX | |
| Enrolled Set [1], n (%)* | XX (XX.X) | XX (XX.X) | (XX XX) XX | |
| Run-in Failures, n (%)* | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Completed Run-In Period, n (%)* | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Safety Set (SAF) [2], n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Full Analysis Set (FAS) [3], n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Completers Analysis Set (CAS) [4], n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Per Protocol Set (PPS) [5], n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Subjects who completed the Safety Phase (week 104) of the study, n $(\$)$ | XX (XX.X) | XX (XX.X) | (X. XX) XX | |
| Subjects who prematurely discontinued study, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Reason for study withdrawal n (%) | | | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Discontinuation of the study by sponsor | (XX.X) | XX (XX.X) | XX (XX.X) | |
| Lost to follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Non-compliance | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Pregnancy | (XX.X) | XX (XX.X) | XX (XX.X) | |
| Protocol Deviation | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Voluntary Withdrawal | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| COVID-19 | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | |

N = the number of subjects enrolled. n = the number of subjects meeting the criterion.

[\*] Percentages based off the Enrolled Set. All other percentages based off the Safety Analysis Set. [\*\*] The calculation of study duration excludes screen failure patients. [4] The Completers Analysis Set includes all subjects from the FAS who have not discontinued the Efficacy Phase (up to Week 24) of the study

<sup>[1]</sup> The Enrolled Set includes all subjects who pass screening and enter into the run-in period, irrespective of whether they receive the study treatment.

<sup>[2]</sup> The Safety Analysis Set includes all subjects who are treated with at least one dose of the IMP. [3] The Full Analysis Set includes all subjects who receive at least one dose of the IMP and who have a baseline and at least one postbaseline measurement of LDL-C.

<sup>[5]</sup> The Per Protocol Set includes all patients from the FAS who reasonably adhere to all protocol conditions (i.e. who have met the early irrespective of the reason for discontinuation.

eligibility criteria and receive planned study medication without important protocol deviations considered to have a serious impact on the efficacy results within the Efficacy Phase of the trial). Source: Listing 16.2.1.1 and Listing 16.2.3.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS

## SQN Clinical study no: OCH19003

Table 14.1.1.1 Subject Disposition (Enrolled Set)

| | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|
| Study duration (weeks) ** | | | |
| n | ×× | ×× | XX |
| Mean | x.xx | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Minimum | x.xx | XX.X | xx.x |
| Median | x.xx | XX.X | xx.x |
| Maximum | XX.X | ×××× | XX.X |
| Treatment duration (weeks) | | | |
| n | XX | XX | ×× |
| Mean | x.xx | XX.X | xx.x |
| SD | XX.XX | XX.XX | XX.XX |
| Minimum | XX.X | XX.X | xx.x |
| Median | x.xx | XX.X | xx.x |
| Maximum | x. xx | XX.X | ××.× |

N = the number of subjects enrolled. n = the number of subjects meeting the criterion.

\* Percentages based off the Enrolled Set. All other percentages based off the Safety Analysis Set.

\*\*] The calculation of study duration excludes screen failure patients.

[1] The Enrolled Set includes all subjects who pass screening and enter into the run-in period, irrespective of whether they receive the study treatment.

[2] The Safety Analysis Set includes all subjects who are treated with at least one dose of the IMP. [3] The Full Analysis Set includes all subjects who receive at least one dose of the IMP and who have a baseline and at least one post-

[4] The Completers Analysis Set includes all subjects from the FAS who have not discontinued the Bfficacy Phase (up to Week 24) of the study baseline measurement of LDL-C.

early irrespective of the reason for discontinuation. [5] The Per Protocol Set includes all patients from the FAS who reasonably adhere to all protocol conditions (i.e. who have met the eligibility criteria and receive planned study medication without important protocol deviations considered to have a serious impact on the

efficacy results within the Efficacy Phase of the trial). Source: Listing 16.2.1.1 and Listing 16.2.3.1

DATE OF EXTRACTION: XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXXX PROGRAM NAME: T XXX 01.SAS

Table 14.1.1.2 Subject Study Visits
 (Enrolled Set)

| | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|
| <pre>Run-in period: Visit 2 (Enrolment), n (%) Visit 3 (Compliance), n (%)</pre> | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| <pre>Efficacy Phase: Visit 4 (Week 0 / Day 0), n (%)</pre> | XX (XX.X) | XX (XX.X) | (XX.X) |
| 5 (Week 4 / Day | | | |
| Visit 6 (Week 8 / Day 56), n (%)<br>Visit 7 (Week 12 / Day 84), n (%) | (X.X)<br>(X.X)<br>(X.X) | (XXXX)<br>XX (XXXX) | XX (XX.X)<br>XX (XX.X) |
| 8 (Week 16 | | | |
| Visit 9 (Week 20 / Day 140), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Visit 10 (Week 24 / Day 168), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Safety Phase: | | | |
| Visit 11 (Week 28 / Day 196), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Visit 12 (Week 32 / Day 224), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Visit 13 (Week 36 / Day 252), n (%) | XX (XX.X) | XX (XX.X) | xx (xx.x) |
| Visit 14 (Week 40 / Day 280), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 15 (Week 44 / Day | | | |
| (Week | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Visit 17 (Week 52 / Day 364), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Visit 18 (Week 56 / Day 392), n (%) | XX (XX.X) | XX (XX.X) | xx (xx.x) |
| Visit 19 (Week 68 / Day 479), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Visit 20 (Week 80 / Day 560), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Visit 21 (Week 92 / Day 644), n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| End Of Treatment: | | | |
| Visit 22 (EOT / Week 104) | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| Follow-up: | | | |
| Visit 23 (Week 108) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | - | | |

N = the number of subjects enrolled, n = the number of subjects meeting the criterion. Percentages based off the Enrolled Set. Source: Listing 16.2.16.1

PROGRAM NAME: T\_XXX\_01.SAS DATE OF

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX

Table 14.1.2.1 Demography (Safety Analysis Set)

| Sex, n (%) Male Female Unknown Missing Age (years) Mean SD Minimum Median Meximum | | 41 | (N=XX) | 4 |
|---|---|---|---|---|
| | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | XX (XX.X) | (XX.X) XX | XX (XX.X) |
| | | XX (XX.X) | (XX.XX) XX | XX (XX.X) |
| | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mean SD Minimum Median Maximum | | ×× | ×× | XX |
| SD<br>Minimum<br>Median<br>Maximum | | x.xx | XX.X | XX.XX |
| Minimum<br>Median<br>Maximum | | XX.XX | XX.XX | XX.XX |
| Median<br>Maximum | | x.xx | XX.X | XX.X |
| Maximum | | x.xx | XX.X | XX.X |
| | | XX.X | XX.X | XX.X |
| Race, n (%) Black or African | African American | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| American Indian | Indian or Alaska Native | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Asian | | XX (XX.X) | (XX.X) XX | XX (XX.X) |
| Native Hawaiian or | iian or other Pacific | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Islander | | | | |
| Arabic | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| White | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | | (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Ethnicity, n (%) Hispanic or Latino | Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Hispanic or Latino | c or Latino | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Reported | T | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unknown | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | | XX (XX.X) | XX (XX.X) | XX (XX.X) |

DATE OF EXTRACTION: XXXXXXXXX

TIME OF RUN: XX:XX:XX

DATE OF RUN:XXXXXXXX

PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Age is calculated in years = [full] age in month (months + years) / 12]


N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100. [1] BMI = {weight(kg) / height(m)^2} [2] BSA (m^2) =  $\sqrt{[height(cm) \times weight(kg)]}$  / 3600] [Mosteller formula] [3] z scores and percentiles calculated using the WHO growth reference indicators for children aged 5 to 19 years Source: Listing 16.2.4.1, Listing 16.2.4.2, Listing 16.2.8.1

Table 14.1.2.1 Demography
(Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Country, n (%) | Germany | XX (XX.X) | XX (XX.X) | (XXX) XX |
| | Jpalii<br>Italv | | | |
| | Saudi Arabia | | | _ |
| | Tunisia | | | |
| | Israel | (X.XX) XX | XX (XX.X) | XX (XX.X) |
| Height (cm) at Baseline | и | XX | XX | XX |
| | Mean | X.XX | xx.x | x.xx |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.XX |
| | 25th percentile | XX.X | XX.X | XX.XX |
| | 75th percentile | x.xx | XX.X | XX.X |
| Weight (kg) at Baseline | ц | × | XX | XX |
| | Mean | XX.X | xx.x | xx.xx |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | X.XX | x.xx | xx.xx |
| | Median | X.XX | xx.x | x.xx |
| | Maximum | XX.X | xx.x | xx.xx |
| | 25th percentile | XX.X | XX.X | xx.xx |
| | 75th percentile | X.XX | XX.X | XX.X |
| $N$ = the number of subjects in the analysis set. n [1] $BMI = \{weight(kg) / height(m)^2\}$ | the analysis set. $n = the number of (m)^2$ | of subjects meeting the criterion. | (%) = $n/N*100$ . | |
| [2] BSA (m^2) = $\sqrt{\{\text{height(cm) x weight(kg)}\}}$ / 3600] [3] z scores and percentiles calculated using the WH Source: Listing 16.2.4.1, Listing 16.2.4.2, Listing | x weight(kg)} / 3600] [Mostell alculated using the WHO growth reing 16.2.4.2, Listing 16.2.8.1 | [2] BSA (m^2) = $V[\{\text{height}(\text{cm}) \times \text{weight}(\text{kg})\}$ / 3600] [Mosteller formula] [3] z scores and percentiles calculated using the WHO growth reference indicators for children aged Source: Listing 16.2.4.1, Listing 16.2.4.2, Listing 16.2.8.1 | ed 5 to 19 years | |
| PROGRAM NAME: T_XXX_01.SAS | DATE OF RUN:XXXXXXXXX TIME OF | TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX | N:XXXXXXXX | |

NOTES: Age is calculated in years = [full age in month (months + years) / 12]

Table 14.1.2.1 Demography
(Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Body mass index (kg/m^2) at<br>Baseline [1] | и | XX | ×× | XX |
| | Mean | XX.X | x.xx | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.XX | xx.xx | XX.XX |
| | Median | XX.XX | XX.X | XX.X |
| | Maximum | x.xx | ××.× | XX.X |
| | 25th percentile | x.xx | ××.× | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X |
| Body surface area (BSA) at Baseline | а | ×× | XX | XX |
| | Mean | ×·×× | × · × × | × · ×× |
| | SD | x | × | ×× ·×× |
| | Minimum | ×.×× | XX.X | XX.X |
| | Median | XX.XX | XX.X | XX.X |
| | Maximum | XX.XX | XX.X | XX.X |
| | 25th percentile | XX.XX | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X |
| Height percentile [3] | ជ | XX | XX | ×× |
| | Mean | xx.xx | ××.×× | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.X | XX.X | XX.XX |
| | Median | XX.XX | XX.X | XX.X |
| | Maximum | XX.XX | ××.×× | XX.X |
| | 25th percentile | XX.X | XX.X | xx.x |
| | 75th percentile | XX.X | XX.X | XX.X |
| N = the number of subjects in the analysis set. n = [1] BMI = {weight(kg) / height(m)^2} $\frac{1}{2}$ [2] BAI = $\frac{1}{2}$ [2] BAI = $\frac{1}{2}$ [3] [3] [4] [5] [5] [6] [6] [6] [7] [6] [7] [7 | lysis set. n = the number of subjects meeting the criterion. (%) = $n/N*100$ . | eting the criterion. | (%) = $n/N*100$ . | |

NOTES: Age is calculated in years = [full] age in month (months + years) / 12]

<sup>[2]</sup> BSA (m^2) =  $\sqrt{[\{\text{height(cm) x weight(kg)}\}}$  / 3600] [Mosteller formula] [3] z scores and percentiles calculated using the WHO growth reference indicators for children aged 5 to 19 years Source: Listing 16.2.4.1, Listing 16.2.4.2, Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN: XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.1.2.1 Demography
(Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years $(N=XX)$ | Overall (N=XX) |
|---|---|---|---|---|
| | | : | : | : |
| Height 2 Score [3] | n | ×× | ×× | ×× |
| | Mean | XX.XX | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.XX | ××.×× | XX.X |
| | Median | XX.XX | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.X |
| | 25th percentile | XX.XX | XX.X | XX.X |
| | 75th percentile | x.xx | XX.X | XX.X |
| BMI percentile [3] | п | XX | XX | ×× |
| | Mean | XX.X | xx.xx | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.XX | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.X |
| | 25th percentile | XX.XX | XX.X | XX.X |
| | 75th percentile | X.XX | XX.X | XX.X |
| BMI Z Score [3] | п | XX | XX | ×× |
| | Mean | x.xx | xx.xx | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.X |
| | 25th percentile | XX.X | XX.X | XX.X |
| | 75th percentile | XX.XX | XX.XX | XX.X |

DATE OF EXTRACTION: XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXXX PROGRAM NAME: T\_XXX\_01. SAS

NOTES: Age is calculated in years = [full age in month (months + years) / 12]

<sup>[2]</sup> BSA (m^2) =  $V[\{\text{height(cm} \times \text{weight(kg)}\} / 3600]$  [Mosteller formula] [3] z scores and percentiles calculated using the WHO growth reference indicators for children aged 5 to 19 years Source: Listing 16.2.4.1, Listing 16.2.4.2, Listing 16.2.8.1

Table 14.1.2.2 Baseline Lipids (Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| | | 4 | | |
| LDL-C (mg/dL) | ч | ×× | ×× | XX |
| | Mean | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.XX | xx.x | XX.XX |
| | Median | XX.X | XX.X | x.xx |
| | Maximum | XX.X | XX.XX | x.xx |
| | 25th percentile | XX.XX | XX.XX | X.XX |
| | 75th percentile | ×××× | XX.X | XX.X |
| Non-HDL-C (mg/dL) | ព | XX | XX | XX |
| | Mean | XX.XX | ××.×× | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.XX | x.xx |
| | Maximum | XX.X | XX.XX | x.xx |
| | 25th percentile | XX.XX | XX.XX | XX.XX |
| | 75th percentile | ×·×× | XX.X | XX.X |
| Total Cholesterol (TC) (mg/dL) | ជ | XX | XX | XX |
| | Mean | XX.XX | XX.XX | X.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.XX | XX.X | XX.XX |
| | Median | XX.X | ××.×× | ×.×× |
| | Maximum | XX.XX | xx.x | XX.XX |
| | 25th percentile | XX.X | ××.×× | ×.×× |
| | 75th percentile | x.xx | xx.xx | XX.XX |

DATE OF RUN:XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS  Date: 28JUN2024 Version: Final 5.0

Table 14.1.2.2 Baseline Lipids (Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| VLDL-C (mg/dL) | а | XX | XX | XX |
| | Mean | ×.×. | XX.XX | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | X.XX | x.xx | XX.X |
| | Median | XX.XX | XX.X | XX.X |
| | Maximum | X.XX | x.xx | XX.X |
| | 25th percentile | X.XX | XX.XX | XX.X |
| | 75th percentile | x.xx | XX.XX | XX.X |
| Apo B (mg/dL) | ч | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | X.XX | XX.XX | XX.X |
| | Median | X.XX | XX.XX | XX.X |
| | Maximum | XX.XX | x.xx | ××.×× |
| | 25th percentile | X.XX | x.xx | XX.X |
| | 75th percentile | x.xx | XX.X | XX.X |
| Triglycerides (TG) (mg/dL) | и | XX | XX | XX |
| | Mean | X.XX | x.xx | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | X.XX | XX.XX | XX.X |
| | Median | x.xx | x.xx | XX.X |
| | Maximum | x.xx | x.xx | XX.X |
| | 25th percentile | XX.X | XX.X | XX.X |
| | 75th percentile | XX.XX | x.xx | XX.X |

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


Table 14.1.2.2 Baseline Lipids (Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Apo Al (mg/dL) | п | XX | XX | ×× |
| | Mean | XXXX | XX.XX | x.xx |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.X | x.xx | x.xx |
| | Median | XX.X | x.xx | x.xx |
| | Maximum | XX.XX | x.xx | xx.x |
| | 25th percentile | XXXX | XX.X | xx.x |
| | 75th percentile | x.xx | XX.X | XX.X |
| HDL-C (mg/dL) | u | ×× | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.XX | XX.X | xx.x |
| | Median | XX.XX | XX.X | xx.x |
| | Maximum | XX.X | x.xx | x.xx |
| | 25th percentile | XX.X | xx.xx | ×.×× |
| | 75th percentile | x.xx | XX.X | XX.X |
| Lp(a) (mg/dL) | u | ×× | XX | XX |
| | Mean | XX.XX | x.xx | xx.x |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.X | XX.X | x.xx |
| | Median | XX.X | XX.X | ××.× |
| | Maximum | XX.X | XX.X | ××.× |
| | 25th percentile | XX.X | XX.X | ×.×× |
| | 75th percentile | x.xx | XX.X | XX.X |

THE TOTAL PRINCE TO THE TO THE TOTAL PRINCE TO

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS  Date: 28JUN2024 Version: Final 5.0

Table 14.1.2.2 Baseline Lipids (Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Lp(a) (nmol/L) | и | XX | XX | XX |
| | Mean | X.XX | XX.XX | ×.×× |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.XX | XX.XX | ××.×× |
| | Median | XX.XX | XX.XX | ××.×× |
| | Maximum | XX.XX | XX.XX | ××.×× |
| | 25th percentile | XX.XX | XX.XX | ××.×× |
| | 75th percentile | x.xx | XX.XX | XX.X |
| TC/HDL-C | ч | ×× | XX | ×× |
| | Mean | XX.X | XX.X | xx.x |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.X | XX.X | x.xx |
| | Median | XX.X | XX.X | x.xx |
| | Maximum | XX.X | XX.X | xx.x |
| | 25th percentile | XX.X | XX.X | xx.x |
| | 75th percentile | XX.X | XX.X | XX.X |

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.1.2.3 Diagnosis of HoFH (Safety Analysis Set)

| | Statistics | 5 to $10 \text{ years}$ $(N=XX)$ | 11 to 17 years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Duration of HoFH diagnosis (weeks) | | | | |
| | п | XX | ×× | XX |
| | Mean | XX.X | XX.X | ×.×. |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | X |
| | Median | XX.X | XX.X | XX.XX |
| | Maximum | XX | XX | XX |
| | 25th percentile | XX.X | XX.X | ×.×. |
| | 75th percentile | XX.X | XX.X | XX.X |
| Genetic confirmation of 2 mutant alleles, n (%) | Kes | (X.XX) XX | (X.X.X) XX | XX (XX.X) |
| | No | XX (XX.X) | XX (XX.X) | (XX.X) |
| Type of mutant allele, n (%) | LDLR gene locus | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Apo B gene locus | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | PCSK9 gene locus | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | LDLRAP1 gene locus | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Unknown | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | (XX.X) |
| LDL receptor function mutation | LDLR-deficient mutation | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | LDLR-defective mutation | XX (XX.X) | XX (XX.X) | XX (XX.X) |

<sup>[1]</sup> Duration of diagnosis is defined as the time in weeks from diagnosis to baseline. Source: Listing 16.2.4.2

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01. SAS

Table 14.1.2.3 Diagnosis of HoFH (Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| An untreated LDL-C >500mg/dL (13mmol/L) or treated LDLC >300mg/dL (8mmol/L) AND cutaneous or tendon xanthoma before age of 10 | Yes | (XX (XX XX) | (XX.X) | XX (XX.X) |
| years? n (%) | No | XX (XX.X) | XX (XX.X) | (XX.X) |
| An untreated LDL-C >500mg/dL (13mmol/L) or treated LDLC >300mg/dL (8mmol/L) aND intreated | K e s | (XX.X) XX | XX (XX.X) | XX (XX.X) |
| LDL-C levels consistent with HoFH in both parents? n (%) | No | XX (XX.X) | (XXX.X) | (x.xx) xx |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100. [1] Duration of diagnosis is defined as the time in weeks from diagnosis to baseline. Source: Listing 16.2.4.2

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS 

Table 14.1.3.1 Medical History (Safety Analysis Set)

Ongoing conditions

| System organ class<br>Preferred term | 5 to 10 years (N=XX) | 11 to 17 years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with any medical history | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| System organ class 1 | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 4 | (XXXX) XX | XX (XX.X) | XX (XX.X) |

Medical history events were coded using the MedDRA Dictionary, version xx.x. System organ classes (SOC) are ordered in decreasing frequency of the total number of subjects with medical histories reported in each SOC and preferred terms are ordered within a SOC in decreasing frequency of the total number of subjects with each medical history. N = the number of subjects in the analysis set. n = the number of subjects with medical history. (%) = n/N\*100. Source: Listing 16.2.4.3

DATE OF RUN:XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for 'Previous conditions'.

Table 14.1.3.2 Cardiovascular History (Safety Analysis Set)

Ongoing conditions

| System organ class<br>Preferred term | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with any cardiovascular history | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| System organ class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 4 | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| System organ class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred term 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Cardiovascular history events were coded using the MedDRA Dictionary, version xx.x.. System organ classes (SOC) are ordered in decreasing frequency of the total number of subjects with cardiovascular histories reported in each SOC and preferred terms are ordered within a SOC in decreasing frequency of the total number of subjects with each cardiovascular history. N = the number of subjects in the analysis set. n = the number of subjects with medical history. (%) = n/N\*100. Cardiovascular History will be identified using pre-specified SOC and PT terms.

Source: Listing 16.2.4.4

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for 'Previous conditions'.

Table 14.1.3.3 Cardiovascular Disease History at Screening (Safety Analysis Set)

XX (XX.X) XX (XX.X) XX (XX.X) ××. ×× × × × (XX.XX) XX (XX.X) XX.X Overall (N=XX)11 to 17 years XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) (X.XX) XX ××.× ××. ×.× XX.X (N=XX)× 5 to 10 years XX (XX.X) XX (XX.X) XX (XX.X) ××.×× ×× XX (XX.X) XX (XX.X) XX.X ××.× XX.X (X=XX)× Duration of cardiovascular disease (months)\* Subjects with cardiovascular history at screening, n (\$)Cardiovascular disease ongoing, n (%) Type of cardiovascular disease Coronary artery disease, n (%) Valvular disease, n (%) 25th percentile 75th percentile Other, n (%) Minimum Maximum Median Mean

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS 

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = m/n\*100. \* Duration of cardiovascular disease (months). For those with ongoing CVD, duration is calculated up to date of screening visit. Source: Listing 16.2.4.4

# SQN Clinical study no: OCH19003

Table 14.1.4.1 Prior and 'Run-in Medications' Medications (Safety Analysis Set)

| Medication class<br>Standardised medication name | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with any prior and/or 'Run-in' medication | (XX.X) | (XX) XX | XX (XX.X) |
| Medication class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Medication class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Medications were coded using WHO Drug Dictionary, version xxx. Medication classes and standardised medication names are ordered by descending frequency.

Prior medications / procedures are defined as those that started and ended prior to the enrolment date visit (visit 2) (i.e. start of the 'run-in period').

Run-in period' medications / procedures are defined as those that are ongoing at the time of starting the 'run-in' period (i.e. Visit 2) or N = the number of subjects in the analysis set receiving the treatment. n = the number of subjects taking a prior/'run-in' medication. (%) started after the start of the 'run-in' period, but before the time of first administration of study treatment.

[\*] Indicates prior medication only. Source: Listing 16.2.4.5

n/N\*100.

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Please flag (\*) medications that are prior only medications.

# SQN Clinical study no: OCH19003

Table 14.1.4.2 Concomitant Medications
(Safety Analysis Set)

| Medication class<br>Standardised medication name | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Subjects with any concomitant medication | XX (XX.X) | XX (XX.X) | (XX.X) |
| Medication class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 1 | XX (XX.X) | XX (XX.X) | (XXXXX) XX |
| Standardised medication name 2 | XX (XX.X) | XX (XX.X) | (XX.X) |
| Standardised medication name 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 4 | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| Medication class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 4 | (X, XX) XX | (X, XX) XX | (XXXX) |

(

Medications were coded using WHO Drug Dictionary, version xxx.

Medication classes and standardised medication names are ordered by descending frequency.

Concomitant medications / procedures are defined as those that are ongoing at the time of first administration of study treatment or started on or after the time of first administration of study treatment or started prior to the end / last dose of study treatment. If medication / procedure dates are incomplete and it is not clear whether the medication / procedure was concomitant, it will be assumed to be concomitant. N = 1 the number of subjects in the analysis set receiving the treatment. n = 1 the number of subjects taking a concomitant medication. (%) =

Source: Listing 16.2.4.5

PROGRAM NAME: T XXX 01.SAS DATE OF RUN: XXXXXXXXX TIME OF F

XXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

Table 14.1.4.3 Lipid-Lowering-Therapy Medications (Safety Analysis Set)

Prior and 'Run-in' LLT medications

| Medication class<br>Standardised medication name | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with any prior and/or 'run-in' LLT medication | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Subjects with $>= 2$ 'run-in' LLT medications | XX (XX.X) | (XX.X) | (XX.X) |
| Subjects with $>=$ 3 'run-in' LLT medications | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Medication class 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 1 | (X. XX) XX | XX (XX.X) | (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Standardised medication name 2 | (XX.XX) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 4 | XX (XX.X) | XX (XX.X) | xx (xx.x) |
| Medication class 2 | XX (XX.X) | XX (XX.X) | (X.XX) XX |
| Standardised medication name 1 | (XX.XX) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Standardised medication name 3 | (XX.XX) | XX (XX.X) | (XX (XX.X) |
| Standardised medication name 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Medications were coded using WHO Drug Dictionary, version xxx.

Medication classes and standardised medication names are ordered by descending frequency. Prior Lipid-lowering therapy medications and procedures are defined as those that started and ended prior to the enrolment visit (visit 2) date (i.e. start of the 'run-in period').

the enrolment visit (visit 2) date (i.e. start of the 'run-in period') and / or started after the start of the 'run-in period', but before the Run-in' periord Lipid-lowering therapy medications and procedures are defined as any lipid-lowering therapy or procedure that are ongoing at time of first administration of study treatment.

N = the number of subjects in the analysis set receiving the treatment. n = the number of subjects with a prior and/or 'run-in' medication.

[\*] Indicates prior medication only. (%) = n/N\*100.

PROGRAM NAME: T\_XXX\_01.SAS

Source: Listing 16.2.4.6

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX DATE OF RUN:XXXXXXXX Repeat for Concomitant LLT medications (efficacy phase); Concomitant LLT medications (safety phase). Update first row table text and footnotes accordingly. Please flag (\*) medications that are prior only medications. NOTES:

SQN Clinical study no: OCH19003

Table 14.1.4.5 Procedures (Safety Analysis Set)

| Procedure category<br>Indication | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with any procedure | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Procedure category 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Indication 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Indication 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Indication 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Indication 4 | XX (XX.X) | XX (XX.X) | xx (xx.x) |
| Procedure category 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Indication 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Indication 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Indication 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Indication 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Etc | | | |
| Procedures were coded using the MedDRA Dictionary, version $xx.x.$ N = the number of subjects in the analysis set receiving the treatment. n = the number of subjects with procedure. (%) = $n/N*100$ . | ry, version xx.x.<br>receiving the treatment. n = the n | number of subjects with procedur | e. (%) = $n/N*100$ . |

Source: Listing 16.2.4.7

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

# SQN Clinical study no: OCH19003

Table 14.1.4.6 Days from most recent apheresis to the corresponding LDL-C primary efficacy assessment (Safety Analysis Set)

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) |
|---|---|---|---|
| Established regimen during run-in | Twice a week | (XX,X) | (X, XX) XX |
| | Weekly | | |
| | Every two weeks | XX (XX.X) | |
| | Other | XX (XX.X) | XX (XX.X) |
| Weighted average number of days from previous LA during run-in (days) $[1]$ | ď | ×× | XX |
| | Mean | XX.XX | XX.X |
| | SD | XX.XX | XX.XX |
| | Minimum | ×× | XX |
| | Median | x.xx | XX.X |
| | Maximum | ×× | XX |
| | 25th percentile | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X |
| Days from most recent apheresis to LDL-C assessment on [2]: | | | |
| Baseline | ч | ×× | ×× |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Minimum | XX | XX |
| | Median | XX.XX | XX.X |
| | Maximum | ×× | XX |
| | 25th percentile | XX.X | XX.X |
| | 75th percentile | XX.X | ××.× |
| Week 24/LOCF | u | XX | ×× |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Minimum | ×× | XX |
| | Median | XX.X | XX.X |
| | Maximum | XX | XX |
| | 25th percentile | XX.X | XX.X |
| | 75th percentile | XX.X | ×.×× |

Only subjects on apheresis at baseline are presented.

<sup>[1]</sup> Established apheresis regimen during run-in in days. The weighted average number of days is summarised.

[2] Days from most recent apheresis to baseline LDL-C assessment and to Week 24 are summarised. For subjects discontinuing before Week 24, the duration between the most recent apheresis and the LDL-C assessment that was carried forward is presented.

N= the number of subjects in the analysis set receiving the treatment. n = the number of subjects with procedure. (%) = n/N\*100.

## Amryt Pharma study no: APH-19

# SQN Clinical study no: OCH19003

Source: Listing 16.2.6.2, Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

For discontinued subjects, note the Week number used for the LOCF in the footnotes. Add categories for established regimen as applicable. NOTES:


Table 14.1.5.1 Study Drug Exposure and Dosing (Safety Analysis Set)

Study Phase

| | | C 7 C + L | | |
|---|---|---|---|---|
| | | o to lu years | II to I/ Years | Overall |
| | SCACISCICS | (N=AA) | (N=AX) | (N=AX) |
| Exposure (weeks) | и | ×× | XX | ×× |
| | Mean | XX.XX | XX.X | ××.×× |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | XX | ×× |
| | Median | XX.X | XX.XX | ××.×× |
| | Maximum | ×× | XX | ×× |
| | 25th percentile | xx.x | XX.XX | x.xx |
| | 75th percentile | XX.X | XX.X | XX.X |
| Exposure (mg / day) | и | ×× | XX | ×× |
| | Mean | xx.x | ××.×× | x.xx |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | ×× |
| | Median | xx.x | XX.XX | x.xx |
| | Maximum | ×× | XX | ×× |
| | 25th percentile | xx.x | XX.XX | x.xx |
| | 75th percentile | XX.X | XX.X | XX.X |
| Maximum Tolerated Dose (mg), n (%) | 5mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 10mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 20mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 30mg | XX (XX.X) | XX (XX.X) | (XX.XX) |
| | 40mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 60mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Exposure to maintenance dose (weeks) | и | ×× | XX | ×× |
| | Mean | XX.XX | XX.X | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | XX | ×× |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | ×× | XX | ×× |
| | 25th percentile | x.x. | ××.× | xx.x |
| | 75th percentile | XX.X | x.xx | XX.X |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100.

## SQN Clinical study no: OCH19003

[1] Subject compliant for IMP dosing has been medically reviewed on a patient level basis. Subjects will be considered compliant if 80% to 100% of IMP doses have been taken.

Source: Listing 16.2.5.1

SOUTH TERRETING TO.Z.O.T

NOTES:

PROGRAM NAME: T XXX 01.SAS DATE OF RUN: XXXXXXXXX TIME OF RUN: XX:XX:XX

DATE OF EXTRACTION:XXXXXXXX

Additional doses may be added to Maximum Tolerated Dose as appropriate. Subject percentage compliance for dosing as per protocol (Efficacy Phase) - Use post-baseline study visits Week 4 to Week 24 inclusive

Subject percentage compliance for dosing as per protocol (Safety Phase) - Use post-baseline study visits Week 28 to Week 104 inclusive

Subject percentage compliance for dosing as per protocol (Overall) - Use post-baseline study visits Week 4 to Week 104 inclusive If a subject discontinues early during the efficacy phase, Use post-baseline study visits Week 4 to Week 24 and EOI/Week 104, as

For the compliant with IMP dosing present only the corresponding to the study phase.

Table 14.1.5.1 Study Drug Exposure and Dosing (Safety Analysis Set)

Study Phase

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Number of Doses Received | £ | XX | XX | XX |
| | Mean | XX.X | X.XX | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX |
| | Median | ××.×× | XX.XX | ××.×× |
| | Maximum | XX | ×× | ×× |
| | 25th percentile | XX.X | XX.X | xx.x |
| | 75th percentile | XX.X | XX.X | XX.X |
| Number of Dose Increases | п | XX | XX | XX |
| | Mean | xx.x | XX.XX | xx.x |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | ×× |
| | Median | xx.x | XX.XX | xx.x |
| | Maximum | XX | XX | ×× |
| | 25th percentile | XX.X | XX.X | xx.x |
| | 75th percentile | XX.X | XX.X | XX.X |
| Number of Dose Reductions | ជ | ×× | XX | XX |
| | Mean | XX.X | x.xx | xx.x |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | ×× |
| | Median | xx.x | XX.XX | xx.x |
| | Maximum | ×× | ×× | XX |
| | 25th percentile | XX.X | ×.×× | xx.x |
| | 75th percentile | XX.X | XX.XX | XX.X |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100. [1] Subject compliant for IMP dosing has been medically reviewed on a patient level basis. Subjects will be considered compliant if 80% to 100% of IMP doses have been taken. Source: Listing 16.2.5.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS NOTES: Additional doses may be added to Maximum Tolerated Dose as appropriate.
Subject percentage compliance for dosing as per protocol (Efficacy Phase) - Use post-baseline study visits Week 4 to Week 24 inclusive
Subject percentage compliance for dosing as per protocol (Safety Phase) - Use post-baseline study visits Week 28 to Week 104

Subject percentage compliance for dosing as per protocol (Overall) - Use post-baseline study visits Week 4 to Week 104 inclusive If a subject discontinues early during the efficacy phase, Use post-baseline study visits Week 4 to Week 24 and EOI/Week 104, as

appropriate. For the compliant with IMP dosing present only the corresponding to the study phase.


Table 14.1.5.1 Study Drug Exposure and Dosing (Safety Analysis Set)

Study Phase

| | | 5 to 10 years | 11 to 17 years | Overall |
|---|---|---|---|---|
| | Statistics | (N=XX) | (N=XX) | (N=XX) |
| | | ; | : | : |
| Number of Dose Interruptions | и | × | × | ×× |
| | Mean | xx.xx | XX.X | xx.x |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | X | XX | XX |
| | Median | ×××× | ×.×× | ××.×× |
| | Maximum | ×× | XX | XX |
| | 25th percentile | XX.X | x.xx | xx.x |
| | 75th percentile | XX.X | x.xx | XX.X |
| Number of Dose Reductions due to concomitant medication | и | X | XX | ×× |
| | Mean | XX.X | x.xx | xx.x |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | XX | XX |
| | Median | ×××× | xx.xx | ××.×× |
| | Maximum | XX | XX | XX |
| | 25th percentile | XX.X | x.xx | xx.x |
| | 75th percentile | XX.X | XX.X | XX.X |
| Number of Dose Reductions due to adverse events | и | XX | XX | XX |
| | Mean | XX.X | x.xx | xx.x |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | XX | XX |
| | Median | ××.×× | XX.X | xx.x |
| | Maximum | XX | XX | XX |
| | 25th percentile | XX.X | XX.XX | xx.x |
| | 75th percentile | XX.X | XX.X | XX.X |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100. [1] Subject compliant for IMP dosing has been medically reviewed on a patient level basis. Subjects will be considered compliant if 80% to 100% of IMP doses have been taken. Source: Listing 16.2.5.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF RUN:XXXXXXXX

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

NOTES: Additional doses may be added to Maximum Tolerated Dose as appropriate.

Subject percentage compliance for dosing as per protocol (Efficacy Phase) - Use post-baseline study visits Week 4 to Week 24 inclusive

Subject percentage compliance for dosing as per protocol (Safety Phase) - Use post-baseline study visits Week 28 to Week 104 inclusive

Subject percentage compliance for dosing as per protocol (Overall) - Use post-baseline study visits Week 4 to Week 104 inclusive If a subject discontinues early during the efficacy phase, use post-baseline study visits Week 4 to Week 24 and EOI/Week 104, as

appropriate. For the compliant with IMP dosing present only the corresponding to the study phase. Date: 28JUN2024 Version: Final 5.0


Table 14.1.5.1 Study Drug Exposure and Dosing (Safety Analysis Set)

Study Phase

| | | 5 to 10 years | 11 to 17 years | Overall |
|---|---|---|---|---|
| | Statistics | (N=XX) | (N=XX) | (N=XX) |
| Number of Dose Interruptions due to concomitant medication | ជ | XX | XX | ×× |
| 1000 | Mean | XX.X | ×××× | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX |
| | Median | XX.X | XX.XX | ×.×× |
| | Maximum | XX | XX | ×× |
| | 25th percentile | XX.X | XX.XX | ×.×× |
| | 75th percentile | XX.X | XX.X | XX.XX |
| Number of Dose Interruptions due to adverse events | g | XX | XX | ×× |
| | Mean | xx.x | XX.X | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | ×× |
| | Median | ××.× | XX.X | ×.×. |
| | Maximum | ×× | XX | XX |
| | 25th percentile | XX.X | XX.X | ×.×× |
| | 75th percentile | XX.X | XX.X | XX.XX |
| Number of Drug Discontinuations due to adverse events | а | XX | XX | XX |
| | Mean | XX.X | ×.×× | ×.×× |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | XX | XX |
| | Median | XX.X | XX.X | ×.×. |
| | Maximum | XX | XX | ×× |
| | 25th percentile | XX.X | x.xx | ×.×× |
| | 75th percentile | XX.X | XX.XX | x.xx |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100. [1] Subject compliant for IMP dosing has been medically reviewed on a patient level basis. Subjects will be considered compliant if 80% to 100% of IMP doses have been taken.

Source: Listing 16.2.5.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Additional doses may be added to Maximum Tolerated Dose as appropriate.

Subject percentage compliance for dosing as per protocol (Efficacy Phase) - Use post-baseline study visits Week 4 to Week 24 inclusive

Subject percentage compliance for dosing as per protocol (Overall) - Use post-baseline study visits Week 4 to Week 104 inclusive If a subject discontinues early during the efficacy phase, use post-baseline study visits Week 4 to Week 24 and EOI/Week 104, as Subject percentage compliance for dosing as per protocol (Safety Phase) - Use post-baseline study visits Week 28 to Week 104 inclusive

appropriate. For the compliant with IMP dosing present only the corresponding to the study phase.


Table 14.1.5.1 Study Drug Exposure and Dosing (Safety Analysis Set)

Study Phase

| | Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Dose at Drug Discontinuation due to adverse events | 2 mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| (11.6) | 5mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 10mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 20mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 30mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 40mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 60mg | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Subject compliant with IMP dosing, n (%) [1] | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| (billoacy Fnase) | NO | (XX.X) | (XX.X) | (XX.X) |
| Subject compliant with IMP dosing, n (%) [1] | Yes | XX (XX.X) | XX (XX.X) | (XX.X) |
| (Salety Flase) | NO | XX (XX.X) | XX (XX.X) | (XX.X) |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100. [1] Subject compliant for IMP dosing has been medically reviewed on a patient level basis. Subjects will be considered compliant if 80% to 100% of IMP doses have been taken. Source: Listing 16.2.5.1

PROGRAM NAME: T\_XXX\_01.SAS DATE OF RUN: XXXXXXXXX

DATE OF RUN:XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX

NOTES: Additional doses may be added to Maximum Tolerated Dose as appropriate.

Subject percentage compliance for dosing as per protocol (Efficacy Phase) – Use post-baseline study visits Week 4 to Week 24 inclusive

Subject percentage compliance for dosing as per protocol (Overall) - Use post-baseline study visits Week 4 to Week 104 inclusive If a subject discontinues early during the efficacy phase, use post-baseline study visits Week 4 to Week 24 and EOI/Week 104, as Subject percentage compliance for dosing as per protocol (Safety Phase) – Use post-baseline study visits Week 28 to Week 104 inclusive

appropriate. For the compliant with IMP dosing present only the corresponding to the study phase.

Table 14.1.5.2 Summary of Compliance to IMP (Safety Analysis Set)

| Visit | m1 | 5 to 10 years (N=XX) | m2 | 11 to 17 years (N=XX) | u. | Overall (N=XX) |
|---|---|---|---|---|---|---|
| Week 4 | XX | XX (XX.X) | ×× | XX (XX.X) | XX | XX (XX.X) |
| Week 8 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Week 12 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Week 16 | ×× | XX (XX.X) | XX | | XX | XX (XX.X) |
| <br>Week 104 | XX | XX (XX.X) | × | XX (XX.X) | XX | XX (XX.X) |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. mx = number of subjects attending the visit. (%) = n/mx\*100. Subject compliant for IMP dosing has been medically reviewed on a patient level basis. Subjects will be considered compliant if 80% to 100% of IMP doses have been taken. Source: Listing 16.2.5.1

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.1.5.3 Time to Dose Reduction and Interruption

(Safety Analysis Set) Overall / Efficacy Phase

| | 5 to 10 years | 11 to 17 years |
|---|---|---|
| Statistics | (N=XX) | (XX=N) |
| Number of subjects with dose reduction, n (%) | XX (XX.X) | XX (XX.X) |
| Number of subjects censored, n (%) | XX (XX.X) | XX (XX.X) |
| Kaplan-Meier estimates of time to dose reduction | | |
| (weeks) | | |
| 25th percentile | XX.X | XX.X |
| 95% CI [1] | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| Median | XX.X | XX.X |
| 95% CI [1] | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| 75th percentile | XX.X | XX.X |
| 95% CI [1] | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| Number of subjects with dose interruption, n (%) | XX (XX.X) | XX (XX.X) |
| Number of subjects censored, n (%) | XX (XX.X) | XX (XX.X) |
| Kaplan-Meier estimates of time to dose interruption | | |
| (weeks) | | |
| 25th percentile | XX.X | XX.X |
| 95% CI [1] | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| Median | XX.X | XX.X |
| 95% CI [1] | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| 75th percentile | XX.X | XX.X |
| 95% CI [1] | (XX.XX, XX.XX) | (XX.XX, XX.XX) |

Time to dose reduction is defined as the time (weeks) from the date of the start of the respective phase to the time of first dose reduction, they will be counted as an event at the time of study discontinuation. If a patient has not had a dose reduction and is still on study drug, they will be censored at their last visit assessment date. if any. For the safety phase, subjects who do not enter the safety phase will be censored at time 0. If a patient discontinues study drug Time to dose interruption is defined as the time (weeks) from the date of the start of the respective phase to the time of first dose

interruption, if any. For the safety phase, subjects who do not enter the safety phase will be censored at time 0. If a patient discontinues study drug they will be counted as an event at the time of study discontinuation. If a patient has not had a dose interruption and is still on study drug, they will be censored at their last visit assessment date. [1] 95% Confidence Interval for Kaplan-Meier estimate.

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100.

Source: Listing 16.2.5.1

DATE OF EXTRACTION: XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for Safety Phase and Overall

Table 14.1.5.4 Distribution of Achieved Doses (Safety Analysis Set)

| Visit | Dose | S to 10 years<br>(N=XX) | II to I/ years<br>(N=XX) |
|---|---|---|---|
| Week 24 | 5 mg | XX (XX.X) | XX (XX.X) |
| | 10 mg | XX (XX.X) | XX (XX.X) |
| | 20 mg | XX (XX.X) | XX (XX.X) |
| | 30 mg | XX (XX.X) | XX (XX.X) |
| | 40 mg | XX (XX.X) | XX (XX.X) |
| | 60 mg | xx (xx.x) | XX (XX.X) |
| Week 56 | 5 mg | XX (XX.X) | XX (XX.X) |
| | 10 mg | XX (XX.X) | XX (XX.X) |
| | 20 mg | XX (XX.X) | XX (XX.X) |
| | 30 mg | XX (XX.X) | XX (XX.X) |
| | 40 mg | XX (XX.X) | XX (XX.X) |
| | 60 mg | xx (xx.x) | XX (XX.X) |
| Week 104 | 5 mg | XX (XX.X) | XX (XX.X) |
| | 10 mg | XX (XX.X) | XX (XX.X) |
| | 20 mg | XX (XX.X) | XX (XX.X) |
| | 30 mg | XX (XX.X) | XX (XX.X) |
| | 40 mg | XX (XX.X) | XX (XX.X) |
| | 60 mg | XX (XX.X) | XX (XX.X) |
| N= the number of subjects in the analysis set. $n=$ the Source: Listing 16.2.5.1 | We number of subjects meeting the criterion. (%) = $\ensuremath{\mathrm{n}}/\ensuremath{\mathrm{N}}^*100$ | iterion. (%) = $n/N*100$ . | |

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Add or remove dose categories as applicable.

Table 14.2.1.1 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks

(Full Analysis Set)

| | | | ( | |
|---|---|---|---|---|
| | | | Overall<br>(N=XX) | <b>⊤</b> |
| | | | Change | |
| | | Observed | from | % Change from |
| Visit | Statistics | value | baseline | baseline |
| ( ) | , | *** | | |
| Baseline | n | XX | | |
| | Mean | xx.x | | |
| | SD | XX.XX | | |
| | Minimum | ×× | | |
| | Median | XX.X | | |
| | Maximum | ×× | | |
| | 25th percentile | ×.×× | | |
| | 75th percentile | XX. | | |
| HAFICACT, MOON 24 | c | ** | >><br>>> | * |
| Analysis Study Week 24) | = | 7777 | ×7×7 | ~~~ |
| | Mean | ××.×× | XX.X | x.xx |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX |
| | Median | ××.×× | XX.X | XX.XX |
| | Maximum | ×× | XX | ×× |
| | 25th percentile | XX.X | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X |
| Efficacy Week 24 | и | XX | XX | XX |
| (Nominal Study Visit 10) | Mean | ×.×× | ×.×× | X.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX |
| | Median | XX.XX | XX.X | XX.XX |
| | Maximum | XX | XX | ×× |
| | 25th percentile | XX.X | XX.X | XX.X |
| | 75th percentile | ××.× | XX.X | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set. n = the number of subjects with a measurement.

[1] 95% confidence interval for mean percentage change.

[\*] Null hypothesis of 0% change. One-sample t-test or Wilcoxon Signed-Rank test.

#### Amryt Pharma study no: APH-19

## SQN Clinical study no: OCH19003

[\*\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [\*\*\*] Missing data has been imputed using Baseline Observation Carried Forward (BOCF).

[\*\*\*\*] Sensitivity analysis: Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect. An unstructured covariance will be used initially. The Akaike Information Criterion (AIC) used to assess model fit for covariance structures.

Percentage change from baseline is interpreted clinically as the greater the negative percentage change from baseline the greater the absolute clinical percentage change (i.e. percentage change of -48.5% is interpreted clinically as a 48.5% decrease from baseline). Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN: XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS 

Table 14.2.1.1 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Full Analysis Set)

| | | | Overall (N=XX) | all<br>(X) |
|---|---|---|---|---|
| | | Observed | Change<br>from | % Change from |
| Visit | Statistics | value | baseline | baseline |
| <pre>Efficacy Week 24 (LOCF)** (Analysis Study Week 24)</pre> | n | × | XX | XX |
| | Mean | ×.×× | x.xx | x.xx |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | XX | ×× |
| | Median | XX.X | XX.X | XX.XX |
| | Maximum | ×× | XX | ×× |
| | 25th percentile | XX.XX | XX.X | xx.xx |
| | 75th percentile | XX.X | xx.x | XX.X |
| <pre>Efficacy Week 24 (LOCF)** (Nominal Study Visit 10)</pre> | п | X | XX | ×× |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | XX | ×× |
| | Median | XX.X | XX.X | xx.xx |
| | Maximum | ×× | XX | ×× |
| | 25th percentile | XX.X | XX.X | XX.X |
| | 75th percentile | ×.× | ×.×. | xx |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set. n = the number of subjects with a measurement.

[1] 95% confidence interval for mean percentage change.

[\*] Null hypothesis of 0% change. One-sample t-test or Wilcoxon Signed-Rank test. [\*\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[\*\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [\*\*\*] Missing data has been imputed using Baseline Observation Carried Forward (BOCF).

[\*\*\*\*] Sensitivity analysis: Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect. An unstructured covariance will be used initially. The Akaike Information Criterion (AIC) used to assess model fit for Percentage change from baseline is interpreted clinically as the greater the negative percentage change from baseline the greater the absolute clinical percentage change (i.e. percentage change of -48.5% is interpreted clinically as a 48.5% decrease from baseline). covariance structures.

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXXX PROGRAM NAME: T XXX 01.SAS Source: Listing 16.2.8.1

Table 14.2.1.1 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Full Analysis Set)

| | | | Overal! (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| | | Observed | | % Change from |
| VISIC | Statistics | value | Daseline | Daseline |
| Efficacy Week 24 (BOCF) *** | ц | XX | XX | XX |
| (Alicalysts seady week 21) | Mean | x. xx | XX.X | X.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX |
| | Median | XX.XX | XX.X | XX.X |
| | Maximum | ×× | XX | XX |
| | 25th percentile | XX.XX | XX.X | xx.x |
| | 75th percentile | xx.x | XX.X | ХХ.Х |
| <pre>Efficacy Week 24 (BOCF)*** (Nominal Study Visit 10)</pre> | п | × | ×× | ×× |
| | Mean | XX.XX | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | XX | XX |
| | Median | xx.xx | XX.X | XX.X |
| | Maximum | ×× | XX | XX |
| | 25th percentile | XX.XX | XX.X | xx.x |
| | 75th percentile | ××.× | XX.X | ××.×× |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set. n = the number of subjects with a measurement. [1] 95% confidence interval for mean percentage change.

[\*] Null hypothesis of 0% change. One-sample t-test or Wilcoxon Signed-Rank test. [\*\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[\*\*\*] Missing data has been imputed using Baseline Observation Carried Forward (BOCF).

[\*\*\*\*] Sensitivity analysis: Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect. An unstructured covariance will be used initially. The Akaike Information Criterion (AIC) used to assess model fit for covariance structures.

Percentage change from baseline is interpreted clinically as the greater the negative percentage change from baseline the greater the absolute clinical percentage change (i.e. percentage change of -48.5% is interpreted clinically as a 48.5% decrease from baseline). Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS

Table 14.2.1.1 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Full Analysis Set)

| | | | Overall (N=XX) | 1.1<br>() |
|---|---|---|---|---|
| Visit | Statistics | Observed<br>value | Change<br>from<br>baseline | % Change from baseline |
| Primary Analysis<br>(Analysis Study Week 24) | Mean percentage change<br>95% Confidence Interval[1]<br>P-Value* | | | x.x<br>(x.xxx, x.xxx)<br>x.xxx |
| Sensitivity Analysis (Wilcoxon signed rank) (LOCF) | P-Value* | | | X.XXXX |
| Sensitivity Analysis (Nominal<br>Study Visit 10) | Mean percentage change<br>95% Confidence Interval[1]<br>P-Value* | | | XX.X<br>(X.XXXX, X.XXXX)<br>X.XXXX |
| Sensitivity Analysis (MMRM) **** | Mean percentage change<br>95% Confidence Interval[1]<br>P-Value* | | | XX.X<br>(X.XXXX, X.XXXX)<br>X.XXXX |
| Sensitivity Analysis (BOCF) *** | Mean percentage change<br>95% Confidence Interval[1]<br>P-Value* | | | XX.X<br>(X.XXXX, X.XXXX)<br>X.XXXX |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set. n = the number of subjects with a measurement. [1] 95% confidence interval for mean percentage change.

[\*] Null hypothesis of 0% change. One-sample t-test or Wilcoxon Signed-Rank test.

[\*\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[\*\*\*] Missing data has been imputed using Baseline Observation Carried Forward (BOCF). fixed effect. An unstructured covariance will be used initially. The Akaike Information Criterion (AIC) used to assess model fit for

Percentage change from baseline is interpreted clinically as the greater the negative percentage change from baseline the greater the absolute clinical percentage change (i.e. percentage change of -48.5% is interpreted clinically as a 48.5% decrease from baseline). Source: Listing 16.2.8.1 covariance structures.

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

# DocuSign Envelope ID: A18FEEF9-59CA-4D21-B668-F2E37C0A9EAE

# SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.1.2 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - per protocol set)

(Per Protocol Set)

Repeat of Table 14.2.1.1

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.1 (as applicable)


## Amryt Pharma study no: APH-19

# SQN Clinical study no: OCH19003

Table 14.2.1.3 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - completer analysis set) (Completers Analysis Set)

Repeat of Table 14.2.1.1

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.1 (as applicable)


Table 14.2.1.4 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups) (Full Analysis Set)

| | | | 5 to 10 years (N=XX) | ears | | 11 to 17 years (N=XX) | ears |
|---|---|---|---|---|---|---|---|
| | | | Change | | | Change | |
| Visit | Statistics | Observed value | from<br>baseline | % Change from baseline | Observed value | from<br>baseline | % Change from baseline |
| | | • | | | ; | | |
| Baseline | п | XX | | | ×× | | |
| | Mean | XX.XX | | | XX.XX | | |
| | SD | XX.XX | | | XX.XX | | |
| | Minimum | XX | | | XX | | |
| | Median | X.XX | | | XX.X | | |
| | Maximum | ×× | | | ×× | | |
| | 25th percentile | XX.XX | | | ×.×× | | |
| | 75th percentile | XX.X | | | x.xx | | |
| Efficacy Week 24<br>(Analysis Study Week 24) | и | XX | XX | XX | XX | XX | XX |
| | Mean | XX.X | x.xx | ××.× | ×.×× | x.xx | XX.X |
| | SD | XX.XX | XX.XX | ××.×× | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | ×× | XX |
| | Median | XX.XX | ××.× | XX.X | ×.×× | ××.× | XX.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 25th percentile | XX.X | x.xx | XX.XX | XX.X | x.xx | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Efficacy Week 24 | ជ | ×× | XX | XX | XX | XX | XX |
| (NOMILIAL SCACY VISIC 10) | Mean | ×·×× | ××× | ××× | ×·× | ××× | ×:× |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | XX.XX | XX.X | ××.× | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX | ×× |
| | 25th percentile | XX.X | x.xx | XX.XX | XX.X | xx.x | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set.

Analysis of Covariance (ANCOVA) model with age group as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX Date: 28JUN2024 Version: Final 5.0


Table 14.2.1.4 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups) (Full Analysis Set)

| | | | 5 to 10 years (N=XX) | ears | | 11 to 17 years (N=XX) | Vears |
|---|---|---|---|---|---|---|---|
| | | | Change | | | Change | |
| Visit | Statistics | Observed | from | % Change from baseline | Observed value | from | % Change from baseline |
| Efficacy Week 24 | r | XX | XX | XX | × | XX | ×× |
| (LOCE)<br>(Analvsis Study Week 24) | | | | | | | |
| 1 | Mean | ×.×× | x.x | XX.XX | XX.XX | xx.xx | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | XX | XX |
| | Median | ×.×× | xx.x | ××.× | XX.X | x.xx | XX.X |
| | Maximum | XX | ×× | ×× | XX | ×× | XX |
| | 25th percentile | XX.X | x.xx | XX.X | XX.XX | x.xx | XX.X |
| | 75th percentile | ××.× | x.xx | XX.X | x.xx | ××.× | XX.X |
| Efficacy Week 24 (LOCF) ** | и | XX | × | XX | XX | XX | XX |
| (Nominal Study Visit 10) | | | | | | | |
| | Mean | ××.×× | ××.× | XX.X | XX.XX | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | ×× | XX |
| | Median | XX.X | ××.× | xx.x | XX.X | XX.X | XX.X |
| | Maximum | ×× | ×× | ×× | XX | ×× | XX |
| | 25th percentile | XX.XX | ××.× | XX.X | XX.XX | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set.
Analysis of Covariance (ANCOVA) model with age group as a categorical fixed effect.
[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).
[1] Mean percentage change at week 24 from baseline
[2] 95% confidence interval for mean percentage change.
Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.1.4 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups) (Full Analysis Set)

| | | | 5 to 10 years (N=XX) | years<br>) | | 11 to 17 years (N=XX) | years |
|---|---|---|---|---|---|---|---|
| Visit | Statistics | Observed<br>value | Change<br>from<br>baseline | % Change from<br>baseline | Observed | Change<br>from<br>baseline | % Change from baseline |
| Analysis Study Week 24 | Mean percentage change [1] | | | x.xx | | | ×.×x |
| | 95% Confidence Interval[2] | | | (X.XXXX,<br>X.XXXX) | | | (X.XXXX,<br>X.XXXX) |
| Nominal Study Visit 10 | Mean percentage change [1] | | | XX.X. | | | XX.X |
| | 95% Confidence Interval[Z] | | | (X.XXXX,<br>X.XXXX) | | | (X.XXXX,<br>X.XXXX) |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set.
Analysis of Covariance (ANCOVA) model with age group as a categorical fixed effect.
[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).
[1] Mean percentage change at week 24 from baseline
[2] 95% confidence interval for mean percentage change.
Source: Listing 16.2.8.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXX

Table 14.2.1.5 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

(Full Analysis Set)

| | | Document | ed cardiova | Documented cardiovascular disease | No doc | cumented car | No documented cardiovascular |
|---|---|---|---|---|---|---|---|
| | | hi | history at screening | reening | diseas | se history a | disease history at screening |
| | | | (N=XX) | • | | (N=XX) | |
| | | | Change | ; | ; | Change | ; |
| Visit | Statistics | Observed | from | % Change from<br>baseline | Observed value | from | % Change from<br>baseline |
| ( | S | >> | | | > | | |
| Baseline | п | ΥΥ | | | ΥΥ | | |
| | Mean | ×.×. | | | XX.X | | |
| | SD | XX.XX | | | XX.XX | | |
| | Minimum | XX | | | XX | | |
| | Median | ×.×× | | | x.xx | | |
| | Maximum | XX | | | XX | | |
| | 25th percentile | ×.×× | | | XX.X | | |
| | 75th percentile | хх. х | | | XX.X | | |
| Efficacy Week 24<br>(Analysis Study Week 24) | п | ×× | XX | ×× | XX | ×× | XX |
| | Mean | ×.×× | xx.x | XX.X | XX.X | x.xx | XX.X |
| | SD | XX.XX | XX.XX | ××.×× | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | XX | XX |
| | Median | ×.×× | ××.× | XX.X | x.xx | ×.×× | XX.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 25th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | ××.×× | XX.X | XX.X | ×.×. | XX.X | XX.X |
| Efficacy Week 24 (Nominal Study Visit 10) | и | × | ×× | XX | XX | ×× | XX |
| , | Mean | XX.XX | ××.× | X.XX | XX.XX | XX.XX | X.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | ×× | XX |
| | Median | ×.×× | xx.x | XX.X | x.xx | ×.×× | XX.X |
| | Maximum | ×× | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | ×.×× | XX.X | XX.X | ××.× | XX.X | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set.

#### Amryt Pharma study no: APH-19

# SQN Clinical study no: OCH19003

Analysis of Covariance (ANCOVA) model with classification of documented cardiovascular disease history as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[1] Mean percentage change at week 24 from baseline

[2] 95% confidence interval for mean percentage change.

Source: Listing 16.2.8.1

DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX


Table 14.2.1.5 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

(Full Analysis Set)

| | | Document | nted cardiovascular chistory at screening | Documented cardiovascular disease | No doo | No documented cardi | No documented cardiovascular |
|---|---|---|---|---|---|---|---|
| | | TI . | (N=XX) | 6111110 | 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 | (N=XX) | |
| | | | Change | | | Change | |
| | | Observed | from | % Change from | Observed | from | % Change from |
| Visit | Statistics | value | baseline | baseline | value | baseline | baseline |
| <pre>Efficacy Week 24 (LOCF) **</pre> | и | XX | ×× | ×× | XX | ×× | XX |
| (Analysis Study Week 24) | | | | | | | |
| | Mean | XX.X | XX.X | XX.X | XX.XX | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | ×× | XX | ×× | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | x.xx | XX.X |
| | Maximum | XX | ×× | ×× | XX | ×× | XX |
| | 25th percentile | XX.X | XX.X | XX.X | XX.XX | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Efficacy Week 24 (LOCF) ** | и | XX | ×× | XX | X | ×× | XX |
| (Nominal Study Visit 10) | | | | | | | |
| | Mean | XX.X | XX.X | XX.X | XX.XX | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | XX | XX |
| | Median | XX.XX | XX.XX | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | ×× | ×× | XX | ×× | XX |
| | 25th percentile | XX.X | xx.x | XX.X | XX.XX | XX.X | XX.X |
| | 75th percentile | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study N = the number of subjects in the analysis set. treatment in the Efficacy Phase (Visit 4).

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION: XXXXXXXX

Analysis of Covariance (ANCOVA) model with classification of documented cardiovascular disease history as a categorical fixed effect. [\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

<sup>[1]</sup> Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

Table 14.2.1.5 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

(Full Analysis Set)

| | | Documented cardiovascular disease history at screening (N=XX) | No documented cardiovascular disease history at screening $(N=XX)$ |
|---|---|---|---|
| Visit | Statistics | Change Observed from % Change from value baseline baseline | Change Observed from % Change from value baseline baseline |
| Analysis Study Week 24 | Mean percentage change [1] | X.XX | XXX |
| | 95% Confidence Interval[2] | (X.XXXX, | (X.XXXX, |
| | | X.XXXX) | X.XXXX) |
| Nominal Study Visit 10 | Mean percentage change [1] | X.XX | X.XX |
| | 95% Confidence Interval[2] | (X.XXXX, | (X.XXXX, |
| | | X.XXXX) | X,XXXX) |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set. Analysis of Covariance (ANCOVA) model with classification of documented cardiovascular disease history as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX


Table 14.2.1.6 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis))

(Full Analysis Set)

| | | Establish | ed cardiova | Established cardiovascular disease | No esta | ablished car | No established cardiovascular |
|---|---|---|---|---|---|---|---|
| | | history | (defined as | history (defined as aortic valve | disease h | istory (def | disease history (defined as aortic |
| | | dise | disease and/or coronary | coronary | valve o | disease and/ | valve disease and/or coronary |
| | | atheros | scierosis) a<br>(N=XX) | atneroscierosis) at screening<br>(N=XX) | atneros | screrosis) a<br>(N=XX) | atneroscierosis) at screening<br>(N=XX) |
| | | | Change | | | Change | |
| | | Observed | from | % Change from | Observed | from | % Change from |
| Visit | Statistics | value | baseline | baseline | value | baseline | baseline |
| Baseline | п | ×× | | | × | | |
| | Mean | ×.×× | | | XX.X | | |
| | SD | XX.XX | | | XX.XX | | |
| | Minimum | XX | | | XX | | |
| | Median | XX.XX | | | XX.X | | |
| | Maximum | ×× | | | XX | | |
| | 25th percentile | ×.×× | | | XX.X | | |
| | 75th percentile | x.xx | | | XX.X | | |
| Efficacy Week 24 (Analysis Study Week 24) | ц | XX | ×× | XX | XX | ×× | ×× |
| | Mean | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | XX | XX | ×× | XX |
| | Median | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX.X |
| | Maximum | ×× | ×× | XX | XX | ×× | XX |
| | 25th percentile | ×.×× | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | хх.х | XX.X |
| Efficacy Week 24 (Nominal Study Visit 10) | u | × | XX | XX | X | ×× | XX |
| | Mean | XX.X | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | XX | XX | ×× | XX |
| | Median | XX.XX | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | Maximum | X | XX | XX | XX | XX | XX |
| | 25th percentile | ×.×× | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

#### Amryt Pharma study no: APH-19

## SQN Clinical study no: OCH19003

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set. Analysis of Covariance (ANCOVA) model with classification of established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis) as a categorical fixed effect.

- [\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).
  [1] Mean percentage change at week 24 from baseline
  [2] 95% confidence interval for mean percentage change.
  Source: Listing 16.2.8.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS


Table 14.2.1.6 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis))
(Full Analysis Set)

| | | Establish | ed cardiova | Established cardiovascular disease | No est | ablished ca: | No established cardiovascular |
|---|---|---|---|---|---|---|---|
| | | history | (defined as | history (defined as aortic valve | disease | history (def | disease history (defined as aortic |
| | | dise | disease and/or coronary | coronary | valve | disease and | valve disease and/or coronary |
| | | מכוועדס | (N=XX) | acheroscretosis) ac screening<br>(N=XX) | aciidic | (N=XX) | acheroscretosis) ac screening<br>(N=XX) |
| | | | Change | | | Change | |
| | | Observed | from | % Change from | Observed | from | % Change from |
| Visit | Statistics | value | baseline | baseline | value | baseline | baseline |
| Efficacy Week 24 | u | ×× | XX | XX | XX | XX | XX |
| (LOCF) ** | | | | | | | |
| (Analysis Study Week 24) | | | | | | | |
| | Mean | XX.X | xx.x | XX.X | XX.XX | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | ×× | XX |
| | Median | XX.XX | ××.× | XX.X | x.xx | ××.× | XX.X |
| | Maximum | XX | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.XX | ××.× | XX.X | XX.XX | x.xx | XX.X |
| | 75th percentile | XX.XX | xx.x | XX.X | XX.X | XX.X | XX.X |
| Efficacy Week 24<br>(LOCF)** | n | XX | ×× | XX | XX | XX | XX |
| (Nominal Study Visit 10) | | | | | | | |
| | Mean | XX.X | ××.× | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | ×× | ×× | XX |
| | Median | XX.XX | ××.× | xx.x | XX.XX | ××.× | xx.x |
| | Maximum | XX | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.X | xx.x | XX.X | XX.XX | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set.

Analysis of Covariance (ANCOVA) model with classification of established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis) as a categorical fixed effect.

<sup>[\*]</sup> Missing data has been imputed using Last Observation Carried Forward (LOCF).
[1] Mean percentage change at week 24 from baseline
[2] 95% confidence interval for mean percentage change.
Source: Listing 16.2.8.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF RUN:XXXXXXXX

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX


Table 14.2.1.6 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis))

(Full Analysis Set)

| | | Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis) at screening (N=XX) | vascular disease as aortic valve r coronary at screening X) | No est<br>disease l<br>valve<br>athero | ablished canistory (def<br>disease and<br>sclerosis) | No established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis) at screening (N=XX) |
|---|---|---|---|---|---|---|
| Visit | Statistics | Change<br>Observed from<br>value baseline | % Change from baseline | Observed | Change<br>from<br>baseline | % Change from baseline |
| Analysis Study Week 24 | Mean percentage change [1]<br>95% Confidence Interval[2] | | XX.X<br>(X.XXXX,<br>X.XXXX) | | | XX.X<br>(X.XXXX,<br>X.XXXX) |
| Nominal Study Visit 10 | Mean percentage change [1]<br>95% Confidence Interval[2] | | xx.x<br>(x.xxxx,<br>x.xxxx) | | | xx<br>(x.xxx,<br>x.xxx) |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

Analysis of Covariance (ANCOVA) model with classification of established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis) as a categorical fixed effect. N = the number of subjects in the analysis set.

- [\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS


Table 14.2.1.7 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

(Full Analysis Set)

| | | <b>H</b> | Had concomitant LLT | ant LLT | H | Had concomitant LLT | ant LLT |
|---|---|---|---|---|---|---|---|
| | | medicatic | ns/procedur | medications/procedures excluding LA | medicatio | ns/procedure | medications/procedures including LA |
| | | | (N=XX) | | | (N=XX) | |
| | | | Change | 4 | C | Change | |
| Visit | Statistics | Ubserved<br>value | rom<br>baseline | & change irom<br>baseline | observed<br>value | rom<br>baseline | s change irom<br>baseline |
| ۵<br>۵<br>د<br>د | ç | >> > | | | <b>&gt;</b> | | |
| 22 23 2 | : : | 4 9 4 4 9 4 9 4 9 4 9 4 9 4 9 9 9 9 9 9 | | | 4 7 4 4 7 | | |
| | Mean | XX.XX | | | XX.X | | |
| | SD | XX.XX | | | XX.XX | | |
| | Minimum | XX | | | XX | | |
| | Median | XX.XX | | | x.xx | | |
| | Maximum | XX | | | XX | | |
| | 25th percentile | XX.XX | | | XX.X | | |
| | 75th percentile | XX.X | | | XX.XX | | |
| Efficacy Week 24<br>(Analysis Study Week 24) | r. | XX | ×× | XX | XX | XX | XX |
| | Mean | XX.XX | xx.x | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | ××. | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | ×× | XX |
| | Median | XX.X | ××.× | XX.X | x.xx | ××.× | XX.X |
| | Maximum | XX | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.X | XX.X | XX.X | XX.XX | XX.X | XX.X |
| | 75th percentile | XX.X | | XX.X | ×.×. | XX.X | XX.X |
| Efficacy Week 24 (Nominal Study Visit 10) | и | × | ×× | XX | XX | ×× | XX |
| | Mean | ×.×× | ××.× | XX.X | XX.XX | ××.× | XX.X |
| | SD | XX.XX | XX.XX | ××. | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | XX.X | x.xx | XX.X | x.xx | x.xx | XX.X |
| | Maximum | XX | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.X | XX.X | XX.XX | XX.XX | XX.X | XX.X |
| | 75th percentile | ×.×. | ××.× | XX.X | xx.x | ××.× | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set.

#### Amryt Pharma study no: APH-19

## SQN Clinical study no: OCH19003

Analysis of Covariance (ANCOVA) model with classification of concomitant LLT medications/procedures as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[1] Mean percentage change at week 24 from baseline

[2] 95% confidence interval for mean percentage change.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


Table 14.2.1.7 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

(Full Analysis Set)

| Visit Stat: Efficacy Week 24 n (LOCE) ** (Analysis Study Week 24) SD | | medicatio | | | | | |
|---|---|---|---|---|---|---|---|
| Week 24) | | | ns/procedure<br>(N=XX) | medications/procedures excluding LA $(N=XX)$ | medicatio | ns/procedure<br>(N=XX) | medications/procedures including LA (N=XX) |
| Week 24) | | | Change | | | Change | |
| Week 24) | | Observed | from | % Change from | Observed | from | % Change from |
| Week 24) | Statistics | value | baseline | baseline | value | baseline | baseline |
| Week 24) | | × | ×× | XX | × | ×× | XX |
| Mean | | | | | | | |
| SD | נ | ×.×× | ××.× | XX.X | XX.X | ××.× | XX.XX |
| | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | rmum | XX | XX | XX | XX | ×× | XX |
| Median | Lan | ×.× | xx.x | ××.× | XX.XX | XX.X | XX.X |
| Maximum | Lmum | XX | XX | XX | XX | XX | XX |
| 25th | 25th percentile | XX.X | xx.x | XX.X | XX.XX | XX.X | XX.XX |
| 75th | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| <pre>Efficacy Week 24</pre> | | × | XX | XX | × | XX | XX |
| (Nominal Study Visit 10) | | | | | | | |
| Mean | נ | XX.X | xx.x | XX.XX | XX.XX | XX.X | XX.XX |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | rmum | XX | ×× | XX | XX | ×× | XX |
| Median | lan | XX.X | XX.X | xx.x | XX.XX | XX.X | XX.X |
| Maximum | rmum | XX | ×× | XX | XX | ×× | XX |
| 25th | 25th percentile | ×.×× | ××.× | XX.XX | XX.XX | XX.X | XX.XX |
| 75th | 75th percentile | XX.XX | XX.X | XX.X | XX.X | xx.x | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study N = the number of subjects in the analysis set. treatment in the Efficacy Phase (Visit 4).

DATE OF EXTRACTION:XXXXXXXX

Analysis of Covariance (ANCOVA) model with classification of concomitant LLT medications/procedures as a categorical fixed effect. [\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

<sup>[1]</sup> Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.1.7 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

(Full Analysis Set)

| | | Had concomitant LLT medications/procedures excluding LA (N=XX) | Had concomitant LLT medications/procedures including LA (N=XX) |
|---|---|---|---|
| Visit | Statistics | Change Observed from % Change from value baseline baseline | Change Observed from % Change from value baseline baseline |
| Analysis Study Week 24 | Mean percentage change [1] | XXX.X | XXX. |
| | 95% Confidence Interval[2] | (X.XXX,<br>X.XXXX) | (X.XXX,<br>X.XXXX) |
| Nominal Study Visit 10 | Mean percentage change [1] | ××××× | ××× |
| | 95% Confidence Interval[2] | (X.XXXX,<br>X.XXXX) | (X.XXXX,<br>X.XXXX) |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set.

Analysis of Covariance (ANCOVA) model with classification of concomitant LLT medications/procedures as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[1] Mean percentage change at week 24 from baseline

[2] 95% confidence interval for mean percentage change.

Source: Listing 16.2.8.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.1.8 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose interruptions)

(Full Analysis Set)

| | | N | No dose reductions | ctions | At le | At least one dose reduction | reduction |
|---|---|---|---|---|---|---|---|
| | | | (N=XX) | | | (N=XX) | |
| | | | Change | | | Change | |
| Visit | Statistics | Observed<br>value | from<br>baseline | % Change from<br>baseline | Observed<br>value | from<br>baseline | % Change from baseline |
| Baseline | п | XX | | | XX | | |
| | Mean | X.XX | | | XX.XX | | |
| | SD | XX.XX | | | XX.XX | | |
| | Minimum | XX | | | XX | | |
| | Median | XX.XX | | | XX.X | | |
| | Maximum | XX | | | XX | | |
| | 25th percentile | XX.XX | | | XX.XX | | |
| | 75th percentile | XX.XX | | | ×. ×. | | |
| Efficacy Week 24<br>(Analysis Study Week 24) | и | X | XX | XX | ×× | ×× | ×× |
| | Mean | XX.XX | ××.× | XX.X | XX.XX | x.xx | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | ×× | XX | ×× | XX |
| | Median | XX.XX | ××.× | ××.× | x.xx | x.xx | x.xx |
| | Maximum | XX | ×× | ×× | XX | ×× | XX |
| | 25th percentile | XX.XX | xx.x | XX.X | XX.XX | x.xx | XX.X |
| | 75th percentile | XX.X | хх.х | XX.X | XX.X | XX.X | XX.X |
| Efficacy Week 24 (Nominal Study Visit 10) | u | X | XX | XX | × | ×× | XX |
| | Mean | XX.X | ××.× | ××.× | ××.× | xx.x | xx.x |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | ×× | XX |
| | Median | XX.X | ××.× | ××.× | ××.× | xx.x | xx.x |
| | Maximum | XX | ×× | ×× | XX | ×× | XX |
| | 25th percentile | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | ××.× | ××.×× | XX.X | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. Analysis of Covariance (ANCOVA) model with classification of dose reduction as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


Table 14.2.1.8 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose (Full Analysis Set) interruptions)

| | | A | No dose reductions (N=XX) | ıctions | At le | ast one dose (N=XX) | At least one dose reduction $(N=XX)$ |
|---|---|---|---|---|---|---|---|
| | | | Change | | | Change | |
| Visit | Statistics | Observed | from | % Change from baseline | Observed | from | % Change from baseline |
| Efficacy Week 24 | n | XX | XX | XX | ×× | × | XX |
| (Analysis Study Week 24) | | | | | | | |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.XX | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | XX | XX | ×× | XX |
| | Median | XX.X | xx.x | XX.X | ×.×× | xx.x | x.xx |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 25th percentile | XX.X | XX.X | XX.X | XX.X | XX.XX | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| <pre>Efficacy Week 24 (LOCF) **</pre> | а | XX | XX | XX | X | × | XX |
| (Nominal Study Visit 10) | | | | | | | |
| | Mean | XX.X | xx.x | XX.X | XX.XX | XX.XX | XX.X |
| | SD | XX.XX | xx.xx | XX.XX | XX.XX | xx.xx | XX.XX |
| | Minimum | XX | ×× | XX | XX | ×× | XX |
| | Median | XX.X | xx.x | XX.X | XX.XX | XX.XX | XX.X |
| | Maximum | XX | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.X | XX.X | XX.X | XX.X | XX.XX | XX.X |
| | 75th percentile | ××× | ××× | × ×× | ××× | * ** | × ×× |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study N = the number of subjects in the analysis set. treatment in the Efficacy Phase (Visit 4).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS

Analysis of Covariance (ANCOVA) model with classification of dose reduction as a categorical fixed effect. [\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1
Table 14.2.1.8 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose interruptions)

(Full Analysis Set)

| | | NO | No dose reductions (N=XX) | uctions<br>) | At le | At least one dose reduction (N=XX) | e reduction |
|---|---|---|---|---|---|---|---|
| Visit | Statistics | Observed<br>value b | Change<br>from<br>baseline | % Change from<br>baseline | Observed<br>value | Change<br>from<br>baseline | % Change from baseline |
| Analysis Study Week 24 | Mean percentage change [1] | | | XX.X | | | ××.× |
| | 95% Confidence Interval[2] | | | (X.XXXX, | | | (X.XXXX, |
| | | | | X.XXXX) | | | X.XXXX) |
| Nominal Study Visit 10 | Mean percentage change [1] | | | XX.X | | | XX.X |
| | 95% Confidence Interval[2] | | | (X.XXXX, | | | (X.XXXX, |
| | | | | X.XXXX) | | | X.XXXX) |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study

treatment in the Efficacy Phase (Visit 4). N = the number of subjects in the analysis set.

Analysis of Covariance (ANCOVA) model with classification of dose reduction as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[1] Mean percentage change at week 24 from baseline

[2] 95% confidence interval for mean percentage change.

Source: Listing 16.2.8.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.1.9 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group)

(Full Analysis Set)

| | | ב ממא<br>ה ממא | AND FOY | מווטאט פטפ | رة<br>د ال | THACK MTD | mid not reach MTD for age groun |
|---|---|---|---|---|---|---|---|
| | | | (XX=N) | 7<br>5<br>1 | )<br>)<br>;<br>;<br>;<br>; | (XX=N) | 13<br>15 |
| | | | Change | | | Change | |
| Visit | Statistics | Observed | from | % Change from baseline | Observed value | from | % Change from baseline |
| Baseline | c | XX | | | XX | | |
| | Mean | XX.XX | | | XX.X | | |
| | SD | XX.XX | | | XX.XX | | |
| | Minimum | XX | | | XX | | |
| | Median | ×.×× | | | XX.X | | |
| | Maximum | XX | | | XX | | |
| | 25th percentile | ××.×× | | | XX.X | | |
| | 75th percentile | XX.X | | | ×.×. | | |
| Efficacy Week 24<br>(Analysis Study Week 24) | и | X | × | XX | XX | × | ×× |
| | Mean | ×.×× | XX.X | xx.x | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | ×× | ×× | ×× | XX |
| | Median | XX.XX | XX.X | xx.x | XX.X | XX.X | XX.X |
| | Maximum | ×× | ×× | ×× | ×× | ×× | XX |
| | 25th percentile | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | xx.x | x. x. | ××.× | XX.X |
| Efficacy Week 24 (Nominal Study Visit 10) | п | XX | × | ×× | XX | ×× | XX |
| | Mean | ×.×× | XX.X | xx.x | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | ×× | ×× | ×× | XX |
| | Median | ×.×× | ××.× | xx.x | XX.X | XX.X | XX.X |
| | Maximum | ×× | ×× | ×× | ×× | ×× | XX |
| | 25th percentile | XX.XX | XX.X | XX.X | XX.XX | XX.X | XX.X |
| | 75th percentile | ×. ×. | XX.X | XX.X | ×. ×. | x.xx | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. Analysis of Covariance (ANCOVA) model with classification of dose reduction as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS  Date: 28JUN2024 Version: Final 5.0

Table 14.2.1.9 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group) (Full Analysis Set)

| | | אממר | (N=XX) | Keached MTD ior age group<br>(N=XX) | Did not | reach MTD i<br>(N=XX) | Did not reach MTD for age group<br>(N=XX) |
|---|---|---|---|---|---|---|---|
| | | | Change | | | Change | |
| 4 7 7 7 14 | | Observed | from | % Change from | Observed | from | % Change from |
| VISIC | SCALLSCICS | value | Daserine | Daseline | value | Daseline | Daserine |
| Efficacy Week 24 | п | XX | XX | XX | XX | XX | XX |
| (LOCE) ** | | | | | | | |
| (Analysis Study Week 24) | ; | | | | | | |
| | Mean | ×.×. | XX.X | ××.× | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | ×× | ×× | ×× | XX |
| | Median | XX.X | ××.× | XX.X | XX.XX | ××.× | XX.X |
| | Maximum | XX | XX | ×× | XX | XX | XX |
| | 25th percentile | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| | 75th percentile | XX.X | xx.x | XX.X | XX.X | xx.x | XX.X |
| Efficacy Week 24 (LOCE) ** | ц | XX | × | XX | × | ×× | XX |
| (Nominal Study Visit 10) | | | | | | | |
| | Mean | XX.XX | XX.X | XX.X | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | ×× | ×× | ×× | XX |
| | Median | XX.X | XX.X | x.xx | XX.XX | XX.X | XX.X |
| | Maximum | XX | ×× | ×× | XX | ×× | XX |
| | 25th percentile | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| | 75th percentile | XX.X | XX.X | x.xx | XX.XX | XX.XX | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study N = the number of subjects in the analysis set. treatment in the Efficacy Phase (Visit 4).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Analysis of Covariance (ANCOVA) model with classification of dose reduction as a categorical fixed effect. [\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

Table 14.2.1.9 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group)

(Full Analysis Set)

| | | Reac | Reached MTD for age group $$({\rm N=XX})$$ | c age group<br>) | Did not | reach MTD (N=XX) | Did not reach MTD for age group $(N=XX)$ |
|---|---|---|---|---|---|---|---|
| Visit | Statistics | Observed<br>value | Change<br>from<br>baseline | % Change from baseline | Observed | Change<br>from<br>baseline | % Change from<br>baseline |
| Analysis Study Week 24 | Mean percentage change [1] | | | X.XX | | | XX.X |
| | 95% Confidence Interval[2] | | | (X.XXXX,<br>X.XXXX) | | | (X.XXXX,<br>X.XXXXX) |
| Nominal Study Visit 10 | Mean percentage change [1] 95% Confidence Interval[2] | | | , xxxx (x) | | | X.XX<br>(X.XXXXX) |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study

treatment in the Efficacy Phase (Visit 4). N = the number of subjects in the analysis set.

Analysis of Covariance (ANCOVA) model with classification of dose reduction as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).

[1] Mean percentage change at week 24 from baseline

[2] 95% confidence interval for mean percentage change.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION: XXXXXXXXX

Table 14.2.1.10 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex) (Full Analysis Set)

| | | | Male<br>(N=XX) | | | Female (N=XX) | |
|---|---|---|---|---|---|---|---|
| | | | Change | | | Change | |
| Visit | Statistics | Observed value | from<br>baseline | % Change from<br>baseline | Observed value | from<br>baseline | % Change from<br>baseline |
| Baseline | n | XX | | | × | | |
| | Mean | X. XX | | | X.XX | | |
| | SD | XX.XX | | | XX.XX | | |
| | Minimum | XX | | | XX | | |
| | Median | XX.XX | | | XX.X | | |
| | Maximum | XX | | | XX | | |
| | 25th percentile | XX.XX | | | XX.X | | |
| | 75th percentile | X.XX | | | x.xx | | |
| Efficacy Week 24<br>(Analysis Study Week 24) | ц | XX | XX | XX | X | ×× | XX |
| | Mean | XX.XX | XX.X | xx.xx | XX.XX | ××.× | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | ×× | XX |
| | Median | XX.XX | xx.x | XX.X | ×.×× | x.xx | XX.X |
| | Maximum | XX | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| | 75th percentile | XX.X | xx.x | XX.X | XX.X | XX.X | xx.x |
| Efficacy Week 24 (Nominal Study Visit 10) | и | × | XX | XX | × | XX | XX |
| 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 | Mean | XX.XX | ×.×× | ×.×× | ×.×× | ××. | XX. |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | XX.XX | xx.x | ××.× | XX.XX | x.xx | XX.X |
| | Maximum | XX | ×× | XX | ×× | ×× | XX |
| | 25th percentile | XX.X | xx.x | XX.X | XX.XX | xx.x | XX.X |
| | 75th percentile | XX.XX | XX.X | XX.X | XX.X | xx.x | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set.

Analysis of Covariance (ANCOVA) model with sex as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF).


[1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS 

Table 14.2.1.10 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex) (Full Analysis Set)

| | | | Male | | | Female | |
|---|---|---|---|---|---|---|---|
| | | | (N=XX) | | | (N=XX) | |
| | | | Change | | | Change | |
| | | Observed | from | % Change from | Observed | from | % Change from |
| Visit | Statistics | value | baseline | baseline | value | baseline | baseline |
| Efficacy Week 24 | и | X | XX | XX | XX | × | ×× |
| (LUCE)<br>(Analysis Study Week 24) | | | | | | | |
| | Mean | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | XX | XX | ×× | XX |
| | Median | ××.×× | XX.X | xx.x | XX.XX | XX.X | XX.X |
| | Maximum | ×× | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| <pre>Efficacy Week 24 (LOCF) **</pre> | а | ×× | × | X | XX | × | ×× |
| (Nominal Study Visit 10) | | | | | | | |
| | Mean | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | ×× | XX | ×× | XX |
| | Median | ××.× | ××.× | xx.x | XX.XX | XX.X | XX.X |
| | Maximum | ×× | ×× | XX | XX | ×× | XX |
| | 25th percentile | XX.XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | ×. ×. | ××.× | XX.X | xx.x | ×.× | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). Analysis of Covariance (ANCOVA) model with sex as a categorical fixed effect.

[1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.1.10 Lipid parameter: LDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex) (Full Analysis Set)

| | | | Male | | | Female | 0 6 |
|---|---|---|---|---|---|---|---|
| | | | (N=AA<br>Change | | | (N=AX)<br>Change | |
| Visit | Statistics | Observed value | from<br>baseline | % Change from<br>baseline | Observed value | from<br>baseline | % Change from baseline |
| Analysis Study Week 24 | Mean percentage change [1] | | | X.XX | | | X.XX |
| | 95% Confidence Interval[2] | | | (X.XXXX, | | | (X.XXXX, |
| | | | | X.XXXX) | | | X.XXXX) |
| Nominal Study Visit 10 | Mean percentage change [1] | | | XX.X | | | XX.XX |
| | 95% Confidence Interval[2] | | | (X.XXXX, | | | (X.XXXX, |
| | | | | X.XXXX) | | | X.XXXX) |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

N = the number of subjects in the analysis set. Analysis of Covariance (ANCOVA) model with sex as a categorical fixed effect.

[\*] Missing data has been imputed using Last Observation Carried Forward (LOCF). [1] Mean percentage change at week 24 from baseline [2] 95% confidence interval for mean percentage change. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN: XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

| f subjects achieving a reduction in f subjects achieving a reduction in f subjects achieving a reduction in any time from Week 8 of: statistics (N=XX) (N=XX) (N=XX) (N=XX) (N=XX) (X (XX.X) (X (XX.X | | | | | - | |
|---|---|---|---|---|---|---|
| n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) XX (XX.X) | | Statistics | | | to 17 years (N=XX) | Overall<br>(N=XX) |
| n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) XX (XX.X) | - | - | | | | |
| n (%) XX (XX.X) n (%) XX (XX.X) n (%) XX (XX.X) x (XX.X) XX (XX.X) x (XX.X) XX (XX.X) n (%) XX (XX.X) x (XX.X) XX (XX.X) x (XX.X) XX (XX.X) | Number of subjects achieving LDL-C at Week 24 of: | g a reduction in | | | | |
| n (%) XX (XX.X) n (%) XX (XX.X) x (XX.X) XX (XX.X) n (%) XX (XX.X) n (%) XX (XX.X) x (XX.X) XX (XX.X) | >15% | (%) u | XX (XX. | (× | XX (XX.X) | XX (XX.X) |
| n (%) XX (XX.X) n (%) XX (XX.X) n (%) XX (XX.X) x (XX.X) XX (XX.X) | >25% | $\overline{}$ | . XX (XX | (× | XX (XX.X) | XX (XX.X) |
| n (%) | >50% | _ | . XX (XX | (× | XX (XX.X) | XX (XX.X) |
| n (%) XX (XX.X) XX (XX.X) n (%) XX (XX.X) | Number of subjects achieving<br>LDL-C at any time from Week | g a reduction in<br>8 of: | | | | |
| n (%) XX (XX.X) XX (XX.X) | >15% | | .xx (xx | (× | xx (xx.x) | XX (XX.X) |
| | >25% | $\overline{}$ | . XX (XX | (X | XX (XX.X) | XX (XX.X) |
| n (%) XX (XX.X) XX (XX.X) XX XX | >50% | | .xx (xx | (X | XX (XX.X) | XX (XX.X) |
| | PROGRAM NAME: T_XXX_01.SAS | DATE OF RUN: XXXXXXXXX | TIME OF RUN: XX:XX:XX | DATE OF EXTRACTION: XXXXXXXXX | : XXXXXXXXX | |

#### SQN Clinical study no: OCH19003

Table 14.2.2.1 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Secondary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.1

PROGRAM NAME: T\_XXX\_01.SAS DATE

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX

Replace Primary Analysis with Secondary Analysis and exclude Sensitivity Analysis (MANRM) Footnotes as per Table 14.2.1.1 (as applicable) NOTES:


#### SQN Clinical study no: OCH19003

Table 14.2.2.2 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - per protocol set)

(Per Protocol Set)

Repeat of Table 14.2.1.2

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.2 (as applicable)

## SQN Clinical study no: OCH19003

Table 14.2.2.3 Lipid parameter: Non-HDL-C value (mg/dL) change from baseline at 24 weeks (Supplementary analysis - completer analysis set)

(Completers Analysis Set)

Repeat of Table 14.2.1.3

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.3 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.2.4 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups)

(Full Analysis Set)

Repeat of Table 14.2.1.4

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.4 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.2.5 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

(Full Analysis Set)

Repeat of Table 14.2.1.5

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.5 (as applicable)

### SQN Clinical study no: OCH19003

Table 14.2.2.6 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis))

(Full Analysis Set)

Repeat of Table 14.2.1.6

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.6 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.2.7 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

(Full Analysis Set)

Repeat of Table 14.2.1.7

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.7 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.2.8 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose interruptions)

(Full Analysis Set)

Repeat of Table 14.2.1.8

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.8 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.2.9 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group)

(Full Analysis Set)

Repeat of Table 14.2.1.9

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.9 (as applicable)

#### SQN Clinical study no: OCH19003

Table 14.2.2.10 Lipid parameter: Non-HDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex)

(Full Analysis Set)

Repeat of Table 14.2.1.10

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

PROGRAM NAME: T\_XXX\_01.SAS DATE OF RUN: XXXXXXXXX

NOTES: Footnotes as per Table 14.2.1.10 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.2.11 Lipid parameter: Non-HDL-C (mg/dL) Responder Analysis (Supplementary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.11

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.11 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.3.1 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Secondary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX

NOTES:

Footnotes as per Table 14.2.1.1 (as applicable)
Replace Primary Analysis with Secondary Analysis and exclude Sensitivity Analysis (MMRM)


#### SQN Clinical study no: OCH19003

Table 14.2.3.2 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - per protocol set)

(Per Protocol Set)

Repeat of Table 14.2.1.2

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.2 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.3.3 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - completer analysis set)

(Completers Analysis Set)

Repeat of Table 14.2.1.3

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.3 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.3.4 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups) (Full Analysis Set)

Repeat of Table 14.2.1.4

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.4 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.3.5 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

(Full Analysis Set)

Repeat of Table 14.2.1.5

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.5 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.3.6 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis))

(Full Analysis Set)

Repeat of Table 14.2.1.6

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.6 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.3.7 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

(Full Analysis Set)

Repeat of Table 14.2.1.7

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.7 (as applicable)

#### SQN Clinical study no: OCH19003

Table 14.2.3.8 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose interruptions) (Full Analysis Set)

Repeat of Table 14.2.1.8

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.8 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.3.9 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group)

(Full Analysis Set)

Repeat of Table 14.2.1.9

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.9 (as applicable)

# DocuSign Envelope ID: A18FEEF9-59CA-4D21-B668-F2E37C0A9EAE

#### SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.3.10 Lipid parameter: TC (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex) (Full Analysis Set)

Repeat of Table 14.2.1.10

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.10 (as applicable)

#### SQN Clinical study no: OCH19003

Table 14.2.3.11 Lipid parameter: TC (mg/dL) Responder Analysis (Supplementary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.11

PROGRAM NAME: T\_XXX\_01.SAS DATE OF RUN

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX

NOTES: Footnotes as per Table 14.2.1.11 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.4.1 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Secondary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.1

DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX

NOTES:

Footnotes as per Table 14.2.1.1 (as applicable)
Replace Primary Analysis with Secondary Analysis and exclude Sensitivity Analysis (MMRM)

#### SQN Clinical study no: OCH19003

Table 14.2.4.2 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - per protocol set) (Per Protocol Set)

Repeat of Table 14.2.1.2

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.2 (as applicable)

# SQN Clinical study no: OCH19003

Table 14.2.4.3 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - completer analysis set) (Completers Analysis Set)

Repeat of Table 14.2.1.3

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.3 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.4.4 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups) (Full Analysis Set)

Repeat of Table 14.2.1.4

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.4 (as applicable)


### SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.4.5 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

(Full Analysis Set)

Repeat of Table 14.2.1.5

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.5 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.4.6 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as acrtic valve disease and/or coronary atherosclerosis))

(Full Analysis Set)

Repeat of Table 14.2.1.6

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.6 (as applicable)


#### SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

(Full Analysis Set)

Table 14.2.4.7 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

Repeat of Table 14.2.1.7

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.7 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.4.8 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose interruptions)

Amryt Pharma study no: APH-19

(Full Analysis Set)

Repeat of Table 14.2.1.8

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.8 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.4.9 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group)

Amryt Pharma study no: APH-19

(Full Analysis Set)

Repeat of Table 14.2.1.9

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.9 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.4.10 Lipid parameter: VLDL-C (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex)

(Full Analysis Set)

Repeat of Table 14.2.1.10

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

PROGRAM NAME: T\_XXX\_01.SAS DATE OF RUN: XXXXXXXXX

NOTES: Footnotes as per Table 14.2.1.10 (as applicable)


SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.4.11 Lipid parameter: VLDL-C (mg/dL) Responder Analysis (Supplementary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.11

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.11 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.5.1 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Secondary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.1

DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX

NOTES:

Footnotes as per Table 14.2.1.1 (as applicable)
Replace Primary Analysis with Secondary Analysis and exclude Sensitivity Analysis (MMRM)

#### SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.5.2 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - per protocol set) (Per Protocol Set)

Repeat of Table 14.2.1.2

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.2 (as applicable)

#### SQN Clinical study no: OCH19003

Table 14.2.5.3 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - completer analysis set)

(Completers Analysis Set)

Repeat of Table 14.2.1.3

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.3 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.5.4 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups) (Full Analysis Set)

Amryt Pharma study no: APH-19

Repeat of Table 14.2.1.4

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.4 (as applicable)


### SQN Clinical study no: OCH19003

Table 14.2.5.5 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

Amryt Pharma study no: APH-19

(Full Analysis Set)

Repeat of Table 14.2.1.5

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.5 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.5.6 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis))

(Full Analysis Set)

Repeat of Table 14.2.1.6

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.6 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.5.7 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

(Full Analysis Set)

Repeat of Table 14.2.1.7

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.7 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.5.8 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose interruptions)

Amryt Pharma study no: APH-19

(Full Analysis Set)

Repeat of Table 14.2.1.8

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.8 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.5.9 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group)

(Full Analysis Set)

Repeat of Table 14.2.1.9

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.9 (as applicable)

#### SQN Clinical study no: OCH19003

Table 14.2.5.10 Lipid parameter: Apo B (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex)

(Full Analysis Set)

Repeat of Table 14.2.1.10

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

PROGRAM NAME: T\_XXX\_01.SAS DATE OF RUN: XXXXXXXXX

NOTES: Footnotes as per Table 14.2.1.10 (as applicable)

#### SQN Clinical study no: OCH19003

Table 14.2.5.11 Lipid parameter: Apo B (mg/dL) Responder Analysis (Supplementary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.11

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.11 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.6.1 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Secondary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX

NOTES:

Footnotes as per Table 14.2.1.1 (as applicable)
Replace Primary Analysis with Secondary Analysis and exclude Sensitivity Analysis (MMRM)


#### SQN Clinical study no: OCH19003

Table 14.2.6.2 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - per protocol set) (Per Protocol Set)

Repeat of Table 14.2.1.2

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.2 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.6.3 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Supplementary analysis - completer analysis set)

(Completers Analysis Set)

Repeat of Table 14.2.1.3

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.3 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.6.4 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups)

(Full Analysis Set)

Repeat of Table 14.2.1.4

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.4 (as applicable)

#### SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.6.5 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

(Full Analysis Set)

Repeat of Table 14.2.1.5

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.5 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.6.6 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis))

(Full Analysis Set)

Repeat of Table 14.2.1.6

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.6 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.6.7 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

(Full Analysis Set)

Repeat of Table 14.2.1.7

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.7 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.6.8 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose interruptions)

(Full Analysis Set)

Repeat of Table 14.2.1.8

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX

NOTES: Footnotes as per Table 14.2.1.8 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.6.9 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group)

(Full Analysis Set)

Repeat of Table 14.2.1.9

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.9 (as applicable)

#### SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.6.10 Lipid parameter: TG (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex) (Full Analysis Set)

Repeat of Table 14.2.1.10

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.10 (as applicable)

#### SQN Clinical study no: OCH19003

Table 14.2.6.11 Lipid parameter: TG (mg/dL) Responder Analysis (Supplementary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.11

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.11 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.7.1 Lipid parameter: Lp(a) and change from baseline at 24 weeks (Secondary analysis) (Full Analysis Set)

<Unit>

Repeat of Table 14.2.1.1 separately by unit

Results are based on local labs rather than central labs.

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES:

Footnotes as per Table 14.2.1.1 (as applicable)
Replace Primary Analysis with Secondary Analysis and exclude Sensitivity Analysis (MARM)
Add a combined p-value using Fisher's method.


#### SQN Clinical study no: OCH19003

Table 14.2.7.2 Lipid parameter: LP(a) and change from baseline at 24 weeks (Supplementary analysis - per protocol set) (Per Protocol Set)

Repeat of Table 14.2.1.2

Results are based on local labs rather than central labs.

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.2 (as applicable)


#### SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.7.3 Lipid parameter: LP(a) and change from baseline at 24 weeks (Supplementary analysis - completer analysis set) (Completers Analysis Set)

Repeat of Table 14.2.1.3

Results are based on local labs rather than central labs.

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.3 (as applicable)


### SQN Clinical study no: OCH19003

Table 14.2.7.4 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 1 - Age groups) (Full Analysis Set)

Repeat of Table 14.2.1.4

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.4 (as applicable)

#### SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.7.5 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 2 - Documented cardiovascular disease history)

(Full Analysis Set)

Repeat of Table 14.2.1.5

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.5 (as applicable)

#### SQN Clinical study no: OCH19003

Table 14.2.7.6 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 3 - Established cardiovascular disease history (defined as aortic valve disease and/or coronary atherosclerosis))

(Full Analysis Set)

Repeat of Table 14.2.1.6

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.6 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.2.7.7 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 4 - Concomitant LLT medications/procedures)

(Full Analysis Set)

Repeat of Table 14.2.1.7

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.7 (as applicable)


# DocuSign Envelope ID: A18FEEF9-59CA-4D21-B668-F2E37C0A9EAE

## SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.7.8 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 5 - Dose reductions / dose interruptions)

(Full Analysis Set)

Repeat of Table 14.2.1.8

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.8 (as applicable)

## SQN Clinical study no: OCH19003

Table 14.2.7.9 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 6 - Reached MTD for age group/ did not reach MTD for age group)

(Full Analysis Set)

Repeat of Table 14.2.1.9

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.9 (as applicable)


## SQN Clinical study no: OCH19003

Table 14.2.7.10 Lipid parameter: LP(a) (mg/dL) and change from baseline at 24 weeks (Subgroup analysis 7 - Sex)

(Full Analysis Set)

Repeat of Table 14.2.1.10

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

PROGRAM NAME: T\_XXX\_01.SAS DATE OF RUN: XXXXXXXXX

NOTES: Footnotes as per Table 14.2.1.10 (as applicable)


# DocuSign Envelope ID: A18FEEF9-59CA-4D21-B668-F2E37C0A9EAE

## SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.2.7.11 Lipid parameter: LP(a) (mg/dL) Responder Analysis (Supplementary analysis)

(Full Analysis Set)

Repeat of Table 14.2.1.11

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.2.1.11 (as applicable)


Table 14.2.8.1 Lipid parameter: LDL-C (mg/dL) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

| | | | 5 to 10 years (N=XX) | 10 years (N=XX) | | | 11 to 17 years (N=XX) | o 17 years<br>(N=XX) | | | Overall<br>(N=XX) | rall<br>XX) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Č | Change | %<br>Change | | - | Change | %<br>Change | | ( | Change | %<br>Change |
| | Statisti | | observe | rom<br>baselin | baselin | | Observe | baselin | rom<br>baselin | | Observe | rom<br>baselin | rrom<br>baselin |
| Visit | CS | Dose | value | Φ | Φ | Dose | value | Φ | Φ | Dose | value | Φ | Φ |
| Baselin | п | XX | × | | | XX | X | | | XX | XX | | |
| υ | Mean | XX.X | | | | XX.X | | | | XX.X | | | |
| | SD | XX.X | | | | XX.X | | | | XX.X | | | |
| | | × | | | | × | | | | × | | | |
| | Minimum | ×× | | | | ×× | | | | XX | | | |
| | Median | XX.X | | | | XX.XX | | | | XX.XX | | | |
| | Maximum | ×× | | | | ×× | | | | ×× | ×× | | |
| | 25th<br>percenti | xx.x | | | | XX.X | X.XX | | | ×.× | X. X | | |
| | 75th<br>Percenti | XX.X | ×.×× | | | × | ×. ×. | | | ×. ×. | ×. ×. | | |
| | Φ. | | | | | | | | | | | | |
| XXX | и | ×× | ×× | ×× | ×× | ×× | ×× | XX | XX | ×× | | XX | ×× |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.XX | XX.XX | XX.X | XX.XX | XX.XX | XX.X | XX.X | XX.XX |
| | SD | XX.X | XX.X | x.xx | ××.× | XX.XX | XX.X | XX.X | XX.X | XX.X | | XX.X | XX.X |
| | | × | × | × | × | × | × | × | × | × | | × | × |
| | Minimum | XX | ×× | ×× | ×× | XX | ×× | ×× | ×× | XX | | ×× | ×× |
| | Median | XX.X | XX.XX | XX.X | XX.X | XX.X | XX.X | ××.×× | XX.X | XX.XX | | XX.X | ××.× |
| | Maximum | ×× | × | × | ×× | ×× | ×× | × | ×× | ×× | | × | ×× |
| | 25th | xx.x | x.x. | x.xx | ××.× | XX.X | ××.× | ×.×× | ×.×× | XX.XX | | ×.×× | ×.×× |
| | percenti | | | | | | | | | | | | |
| | re<br>75th | × ×× | ><br>>> | × × × | > >> | × ×× | > >> | ><br>>> | > | × ×× | > > | × ×× | ><br>>> |
| | percenti | | 4<br>4<br>4<br>4<br>4<br>4<br>4 | 4 9 • | 4 9 • | 4<br>•<br>4<br>4<br>4<br>4 | 4 | 4<br>4<br>4<br>4<br>4<br>4<br>4<br>4 | 4 7 | 4<br>•<br>4<br>4<br>4<br>4 | 4 | 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 | |
| | Fe | | | | | | | | | | | | |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. n = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX


Table 14.2.8.1 Lipid parameter: LDL-C (mg/dL) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

| Statistic Statistic Change Chan | | | | 5 to $10 \text{ years}$ (N=XX) | 10 years<br>(N=XX) | | | 11 to 17 years $(N=XX)$ | o 17 years<br>(N=XX) | | | Overal<br>(N=XX) | verall<br>(N=XX) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Statistic Change | | • | | | | 0/0 | | | | 0/0 | | | | 0/0 |
| Statistic Dose Value e Dose From Goserve from Goserve from d Dose Value e Dose Value e Dose From Goserve from Goserve from Goserve from Goserve from Goserve G | | | | | Change | Change | | | Change | Change | | | Change | Change |
| Statistic d baselin d baselin baselin d baselin s Dose value e e bose value e e bose value e . | | | | Observe | from | from | | Observe | from | from | | Observe | from | from |
| Dose Value e e Dose Value e e Dose Value e | | Statistic | | ಶ | baselin | baselin | | で | baselin | baselin | | ಶ | baselin | baselin |
| n XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX XX </th <th>Visit</th> <th>w</th> <th>Dose</th> <th>value</th> <th>Φ</th> <th>Φ</th> <th>Dose</th> <th>value</th> <th>Φ</th> <th>Φ</th> <th>Dose</th> <th>value</th> <th>Φ</th> <th>Φ</th> | Visit | w | Dose | value | Φ | Φ | Dose | value | Φ | Φ | Dose | value | Φ | Φ |
| n xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx </td <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> <td></td> | | | | | | | | | | | | | | |
| n XXX XXX XXX XXXX XXXX XXXXX | Etc | | | | | | | | | | | | | |
| Mean XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X <th< td=""><td>·</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></th<> | · | | | | | | | | | | | | | |
| Mean XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X XX.X <th< td=""><td>EOT /<br/>Week</td><td>ď</td><td>XX</td><td>×</td><td>×</td><td>×</td><td>XX</td><td>X</td><td>×</td><td>×</td><td>×</td><td>XX</td><td>×</td><td>×</td></th<> | EOT /<br>Week | ď | XX | × | × | × | XX | X | × | × | × | XX | × | × |
| XXXX | 4<br>) | | XX.X | XX.X | XX.X | XX.X | X. XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| XX | | | xx.x | ×.×× | ××.× | x.xx | x.xx | xx.xx | xx.x | xx.x | ××.× | ×.×× | XX.X | XX.X |
| XX | | | × | × | × | × | × | × | × | × | × | × | × | × |
| xx xx.x xx.x xx.x xx.x xx.x xx.x xx.x | | | XX | ×× | ×× | ×× | XX | ×× | ×× | ×× | XX | XX | ×× | XX |
| xx | | | ×.×× | ×.×× | ×.×× | ×.×× | ×.×× | ×.×× | ×.× | ××.× | ××.× | ×.×× | ××.× | XX.X |
| 1 | | | XX | ×× | ×× | ×× | XX | ×× | ×× | ×× | XX | ×× | ×× | ×× |
| X:XX X:XX X:XX X:XX X:XX X:XX X:XX X:X | | | ×.×× | ×.×× | ×.×× | ×××× | ×.×× | ××.× | ××.× | ×××× | ×.×× | ××.×× | ×.×× | ×. ×× |
| X.XX X.XX X.XX X.XX X.XX X.XX X.XX X.X | | percentil | | | | | | | | | | | | |
| XXX XXXX | | Φ | | | | | | | | | | | | |
| | | 75th | ×××× | ×××× | ×.×× | ××× | ×.× | ××.× | ××.× | ××.× | ×.×× | ××. | ×.×× | ××× |
| | | percentil | | | | | | | | | | | | |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

### SQN Clinical study no: OCH19003

Table 14.2.8.2 Lipid parameter: Non-HDL-C (mg/dL) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

#### Repeat of Table 14.2.8.1

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


### SQN Clinical study no: OCH19003

Table 14.2.8.3 Lipid parameter: TC (mg/dL) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

#### Repeat of Table 14.2.8.1

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

### SQN Clinical study no: OCH19003

Table 14.2.8.4 Lipid parameter: VLDL-C (mg/dL) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

#### Repeat of Table 14.2.8.1

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


### SQN Clinical study no: OCH19003

Table 14.2.8.5 Lipid parameter: Apo B (g/L) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

#### Repeat of Table 14.2.8.1

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


### SQN Clinical study no: OCH19003

Table 14.2.8.6 Lipid parameter: TG (mg/dL) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

#### Repeat of Table 14.2.8.1

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


### SQN Clinical study no: OCH19003

Table 14.2.8.7 Lipid parameter: Lp(a) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

#### Repeat of Table 14.2.8.1

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS 

### SQN Clinical study no: OCH19003

Table 14.2.8.8 Lipid parameter: TC/HDL-C ratio and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

#### Repeat of Table 14.2.8.1

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.9.1 Lipid parameter: LDL-C (mg/dL) and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis) (Full Analysis Set)

| | | OO<br>(1) | Overall (N=XX) | | |
|---|---|---|---|---|---|
| Visit | Least Square Means Estimate[1] | Standard Error | 95% Confidence<br>Interval | | P-Value* |
| Week 4 | XX.XX | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 8 | XX.X | XX.XX | (X.XXXX, X.XXXXX) | XXXXX (XXX | XXX |
| Week 12 | XX.XX | XX.XX | (XXXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 16 | XX.XX | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 20 | ×.×× | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 24 | ×.×× | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 28 | XX.XX | XX.XX | (XXXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 32 | xx.x | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 36 | XX.X | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 40 | XX.X | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 44 | XX.XX | XX.XX | (XXXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 48 | XX.XX | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 52 | XX.XX | XX.XX | (XXXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 56 | XX.XX | XX.XX | (XXXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 68 | XX.XX | XX.XX | (X.XXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 80 | XX.XX | XX.XX | (XXXXX, X.XXXX) | XXXXX (XXX | XXX |
| Week 92 | XX.XX | XX.XX | (XXXXX, X.XXXX) | XXXXX (XXX | XXX |
| EOT / Week 104 | XX.X | XX.XX | (XXXXX, X.XXXX) | XXXXX (XXX | XXX |

N = the number of subjects in the analysis set.

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to assess model fit for covariance structures.

[1] Mean percentage change from baseline

[\*] Null hypothesis of 0% change.

Source: Listing 16.2.8.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS

### SQN Clinical study no: OCH19003

Table 14.2.9.2 Lipid parameter: Non-HDL-C (mg/dL) and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis) (Full Analysis Set)

Repeat of Table 14.2.9.

N = the number of subjects in the analysis set.

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect, baseline as a covariate and subject as a random effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to assess model fit for covariance structures.

[1] Mean percentage change from baseline

[\*] Null hypothesis of 0% change.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

### SQN Clinical study no: OCH19003

Table 14.2.9.3 Lipid parameter: TC (mmol/L) and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis) (Full Analysis Set)

Repeat of Table 14.2.9.1

N = the number of subjects in the analysis set.

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect, baseline as a covariate and subject as a random effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to assess model fit for covariance structures.

[1] Mean percentage change from baseline

[\*] Null hypothesis of 0% change.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


### SQN Clinical study no: OCH19003

Table 14.2.9.4 Lipid parameter: VLDL-C (mg/dL) and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis)

(Full Analysis Set)

#### Repeat of Table 14.2.9.1

N = the number of subjects in the analysis set.

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect, baseline as a covariate and subject as a random effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to assess model fit for covariance structures.

[1] Mean percentage change from baseline

[\*] Null hypothesis of 0% change.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

### SQN Clinical study no: OCH19003

Table 14.2.9.5 Lipid parameter: Apo B (g/L) and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis) (Full Analysis Set)

Repeat of Table 14.2.9.1

N = the number of subjects in the analysis set.

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect, baseline as a covariate and subject as a random effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to assess model fit for covariance structures.

[1] Mean percentage change from baseline

[\*] Null hypothesis of 0% change.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

### SQN Clinical study no: OCH19003

Table 14.2.9.6 Lipid parameter: TG (mg/dL) and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis)

(Full Analysis Set)

#### Repeat of Table 14.2.9.1

N = the number of subjects in the analysis set.

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect, baseline as a covariate and subject as a random effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to assess model fit for covariance structures.

[1] Mean percentage change from baseline

[\*] Null hypothesis of 0% change.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

#### SQN Clinical study no: OCH19003

Table 14.2.9.7 Lipid parameter: LP(a) and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis) (Full Analysis Set)

#### Repeat of Table 14.2.9.1

N = the number of subjects in the analysis set.

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect, baseline as a covariate and subject as a random effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to assess model fit for covariance structures.

[1] Mean percentage change from baseline

[\*] Null hypothesis of 0% change.

Results are based on local labs rather than central labs.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX


#### SQN Clinical study no: OCH19003

Table 14.2.9.8 Lipid parameter: TC/HDL-C ratio and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis)

(Full Analysis Set)

#### Repeat of Table 14.2.9.1

N = the number of subjects in the analysis set.

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect, baseline as a covariate and subject as a random effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to assess model fit for covariance structures.

[1] Mean percentage change from baseline

[\*] Null hypothesis of 0% change.

Results are based on local labs rather than central labs.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX


Table 14.2.10.1 Treated with standard Lipid Lowering Therapy (LLT) (including Lipoprotein Apheresis (LA) (Full Analysis Set)

| | Number | | LLT | | | LA | |
|---|---|---|---|---|---|---|---|
| Visit | attending visit (m) | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
| Baseline | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XXXX) XX | XX (XX.X) |
| Week 4 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) | XX (XX.X) |
| Week 8 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 12 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) | XX (XX.X) |
| Week 16 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 20 | XX | (XX.XX) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 24 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) | XX (XX.X) |
| Week 28 | XX | (XX.X) | (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 32 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) | XX (XX.X) |
| Week 36 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 40 | ×× | (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 44 | XX | (XX.X) | (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 48 | XX | (XX.XX) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 52 | XX | (XX.X) | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 56 | XX | (XX.XX) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 68 | XX | (XX.XX) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 80 | XX | (XX.X) | (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 92 | ×× | (XX.X) | (X.X.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| EOT / | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 104 | | | | | | | |

N = the number of subjects in the analysis set. m = the number of subjects attending visit. n = the number of subjects meeting the criterion. (%) = n/m\*100.


Source: Lising 16.2.4.6

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX

Table 14.2.10.2 Reduction in dose of standard Lipid Lowering Therapy (LLT) / Reduced need for Lipoprotein Apheresis (LA) compared to Week 24 (end of Efficacy Phase)

(Full Analysis Set)

| | | LLT | | | LA | |
|---|---|---|---|---|---|---|
| Visit | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
| Number of | ×× | XX | ×× | XX | XX | XX |
| patients treated | | | | | | |
| Week 24 (m) | | | | | | |
| Week 28 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High LDL-C | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Low LDL-C | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| : | | | | | | |
| Week 32 | (XXXX) XX | XX (XX.X) | XX (XX.X) | (XX.XX) | (XX.X) | XX (XX.X) |
| High LDL-C | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| LOW LDL-C | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

N = the number of subjects in the analysis set. m = number of patients treated with LLT (including LA) at Week 24. n = the number of subjects meeting the criterion. (%) = n/m\*100. Source: Lising 16.2.4.6

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.10.3 Discontinue standard Lipid Lowering Therapy (LLT) / Discontinue need for Lipoprotein Apheresis (LA) compared to Week 24 (end of Efficacy Phase)

(Full Analysis Set)

| | | LLT | | | LA | |
|---|---|---|---|---|---|---|
| ] | 5 to 10 years | 11 to 17 years | Overall | 5 to 10 years | 11 to 17 years | Overall |
| Visit | (N=XX) | (X=XX) | (N=XX) | (N=XX) | (X=XX) | (N=XX) |
| Number of | XX | XX | XX | XX | XX | XX |
| patients treated | | | | | | |
| with LLT / LA at | | | | | | |
| Week 24 (m) | | | | | | |
| Week 28 | XX (XX.X) | (XX.XX) XX | XX (XX.X) | XX (XX.X) | (X.XX) XX | XX (XX.X) |
| High LDL-C | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Low LDL-C | XX (XX.X) | (XX.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| : | | | | | | |
| Week 32 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High LDL-C | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Low LDL-C | XX (XX.X) | (X.XX) XX | XX (XX.X) | (X.XX) XX | XX (XX.X) | XX (XX.X) |
| : | | | | | | |
| : | | | | | | |

N = the number of subjects in the analysis set. m = number of patients treated with LLT (including LA) at Week 24. n = the number of subjects meeting the criterion. (%) = n/m\*100. Source: Lising 16.2.4.6

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS 

Table 14.2.10.4 Increase dose of standard Lipid Lowering Therapy (LLT) / Increased need for Lipoprotein Apheresis (LA) compared to Week 24 (end of Efficacy Phase)

(Full Analysis Set)

| | | LLT | | | LA | |
|---|---|---|---|---|---|---|
| Visit | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
| Number of | ×× | XX | XX | XX | ×× | X |
| patients treated | | | | | | |
| with LLT / LA at | | | | | | |
| Week 24 (m) | | | | | | |
| Week 28 | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) |
| High LDL-C | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) |
| LOW LDL-C | XX (XX.X) | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| : | | | | | | |
| Week 32 | (XXXXX) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) |
| High LDL-C | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) |
| Low LDL-C | XX (XX.X) | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| ÷ | | | | | | |
| : | | | | | | |

N = the number of subjects in the analysis set. m = number of patients treated with LLT (including LA) at Week 24. n = the number of subjects meeting the criterion. (%) = n/m\*100. Source: Lising 16.2.4.6


DATE OF RUN:XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.11.1 Recommended target of LDL-C of <135 mg/dL (i.e. 3.5 mmol/L) - EAS recommendation (Full Analysis Set)

| | -1 | | | |
|---|---|---|---|---|
| | Number | | | |
| | attending | 5 to 10 years | 11 to 17 years | Overall |
| Visit | visit (m) | (N=XX) | (N=XX) | (N=XX) |
| Baseline | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 4 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 8 | ×× | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 12 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 16 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 20 | ×× | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 24 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 28 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 32 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 36 | ×× | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 40 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 44 | ×× | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 48 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 52 | ×× | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 56 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 68 | ×× | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 80 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 92 | ×× | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| EOT / Week 104 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Anytime up to Week 24 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Anytime up to Week 104 | XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |

N = the number of subjects in the analysis set. m = number of patients attending the study visit, n = the number of subjects meeting the criterion. (%) = n/m\*100. Source: Listing 16.2.8.1


DATE OF EXTRACTION: XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.2.11.2 Recommended target of LDL-C of <135 mg/dL (i.e. 3.5 mmol/L) by age group and Lomitapide dose - EAS recommendation (Full Analysis Set)

Age Group = 5 to 10 years

| | Number | | | Lomitap | Lomitapide dose at time | time when LDL-C < 135 mg/dL | 5 mg/dL | |
|---|---|---|---|---|---|---|---|---|
| Visit | attending visit (m) | 2mg | 5mg | 10mg | 20mg | 30mg | 40mg | 60mg |
| - | | | | | | | | |
| Baseline | ×× | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| Week 4 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 8 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 12 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 16 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 20 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 24 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 28 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 32 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 36 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 40 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 44 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 48 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 52 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 56 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 68 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 80 | XX | XX | XX | XX | XX | XX | XX | XX |
| Week 92 | XX | ×× | ×× | XX | ×× | ×× | XX | XX |
| EOT / Week 104 | XX | XX | XX | XX | XX | XX | XX | XX |

m= number of patients attending the study visit. n= the number of subjects meeting the criterion. Source: Listing 16.2.8.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for Age Group = 11 to 17 years.

Only include applicable Lomitapide doses applicable for age group Additional doses may be added in to Lomitapide dose at time when LDL-C  $< 135 \, \mathrm{mg/dL}$  as appropriate

Table 14.2.11.3 Recommended targets of LDL-C - Exploratory endpoints

(Full Analysis Set)

| Visit | Number<br>attending<br>visit (m) | Recommended target | 5 to 10 years (N=XX) | 11 to 17 years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| Baseline | ×× | < 115 mg/dL<br>< 110 mg/dL | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | (X.XX) XX XX (XX.X) XX |
| Week 4 | ×× | <pre></pre> | | | (X. XX X |
| Week 8 | ×× | < 115 mg/dL<br>< 110 mg/dL | | | XX (XX.X)<br>XX (XX.X) |
| <br>EOT / Week 104 | XX | < 115 mg/dL<br>< 110 mg/dL | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Anytime up to Week 24 | ×× | < 115 mg/dL<br>< 110 mg/dL | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Anytime up to Week 104 | XX | < 115 mg/dL<br>< 110 mg/dL | XX (XX.X)<br>XX (XX.X) | (X. XX) XX | (X XX X |
| $N$ = the number of subjects in the analysis set. m criterion. (%) = $n/m \star 100$ . Source: Listing 16.2.8.1 | ts in the ana. | | ients attending the study | = number of patients attending the study visit. n = the number of subjects meeting the | subjects meeting the |

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for each visit

Table 14.2.11.4 Recommended targets of LDL-C by age group and Lomitapide dose - Exploratory endpoints

(Full Analysis Set)

Age Group = 5 to 10 years

| | Number | | | Lomit | Lomitapide dose at time when LDL-C recommended target was reached | time when LDL- | .C recommended | target was rea | ıched |
|---|---|---|---|---|---|---|---|---|---|
| Visit | attending<br>visit (m) | Recommended<br>target | 2mg | 5mg | 10mg | 20mg | 30mg | 4 0mg | 60mg |
| Baseline | XX | < 115 mg/dL | XX | ×× | XX | ×× | ×× | XX | × |
| | | < 110 mg/dL | XX | XX | ×× | XX | XX | XX | XX |
| Week 4 | XX | < 115 mg/dL | XX | XX | XX | XX | XX | XX | XX |
| | | < 110 mg/dL | XX | XX | XX | XX | XX | ×× | XX |
| Week 8 | XX | < 115 mg/dL | XX | XX | XX | XX | XX | XX | XX |
| | | < 110 mg/dL | XX | XX | XX | XX | XX | XX | XX |
| EOT / Week | XX | < 115 mg/dL | XX | XX | XX | XX | XX | XX | XX |
| H<br>D<br>Tr | | < 110 mg/dL | XX | ×× | XX | XX | XX | XX | ×× |

 $m=number\ of\ patients\ attending\ the\ study\ visit.$   $n=the\ number\ of\ subjects\ meeting\ the\ criterion.$  Source: Listing 16.2.8.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES:

Repeat for Age Group = 11 to 17 years. Only include applicable Lomitapide doses applicable for age group Additional doses may be added in to Lomitapide dose at time as appropriate


## SQN Clinical study no: OCH19003

Table 14.2.12.1 Lipid parameter: HDL-C (mg/dL) and change from Baseline to EOT / Week 104 by age group (Summary Measures) (Full Analysis Set)

#### Repeat of Table 14.2.8.1

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects with a measurement. Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


Table 14.2.12.2 Lipid parameter: HDL-C (mg/dL) and change from Baseline to EOT / Week 104 (Mixed Model Repeated Measures analysis) (Full Analysis Set)

#### Repeat of Table 14.2.9.1

Mixed Model Repeated Measures model with missing at random assumption. Model includes visit as a categorical fixed effect, baseline as a covariate and subject as a random effect. An unstructured covariance will be used initially. The Alkaike Information Criterion (AIC) used to N = the number of subjects in the analysis set. assess model fit for covariance structures. [1] Mean percentage change from baseline [\*] Null hypothesis of 0% change.

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS Date: 28JUN2024 Version: Final 5.0


Table 14.3.1.1 Summary of Treatment-Emergent Adverse Events

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| | 5 t | to 10 years (N=XX) | 11 | 11 to 17 years (N=XX) | | Overall (N=XX) |
|---|---|---|---|---|---|---|
| | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects (%) |
| Total number of TEAEs | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Total number of Non-TEAEs | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Serious TEAEs | × | (X.X.X) | XX | XX (XX.X) | × | (XX.XX) |
| Serious Related TEAEs [3] | × | (X.XX) XX | XX | (XX.X) | × | (XX.XX) |
| TEAEs leading to study discontinuation | × | (X.XX) XX | XX | (XX.X) | × | (XX.XX) |
| Serious TEAEs leading to study discontinuation | × | (X.XX) XX | XX | (XX.X) | × | (XX.XX) |
| Related TEAEs leading to study discontinuation [3] | ×× | (X.X.X) | XX | (X.XX) XX | ×× | (XX.X) |
| Serious Related TEAEs leading to study discontinuation [3] | XX | (X.X.) XX | XX | (X.XX) XX | ×× | (XX.X) |
| TEAEs leading to death | XX | (XX.X) | XX | (XX.X) | × | (XX.X) |
| Adverse Events of Special Interest (AESI) | ×× | (XX.X) | XX | (XX.X) | × | (XX.X) |
| AESI leading to study discontinuation | ×× | (XX.X) | XX | (XX.X) | × | (XX.X) |
| Study treatment-related AESI | ×× | (XXXX) XX | XX | (XXXX) XX | × | (XX.X) |
| NTEAEs leading to death | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |

Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug. [1] If a subject experienced more than one TEAE, the subject is counted once at the most severe or most related event. [2] Unrelated adverse events are those classified as having a non-reasonable causal relationship to the study treatment. [3] Related adverse events are those classified as having a reasonable causal relationship to the study treatment. N = the number of subjects in the analysis set. (%) = Subjects/N\*100. \*Major Adverse Cardiac Events are defined by the clinical team Source: Listing 16.2.7.1 and Listing 16.2.7.2

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.1.1 Summary of Treatment-Emergent Adverse Events

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| | | to 10 years (N=XX) | □□ | 11 to 17 years $(N=XX)$ | | Overall (N=XX) |
|---|---|---|---|---|---|---|
| | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects (%) |
| Major Adverse Cardiac Events (MACE)* | XX | (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| Severity [1] | 444 | | *** | | *** | |
| MILG | ×× | | XX | _ | ×× | |
| Moderate | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Severe | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| Life Threatening | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Death | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Relationship to study treatment [1] | | | | | | |
| Related [3] | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Unrelated [2] | XX | XX (XX.X) | ×× | XX (XX.X) | XX | XX (XX.X) |
| Action taken with study treatment | | | | | | |
| Dose Decreased | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Dose not Changed | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| Drug Withdrawn | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Not Applicable | X | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Unknown | | | | | | |
| () サンプラン | | | | | | |

Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug. [1] If a subject experienced more than one TEAE, the subject is counted once at the most severe or most related event. [2] Unrelated adverse events are those classified as having a non-reasonable causal relationship to the study treatment. [3] Related adverse events are those classified as having a reasonable causal relationship to the study treatment.

DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

N = the number of subjects in the analysis set. (%) = Subjects/N\*100. \*Major Adverse Cardiac Events are defined by the clinical team Source: Listing 16.2.7.1 and Listing 16.2.7.2

Table 14.3.1.2 Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| Svstem ordan class | 5 + | 5 to 10 years (N=XX) | 11 | 11 to 17 years $(N=XX)$ | | Overall (N=XX) |
|---|---|---|---|---|---|---|
| Preferred term | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects (%) |
| Total number of TEAEs | XX | XX (XX.X) | XX | (XX.X) | XX | XX (XX.X) |
| System organ class 1 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 1 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 2 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 3 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 4 | XX | XX (XX.X) | ×× | XX (XX.X) | XX | (XX.X) |
| System organ class 2 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 1 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 2 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 3 | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 4 | ×× | XX (XX.X) | ×× | XX (XX.X) | XX | (XX,XX) |

(PT).

Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug. If a subject experienced more than one TEAE, the subject is counted once for each system organ class (SOC) and once for each preferred term

SOCs are ordered in decreasing frequency of the total number of subjects with TEAEs reported in each SOC and PTs are ordered within a SOC in decreasing frequency of the total number of subjects with each TEAE.

Adverse events were coded using the MedDRA Dictionary, version xx.x. N = the number of subjects in the analysis set. (%) = Subjects/N\*100. Source: Listing 16.2.7.1 and Listing 16.2.7.2

PROGRAM NAME: T XXX 01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX
#### SQN Clinical study no: OCH19003

Table 14.3.1.3 Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Class and Preferred Term

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

Repeat of Table 14.3.1.2

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.3.1.2 (as applicable)


Table 14.3.1.4 Summary of Treatment-Emergent Adverse Events by MedDRA Preferred Term

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| | r. | 5 to 10 years (N=XX) | 11 | 11 to 17 years (N=XX) | | Overall (N=XX) |
|---|---|---|---|---|---|---|
| Preferred term | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects (%) |
| Total number of TEAEs | XX | XX (XX.X) | × | (XX.X) | XX | XX (XX.X) |
| Preferred term 1 | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 2 | ×× | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 3 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 4 | ×× | XX (XX,X) | ×× | (XXX,X) | XX | (XX,XX) |

Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug. If a subject experienced more than one TEAE, the subject is counted once for each preferred term (PT). PTs are ordered in decreasing frequency of subject incidence.

Adverse events were coded using the MedDRA Dictionary, version xx.x. N = the number of subjects in the analysis set. (%) = Subjects/N\*100. Source: Listing 16.2.7.1

PROGRAM NAME: T XXX 01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX 

# DocuSign Envelope ID: A18FEEF9-59CA-4D21-B668-F2E37C0A9EAE

#### SQN Clinical study no: OCH19003

Table 14.3.1.5 Summary of Serious Adverse Events (SAEs) by MedDRA Preferred Term

Amryt Pharma study no: APH-19

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

Repeat of Table 14.3.1.4

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.3.1.4 (as applicable)


Table 14.3.1.6 Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class, Preferred Term and Severity

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| System ordan class | | N | to 10 years (N=XX) | 11 | to 17 years (N=XX) | | Overall (N=XX) | |
|---|---|---|---|---|---|---|---|---|
| Preferred term | Severity | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects | (%) |
| Total number of TEAEs | Overall | XX | XX (XX.X) | × | XX (XX.X) | ×× | (XXXX) | ŝ |
| | Mild | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.XX) | (X |
| | Moderate | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X | (× |
| | Severe | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X | × |
| | Life-threatening | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.XX) | (X |
| | Death | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) | (× |
| System organ class 1 | Overall | XX | XX (XX.X) | ×× | XX (XX.X) | X | XX (XX.X) | (X |
| | Mild | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.XX) | × |
| | Moderate | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X | × |
| | Severe | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X | × |
| | Life-threatening | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) | × |
| | Death | XX | XX (XX.X) | ×× | XX (XX.X) | × | XX (XX.X) | $\widehat{\times}$ |
| Preferred term 1 | Overall | XX | XX (XX.X) | XX | XX (XX.X) | ×× | (XXXX) XX | (× |
| | Mild | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.XX) | × |
| | Moderate | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) | × |
| | Severe | XX | XX (XX.X) | ×× | XX (XX.X) | XX | XX (XX.X) | (X |
| | Life-threatening | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) | × |
| | Death | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | (X.XX) XX | × |

Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug. If a subject experienced more than one TEAE, the subject is counted once for each system organ class (SOC) and once for each preferred term (PT) at the most severe.

SOCs are ordered in decreasing frequency of the total number of subjects with TEAEs reported in each SOC and PTs are ordered within a SOC in decreasing frequency of the total number of subjects with each TEAE.

Adverse events were coded using the MedDRA Dictionary, version xx.x. N = the number of subjects in the analysis set. (%) = Subjects/N\*100. Source: Listing 16.2.7.1

DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX

DATE OF EXTRACTION:XXXXXXXX

#### SQN Clinical study no: OCH19003

Table 14.3.1.7 Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Class, Preferred Term and Severity

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

Repeat of Table 14.3.1.6

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.3.1.6 (as applicable)

Table 14.3.1.8 Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class, Preferred Term and Relationship to Study Treatment

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| System ordan class | Relationship to | 5 | 5 to 10 years (N=XX) | 11 | 11 to 17 years (N=XX) | | Overall (N=XX) |
|---|---|---|---|---|---|---|---|
| Preferred term | study treatment | Events | Events Subjects (%) | Events | Subjects (%) | Events | Events Subjects (%) |
| Total number of TEAEs | Overall | ×× | XX (XX.X) | ×× | (XX.X) | XX | XX (XX.X) |
| | Unrelated [1] | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| | Related [2] | ×× | XX (XX.X) | × | (XX.X) | × | XX (XX.X) |
| System organ class 1 | Overall | ×× | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| | Unrelated [1] | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| | Related [2] | ×× | XX (XX.X) | ×× | (XX.X) | ×× | XX (XX.X) |
| Preferred term 1 | Overall<br>Etc | XX | XX (XX.X) | XX | (XX.X) | XX | XX (XX.X) |
| E | | | | | | | |

If a subject experienced more than one TEAE, the subject is counted once for each system organ class (SOC) and once for each preferred term Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug. (PT) using the most related event.

SOCs are ordered in decreasing frequency of the total number of subjects with TEAEs reported in each SOC and PTs are ordered within a SOC in decreasing frequency of the total number of subjects with each TEAE.

[1] Unrelated adverse events are those classified as having no reasonable causal relationship to the study treatment. [2] Related adverse events are those classified as having a reasonable causal relationship to the study treatment. Adverse events were coded using the MedDRA Dictionary, version xx.x.

N = the number of subjects in the analysis set. (%) = Subjects/N\*100.

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Source: Listing 16.2.7.1

Table 14.3.1.9 Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Class, Preferred Term and Relationship to Study Treatment

(Safety Analysis Set)

Amryt Pharma study no: APH-19

Overall / Efficacy Phase / Safety Phase / Follow-up

Repeat of Table 14.3.1.8

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.3.1.8 (as applicable)


Table 14.3.1.10 Summary of Adverse Events of Special Interest (AESI) by AESI Category, MedDRA System Organ Class and Preferred Term

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| System ordan class | 5 | to 10 years (N=XX) | 11 | 11 to 17 years $(N=XX)$ | | Overall (N=XX) |
|---|---|---|---|---|---|---|
| Preferred term | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects (%) |
| Total number of AESI | XX | (XX.X) | XX | (X.XX) XX | XX | XX (XX.X) |
| AESI category 1 | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| System organ class 1 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 1 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 2 | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 3 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 4 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| System organ class 2 | XX | XX (XX.X) | ×× | XX (XX.X) | XX | (XX.X) |
| Preferred term 1 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 2 | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 3 | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 4 | × | (XX,X) | XX | (X, XX) XX | ×× | (X X X X X X X X X X X X X X X X X X X |

abnormalities, gastrointestinal effects and major congenital abnormality AEs. If a subject experienced more than one TEAE, the subject is counted once for each system organ class (SOC) and once for each preferred term Adverse events of special interest (AESI) are defined as hepatic, small bowel/intestinal, pancreatic and colorectal tumours, hepatic

SOCs are ordered in decreasing frequency of the total number of subjects with TEAEs reported in each SOC and PTs are ordered within a SOC in decreasing frequency of the total number of subjects with each TEAE.

Adverse events were coded using the MedDRA Dictionary, version xx.x. N = the number of subjects in the analysis set. (%) = Subjects/N\*100.

Source: Listing 16.2.7.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.1.11 Summary of Gastrointestinal (GI) Adverse Events by MedDRA System Organ Class and Preferred Term

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| System ordan class | 5 + | 5 to 10 years (N=XX) | 11 | 11 to 17 years $(N=XX)$ | | Overall (N=XX) |
|---|---|---|---|---|---|---|
| Preferred term | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects (%) |
| Total number of GI Adverse Events | XX | (XX.X) | XX | (X.XX) XX | × | XX (XX.X) |
| System organ class l | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 1 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 2 | ×× | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 3 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 4 | XX | XX (XX.X) | XX | XX (XX.X) | × | XX (XX.X) |
| System organ class 2 | ×× | XX (XX.X) | XX | XX (XX.X) | × | XX (XX.X) |
| Preferred term 1 | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 2 | ×× | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 3 | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 4 | ×× | (XXX, XX) | ×× | (XX.X) | X | (XXXXX) |

τ + If a subject experienced more than one TEAE, the subject is counted once for each system organ class (SOC) and once for each preferred term (PT).

SOCs are ordered in decreasing frequency of the total number of subjects with TEAEs reported in each SOC and PTs are ordered within a SOC in decreasing frequency of the total number of subjects with each TEAE.

Adverse events were coded using the MedDRA Dictionary, version xx.x. N = the number of subjects in the analysis set. (%) = Subjects/N\*1000.

Source: Listing 16.2.7.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.1.12 Summary of Most Frequent Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| System ordan class | 5 t | 5 to 10 years (N=XX) | 11 | 11 to 17 years (N=XX) | | Overall (N=XX) |
|---|---|---|---|---|---|---|
| Preferred term | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects (%) |
| Total number of TEAEs | XX | (XX.X) | × | (X.XX) XX | ×× | XX (XX.X) |
| System organ class 1 | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 1 | ×× | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 2 | ×× | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 3 | ×× | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 4 | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| System organ class 2 | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 1 | ×× | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| Preferred term 2 | ×× | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 3 | ×× | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| Preferred term 4 | ×× | XX (XX,X) | × | (XXX,X) | ×× | (XXXXX) |

Etc.

Only TEAEs that occurred in at least 2 subjects are presented.

Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug. If a subject experienced more than one TEAE, the subject is counted once for each system organ class (SOC) and once for each preferred term

SOCs are ordered in decreasing frequency of the total number of subjects with TEAEs reported in each SOC and PTs are ordered within a SOC in decreasing frequency of the total number of subjects with each TEAE.

Adverse events were coded using the MedDRA Dictionary, version xx.x. N = the number of subjects in the analysis set. (%) = Subjects/N\*100.

Source: Listing 16.2.7.1 and Listing 16.2.7.2

PROGRAM NAME: T\_XXX\_01.SAS DATE OF RUN: XXXXXXXXXX TIME OF RUN: XX:XX:XX

DATE OF EXTRACTION: XXXXXXXXX

NOTES: Present only TEAEs that occured in at least 2 subjects.

Table 14.3.1.13 Time to First Gastrointestinal Treatment-Emergent Adverse Events (Safety Analysis Set)

| Statistics | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|
| Number of subjects with a gastrointestinal TEAE, n (%) | (X.XX) XX | (XX.X) | (X.X) XX |
| Number of subjects censored, n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Kaplan-Meier estimates of time to first gastrointestinal TEAE (days) [1] | | | |
| 25tn percentile<br>95% CI [3] | XX.XX<br>(XX.XX, XX.XX) | XX.X<br>(XX.XX, XX.XX) | XX.X<br>(XX.XX, XX.XX) |
| Median | XX.X | XX.X | XX.X |
| 95% CI [3] | (XX.XX, XX.XX) | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| 75th percentile | XX.XX | XX.XX | XX.XX |
| 95% CI [3] | (XX.XX, XX.XX) | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| Kaplan-Meier estimates of duration of | | | |
| gastrointestinal TEAE (days) [2] | | | |
| 25th percentile | XX.X | XX.X | XX.X |
| 95% CI [3] | (XX.XX, XX.XX) | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| Median | XX.XX | XX.XX | XX.XX |
| 95% CI [3] | (XX.XX, XX.XX) | (XX.XX, XX.XX) | (XX.XX, XX.XX) |
| 75th percentile | XX.XX | XX.XX | XX.XX |
| 95% CI [3] | (XX.XX, XX.XX) | (XX.XX, XX.XX) | (XX.XX, XX.XX) |

<sup>[1]</sup> Time to first gastrointestinal TEAE is defined as the time (days) from the first dose to the time of first gastrointestinal TEAE, if any. [2] Duration is derived as: Date of resolution of the TEAE - Date of start of TEAE. Subjects with an ongoing TEAE will be censored at their last assessment date.

<sup>[3] 95%</sup> Confidence Interval for Kaplan-Meier estimate. N = the number of subjects meeting the criterion.

<sup>(%) =</sup> n/N\*100. Source: Listing 16.2.7.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS

# DocuSign Envelope ID: A18FEEF9-59CA-4D21-B668-F2E37C0A9EAE

SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Table 14.3.1.14 Time to First Hepatic Treatment-Emergent Adverse Events

(Safety Analysis Set)

Repeat of Table 14.3.1.13

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Footnotes as per Table 14.3.1.13 (as applicable)


Table 14.3.1.15 Summary of Treatment-Emergent Adverse Events, by Sex

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

Repeat of Table 14.3.1.1 by sex

Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug.

[1] If a subject experienced more than one TEAE, the subject is counted once at the most severe or most related event. [2] Unrelated adverse events are those classified as having a non-reasonable causal relationship to the study treatment. [3] Related adverse events are those classified as having a reasonable causal relationship to the study treatment.

N = the number of subjects in the analysis set. (%) = Subjects/N\*100.

\*Major Adverse Cardiac Events are defined by the clinical team Source: Listing 16.2.7.1 and Listing 16.2.7.2

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN: XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat of Table 14.3.1.1 by sex (Male, Female) instead of age group


#### SQN Clinical study no: OCH19003

Table 14.3.1.16 Summary of Adverse Events of Special Interest (AESI) by AESI Category, MedDRA System Organ Class and Preferred Term, by Sex

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

### Repeat of Table 14.3.1.10 by sex

abnormalities, gastrointestinal effects and major congenital abnormality AEs. If a subject experienced more than one TEAE, the subject is counted once for each system organ class (SOC) and once for each preferred term Adverse events of special interest (AESI) are defined as hepatic, small bowel/intestinal, pancreatic and colorectal tumours, hepatic

SOCs are ordered in decreasing frequency of the total number of subjects with TEAEs reported in each SOC and PTs are ordered within a SOC in decreasing frequency of the total number of subjects with each TEAE. (PT).

Adverse events were coded using the MedDRA Dictionary, version xx.x. N = the number of subjects in the analysis set. (%) = Subjects/N\*100.

Source: Listing 16.2.7.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat of Table 14.3.1.10 by sex (Male, Female) instead of age group


Table 14.3.1.17 Summary of Elevation in Serum Transaminases Related Treatment-Emergent Adverse Events by MedDRA System Organ Class and

Preferred Term, by Country

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| | | 5 t | 5 to 10 years | 11 t | 11 to 17 years | | Overall |
|---|---|---|---|---|---|---|---|
| System organ class | Country | | (N=XX) | | (N=XX) | | (N=XX) |
| Preferred term | | Events | Subjects (%) | Events | Subjects (%) | Events | Subjects (%) |
| Total number of TEAEs | Overall | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| | Germany | XX | XX (XX.X) | XX | XX (XX.X) | XX | XX (XX.X) |
| | Spain | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| | : | | | | | | |
| System organ class 1 | Overall | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| | Germany | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| | Spain | XX | XX (XX.X) | ×× | XX (XX.X) | × | XX (XX.X) |
| | : | | | | | | |
| Preferred term 1 | Overall | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| | Germany | XX | XX (XX.X) | XX | XX (XX.X) | ×× | XX (XX.X) |
| | Spain | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| | : | | | | | | |
| Preferred term 2 | Overall | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| | Germany | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| | Spain | XX | XX (XX.X) | ×× | XX (XX.X) | ×× | XX (XX.X) |
| : | : | | | | | | |

Only elevated serum transaminases related TEAEs are presented.

Treatment emergent adverse events (TEAEs) are defined as an adverse event that started after administration of study drug. If a subject experienced more than one TEAE, the subject is counted once for each system organ class (SOC) and once for each preferred term

SOCs are ordered in decreasing frequency of the total number of subjects with TEAEs reported in each SOC and PTs are ordered within a SOC in decreasing frequency of the total number of subjects with each TEAE.

Adverse events were coded using the MedDRA Dictionary, version xx.x. N = the number of subjects in the analysis set. (%) = Subjects/N\*100.

Source: Listing 16.2.7.1 and Listing 16.2.7.2

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS

Repeat for overall and all study phases. Include all countries as applicable NOTES:

Elevated serum transaminases defined as: aedecod in ("Alanine aminotransferase increased", "Aspartate aminotransferase increased", Include related events only

"Hypertransaminasaemia", "Transaminases increased")

Table 14.3.2.1 Haematology Values and Change from Baseline over Time

(Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | | 5 to 10 years (N=XX) | years<br>X) | 11 to 17 years $(N=XX)$ | 7 years<br>XX) | Overall (N=XX) | all<br>(X) |
|---|---|---|---|---|---|---|---|
| | • | Observed | Change | Observed | Change | | Change |
| Visit | Statistics | value | baseline | value | baseline | value | baseline |
| XXX | ជ | XX | | ×× | | ×× | |
| | Mean | XX.XX | | XX.XX | | XX.XX | |
| | SD | XX.XX | | XX.XX | | XX.XX | |
| | Minimum | ×× | | ×× | | ×× | |
| | Median | XX.X | | XX.X | | XX.XX | |
| | Maximum | XX | | ×× | | XX | |
| | 25th percentile | x.xx | | ×.×× | | ×.×× | |
| | 75th percentile | ×.<br>×. | | хх. х | | хх. х | |
| XXX | n | ×× | ×× | ×× | ×× | ×× | ×× |
| | Mean | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | × | ×× | ×× | ×× | ×× | ×× |
| | Median | xx.x | XX.X | ××.×× | XX.X | ××.×× | XX.X |
| | Maximum | XX | ×× | ×× | XX | XX | ×× |
| | 25th percentile | XX.XX | XX.X | XX.XX | XX.X | XX.XX | XX.X |
| | 75th percentile | ××.× | xx.x | ×.× | ××.× | ××.× | ××.× |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). At each time point, only subjects with a value at both baseline and that time point are included in the change from baseline column. N = 1 the number of subjects in the analysis set. n = 1 the number of subjects with a measurement.

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T XXX 01.SAS

Source: Listing 16.2.8.9

NOTES: Repeat for all visits and parameters.


Table 14.3.2.2 Clinical Significance of Haematology Values over Time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| Visit | Result | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| XXX | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Normal | (X.XX) XX | XX (XX.X) | XX (XX.X) |
| | NCS | (XX.X) | XX (XX.X) | (XX.X) XX |
| | CS | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXX | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | NCS | (X.XX) XX | XX (XX.X) | XX (XX.X) |
| | CS | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXX | Total | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | NCS | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | CS | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| ÷ | | | | |

CS = clinically significant, NCS = not clinically significant. NCS = not clinically significant. NCS = not clinically significant. NCS = not clinically significant. NCS = (n/number virt) and (3) = (3) and (3) = (Source: Listing 16.2.8.9

PROGRAM NAME:T\_XXX\_01.SAS

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX

NOTES: Repeat for all visits and parameters.

Table 14.3.2.3 Shift in Haematology Values over Time (Safety Analysis Set)

Age Group = XXX
Parameter: <Parameter (Unit)>

| Normal | | | | | Base | Baseline | | |
|---|---|---|---|---|---|---|---|---|
| Normal XX (XX.X) X | Visit | Result | Normal<br>n (%) | CS & Low<br>n (%) | CS & High<br>n (%) | NCS & Low<br>n (%) | NCS & High<br>n (%) | Total<br>n (%) |
| CS & Low | XXX | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| CS & High XX (XX.X) NCS & Low XX (XX.X) | | CS & Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| NCS & Low | | CS & High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| NCS & High XX (XX.X) XX (X | | NCS & Low | XX (XX.X) | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total XX (XX.X) | | NCS & High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal XX (XX.X) | | Total | XX (XX.X) | | XX (XX.X) | XX (XX.X) | (XX.X) | XX (XX.X) |
| XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX X | XXX | Normal | (XX.XX) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | | CS & Low | (XXXX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | (X.XX) XX | XX (XX.X) |
| XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | | CS & High | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | | XX (XX.X) |
| XX (XX.X) XX (XX | | NCS & Low | (XXXX) XX | | XX (XX.X) | XX (XX.X) | (X.XX) XX | |
| xx (xx.x) | | NCS & High | XX (XX.X) | | | XX (XX.X) | | |
| | | Total | (XXXX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | (X.XX) XX | XX (XX.X) |

CS = clinically significant, NCS = not clinically significant.

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = [(n/number with a value at that visit)\*100].treatment in the Efficacy Phase (Visit 4).

Source: Listing 16.2.8.9

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Repeat for all treatment groups, post-baseline visits and parameters. NOTES:

Age group = 5 to 10 years; 11 to 17 years; Overall

Table 14.3.3.1 Serum Clinical Chemistry Values and Change from Baseline over Time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | | 5 to 10 years (N=XX) | years (XX) | | 11 to 1 (N= | 11 to 17 years (N=XX) | | Ove | Overall (N=XX) | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Change | % Change | • | Change | % Change | | | |
| Visit | Statistics | Observed<br>value | from<br>baseline | from<br>baseline | Observed value | from<br>baseline | from<br>baseline | Observed<br>value | from<br>baseline | % Change from<br>baseline |
| XXX | ជ | X | | | × | | | × | | |
| | Mean | ×.×× | | | ××. | | | XX.X | | |
| | SD | XX.XX | | | XX.XX | | | XX.XX | | |
| | Minimum | XX | | | XX | | | XX | | |
| | Median | ×.×. | | | ×.×× | | | ×××× | | |
| | Maximum | XX | | | XX | | | XX | | |
| | 25th | XX.X | | | XX.X | | | ××.× | | |
| | percentile | | | | | | | | | |
| | 75th | ××.× | | | ××.× | | | ×××× | | |
| | percentile | | | | | | | | | |
| ××× | ជ | × | XX | ×× | ×× | ×× | ×× | ×× | ×× | XX |
| | Mean | ××.× | ××.× | ××.× | ××.× | ××.× | ××.× | ×.×× | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | ×× | ×× | XX | XX | ×× | ×× | XX |
| | Median | ××.× | ××.× | ×.×× | ××.× | ××.× | xx.x | ×.×× | XX.X | XX.XX |
| | Maximum | XX | ×× | XX | × | ×× | XX | XX | XX | XX |
| | 25th | XX.X | ××.× | ××.× | ×××× | ××. | ×.× | ××.× | ×.×× | XX.X |
| | percentile | | | | | | | | | |
| | 75th | XX.X | XX.XX | XX.X | ×.×× | XX.X | XX.X | XX.XX | XX.XX | XX.XX |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). percentile

At each time point, only subjects with a value at both baseline and that time point are included in the change from baseline column. N = the number of subjects in the analysis set. n = the number of subjects with a measurement.

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Repeat for all visits and parameters (metabolic panel, LFTS, Fasting Lipid panel (local and central), EFAs, Fat-soluble vitamin Source: Listings 16.2.8.1, 16.2.8.2, 16.2.8.3, 16.2.8.4, 16.2.8.5, 16.2.8.6, 16.2.8.7, 16.2.8.8 levels, hormones, sex hormones, serum lipase). Footnotes as per Table 14.3.2.1 (as applicable) NOTES:

#### SQN Clinical study no: OCH19003

Table 14.3.3.2 Clinical Significance of Serum Clinical Chemistry Values over Time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

Repeat of Table 14.3.2.2

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS Source: Listings 16.2.8.1, 16.2.8.2, 16.2.8.3, 16.2.8.4, 16.2.8.5, 16.2.8.6, 16.2.8.7, 16.2.8.8 Repeat for all visits and parameters (metabolic panel, LFTS, Fasting Lipid panel (local and central), EFAs, Fat-soluble vitamin NOTES:

levels, hormones, sex hormones, serum lipase). Footnotes as per Table 14.3.2.1 (as applicable)


#### SQN Clinical study no: OCH19003

Table 14.3.3.3 Shift in Clinical Chemistry Values over Time

(Safety Analysis Set)

Age Group = XXX
Parameter: <Parameter (Unit)>

Repeat of Table 14.3.2.3

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS Source: Listings 16.2.8.1, 16.2.8.2, 16.2.8.3, 16.2.8.4, 16.2.8.5, 16.2.8.6, 16.2.8.7, 16.2.8.8 Repeat for all visits and parameters (metabolic panel, LFTS, Fasting Lipid panel (local and central), EFAs, Fat-soluble vitamin NOTES:

levels, hormones, sex hormones, serum lipase). Footnotes as per Table 14.3.2.1 (as applicable) Age group = 5 to 10 years; 11 to 17 years; Overall

Table 14.3.3.4 Summary of Maximum Clinical Chemistry Values

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| | | 5 to 10 years | 11 to 17 years |
|---|---|---|---|
| Parameter | Statistics | (N=XX) | (N=XX) |
| Alanine Transaminase | ٤ | × | * |
| | • | • | 4 4 4 4 4 |
| | Mean | XX.XX | XX.X |
| | SD | XX.XX | XX.XX |
| | Minimum | XX | XX |
| | Median | XX.X | XX.X |
| | Maximum | XX | XX |
| | 25th percentile | XX.XX | XX.X |
| | 75th percentile | X.XX | XX.X |
| Aspartate Aminotransferase | ជ | XX | ×× |
| | Mean | ×. ×. | XX.X |
| | SD | XX.XX | XX.XX |
| | Minimum | XX | XX |
| | Median | ××.× | XX.XX |
| | Maximum | XX | XX |
| | 25th percentile | XX.XX | XX.X |
| | 75th percentile | XX.X | XX.X |
| N = the number of subjects in the analysis set. n Source: Listing 16.2.8.3 | e analysis set. $n$ = the number of subjects with a measurement. | th a measurement. | |
| PROGRAM NAME:T_XXX_01.SAS Di | DATE OF RUN:XXXXXXXXX TIME OF RUN: XX:XX:XX | X DATE OF EXTRACTION:XXXXXXXX | × |

NOTES: Maximum post-baseline values for ALT, AST, ALP and TBL

Table 14.3.3.4 Summary of Maximum Clinical Chemistry Values (Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

| Parameter | Statistics | 5 to 10 years<br>(N=XX) | 11 to 17 years<br>(N=XX) |
|---|---|---|---|
| Alkaline Phosphatase | ជ | ×× | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Minimum | XX | XX |
| | Median | XX.X | XX.X |
| | Maximum | XX | XX |
| | 25th percentile | XX.X | XX.X |
| | 75th percentile | x.xx | XX.X |
| Total Bilirubin | и | XX | ×× |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Minimum | XX | XX |
| | Median | XX.X | XX.X |
| | Maximum | XX | XX |
| | 25th percentile | XX.X | XX.X |
| | 75th percentile | ×.×× | XX.X |

N = the number of subjects Source: Listing 16.2.8.3

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Maximum post-baseline values for ALT, AST, ALP and TBL NOTES:

Table 14.3.3.5 Summary of Subjects Exceeding Hepatotoxicity Thresholds over Time (Safety Analysis Set)

| XXX | | | 4 | 4 | |
|-----|-----|-------------|-----------|-----------|-----------|
| | AST | > 3 × ULN | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| | | > 5 × ULN | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | > 10 x ULN | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | > 20 x ULN | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | ALT | > 3 × ULN | XX (XX.X) | XX (XX.X) | (XX.X) |
| | | > 5 × ULN | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | > 10 x ULN | (XX.X) XX | XX (XX.X) | XX (XX.X) |
| | | > 20 x ULN | XX (XX.X) | XX (XX.X) | (XX.X) |
| | ALP | > 1.5 x ULN | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | TBL | > 1.5 x ULN | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | > 2 × UIN | XX (XX.X) | XX (XX.X) | XX (XX.X) |

ALP = Alkaline Phosphatase. ALT = Alanine Transaminase. AST = Aspartate Aminotransferase. TBL = Total Bilirrubin. N = the number of subjects in the analysis set. n = the number of subjects with a measurement. Source: Listing 16.2.8.3

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for each post-baseline visit.

Table 14.3.3.6 Time to Onset of Liver Function Test Abnormality

(Safety Analysis Set)

);;;;

Parameter: <Parameter (Unit)>

| | 5 to 10 years (N=XX) | 11 to 17 years<br>(N=XX) |
|---|---|---|
| Number of subjects with LFT $> x$ 3 ULN, n (%) | XX (XX.X) | XX (XX.X) |
| Time to onset (days) [1] | | |
| u. | XX | XX |
| Mean | XX.XX | XX.X |
| SD | XX.XX | XX.XX |
| Minimum | XX | XX |
| Median | XX.X | XX.X |
| Maximum | XX | XX |
| 25th percentile | XX.X | XX.X |
| 75th percentile | XX.X | X.X.X |
| Number of subjects with ongoing elevation, n (%) | xx (xx.x) | xx (xx.x) |
| Duration of abnormality (days) [2] | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Minimum | XX | XX |
| Median | XX.X | XX.X |
| Maximum | XX | XX |
| 25th percentile | XX.X | XX.X |
| 75th percentile | XX.X | X.XX |
| CI = Confidence Interval. LFT = Liver Function Test. ULN = Upper Limit of Normal. [1] Time to first LFT abnormality is derived as: Date of the first LFT assessment that is $>= 3 \times \text{ULN}$ or greater - Date of first LFT assessment that is $>= 3 \times \text{ULN}$ or greater - Date of first LFT assessment that is $>= 3 \times \text{ULN}$ assessment date of resolution of the first LFT abnormality (resolution defined as $>= 3 \times \text{ULN}$ ). Subjects with an ongoing elevation will be censored at their last laboratory assessment date containing and ALT results. N = the number of subjects meeting the criterion. (%) = $n/N*100$ . Source: Listing 16.2.8.3 | that is >= 3 lution defined at their last g the criteric | x ULN or greater - Date of first dose + 1.<br>l as <3 x ULN) - Date of the first LFT<br>laboratory assessment date containing both AST<br>on. |

PROGRAM NAME: T\_XXX\_01.SAS DATE OF RUN: XXXXXXXXXX TIME OF RUN: XX:XX:XX

DATE OF EXTRACTION: XXXXXXXX

NOTES: Present for ALT and AST abnormalities.

#### SQN Clinical study no: OCH19003

Table 14.3.4.1 Urinalysis Values and Change from Baseline over Time

(Safety Analysis Set)

Parameter: <Parameter (Unit)>

Repeat of Table 14.3.2.1

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Footnotes as per Table 14.3.2.1 (as applicable) Repeat for all visits and parameters. Source: Listing 16.2.8.10 NOTES:

#### SQN Clinical study no: OCH19003

Table 14.3.4.2 Clinical Significance of Urinalysis Values over Time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

Repeat of Table 14.3.2.2

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Footnotes as per Table 14.3.2.2 (as applicable) Repeat for all visits and parameters. Source: Listing 16.2.8.10 NOTES:


#### SQN Clinical study no: OCH19003

Table 14.3.4.3 Shift in Urinalysis Values over Time

(Safety Analysis Set)

Age Group = XXX Parameter: <Parameter (Unit)>

Repeat of Table 14.3.2.3

DATE OF EXTRACTION:XXXXXXXX

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Footnotes as per Table 14.3.2.3 (as applicable) Repeat for all visits and parameters. Source: Listing 16.2.8.10 Age group = 5 to 10 years; 11 to 17 years; Overall NOTES:

Table 14.3.5.1 Vital Signs and Change from Baseline over Time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | | Ω | 5 to 10 years (N=XX) | Ø | T | <pre>11 to 17 years (N=XX)</pre> | rs | | Overall (N=XX) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Statistics | Observed | Change<br>from<br>baseline | % Change<br>from<br>baseline | Observed<br>value | Change<br>from<br>baseline | % Change<br>from<br>baseline | Observed<br>value | Change<br>from<br>baseline | % Change<br>from<br>baseline |
| XXX | и | ×× | | | × | | | × | | |
| | Mean | ×.×. | | | ×.×× | | | ×.×× | | |
| | SD | XX.XX | | | XX.XX | | | XX.XX | | |
| | Minimum | ×× | | | ×× | | | ×× | | |
| | Median | xx.x | | | ××.× | | | x.xx | | |
| | Maximum | ×× | | | ×× | | | XX | | |
| | 25th percentile | ×.×× | | | ×.×× | | | ×.×× | | |
| | 75th percentile | XX.X | | | XX.X | | | XX.X | | |
| XXX | п | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Mean | xx.x | ×.×× | ×.×× | ××.× | ×.×. | ××.× | ×.×× | ××.×× | ××.× |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | ×× | ×× | × | ×× | ×× | ×× | ×× | ×× |
| | Median | ×.×× | ×.×× | ×.×× | ×.×× | ×.×× | ××.× | ×.×× | ×.×× | ××.× |
| | Maximum | ×× | ×× | ×× | × | ×× | ×× | ×× | ×× | ×× |
| | 25th percentile | XX.X | ××.×× | XX.XX | XX.XX | XX.X | XX.X | ×.×× | ××.×× | ××.× |
| | 75th percentile | XX.X | x.xx | XX.X | XX.X | ××.×× | ××.× | XX.X | ××.× | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). At each time point, only subjects with a value at both baseline and that time point are included in the change from baseline column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement.Source: Listing 16.2.9.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits and parameters.

\* Present change from baseline for Maximum, Minimum and Last post baseline value for height/BMI percentiles and z-scores only.


Table 14.3.5.1 Vital Signs and Change from Baseline over Time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | | N | to 10 years | Ø | 11 | to 17 years | rs | | Overall | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | (N=XX) | | | (N=XX) | | | (N=XX) | |
| | | Observed | Change | % Change<br>from | Observed | Change | % Change<br>from | heyyaed | Change | % Change<br>from |
| Visit | Statistics | value | baseline | baseline | value | baseline | baseline | value | baseline | baseline |
| Maximum Post-baseline<br>Value * | и | XX | XX | XX | XX | XX | ×× | XX | XX | XX |
| | Mean | ×.×× | ××.× | ×.×× | ×.×× | ×.×× | xx.x | x.xx | ××.× | XX.X |
| | SD | xx.xx | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX |
| | Minimum | ×× | XX | XX | XX | ×× | XX | XX | XX | XX |
| | Median | x.xx | ×.×× | ×.×× | x.xx | ×.×× | xx.x | ×.×× | ×.× | x.xx |
| | Maximum | ×× | ×× | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| | 25th percentile | x.xx | XX.X | XX.XX | XX.XX | XX.XX | ××.× | XX.XX | XX.XX | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Minimum Post-baseline<br>Value * | и | XX | XX | XX | XX | XX | XX | XX | XX | ×× |
| | Mean | XX.XX | XX.X | XX.XX | XX.XX | XX.X | ××.× | XX.XX | XX.XX | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | × | ×× | × | ×× | ×× | ×× | ×× | ×× |
| | Median | ××.× | ××.× | ×.×× | ××.× | ×.×× | XX.X | ×.×× | ××.× | ××.× |
| | Maximum | ×× | × | ×× | × | ×× | ×× | ×× | ×× | ×× |
| | 25th percentile | ××.× | ×.×× | XX.XX | ××.× | XX.XX | XX.X | XX.XX | XX.XX | XX.XX |
| | 75th percentile | XX.X | x. x. | ×.× | ×. × | ×. ×. | XX.X | XX.XX | ×. ×. | X. XX |
| Last Post-baseline Value * | п | XX | XX | XX | X | XX | XX | XX | XX | XX |
| | Mean | ××.× | ×.×× | XX.XX | ××.× | XX.XX | XX.X | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | × | ×× | × | ×× | ×× | ×× | ×× | ×× |
| | Median | XX.XX | XX.X | XX.XX | XX.XX | XX.XX | XX.X | XX.XX | XX.XX | XX.X |
| | Maximum | ×× | × | ×× | × | ×× | ×× | ×× | ×× | ×× |
| | 25th percentile | x.xx | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | ××.× | ××.× | xx.x | ××.× | xx.x | ××.× | xx.x | ×.× | xx.x |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). At each time point, only subjects with a value at both baseline and that time point are included in the change from baseline column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement.

Source: Listing 16.2.9.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits and parameters.
\* Present change from baseline for Maximum, Minimum and Last post baseline value for height/BMI percentiles and z-scores only.


Table 14.3.6.1 Summary of Overall ECG Interpretation over Time (Safety Analysis Set)

| Visit | Result | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| XXX | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Normal | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Abnormal, NCS | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Abnormal, CS | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| XXX | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Abnormal, NCS | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Abnormal, CS | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| :: | | | | |

NCS = not clinically significant, CS = clinically significant. N = 1 is the number of subjects in the analysis set. N = 1 the number of subjects in the analysis set. N = 1 is the number of subjects in the analysis set. N = 1 is the number of subjects in the analysis set. N = 1 is the number of subjects in the analysis set. N = 1 is the number of subjects in the analysis set. N = 1 is the number of subjects in the analysis set. Source: Listing 16.2.10.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits.

Table 14.3.6.2 Shift in Overall ECG Interpretation over Time (Safety Analysis Set)

Age Group = XXX

| | | | Base | Baseline | |
|---|---|---|---|---|---|
| Visit | Result | Normal<br>n (%) | Abnormal, NCS<br>n (%) | Abnormal, CS<br>n (%) | Total<br>n (%) |
| XXX | Normal | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Abnormal, NCS | (X.XX) XX | (XXXX) XX | XX (XX.X) | XX (XX.X) |
| | Abnormal, CS | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXX | Normal | (XXXXX) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Abnormal, NCS | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Abnormal, CS | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | (X.XX) XX | (XX.X) | XX (XX.X) | XX (XX.X) |
| : | | | | | |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study

treatment in the Efficacy Phase (Visit 4)..

NCS = not clinically significant.

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = [(n/number who have a value at that visit)\*100].

Source: Listing 16.2.10.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Overall.

NOTES: Repeat for all post-baseline visits.

Age group = 5 to 10 years; 11 to 17 years;


Table 14.3.7.1 Summary of Echocardiography (Standard of Care) over Time (Safety Analysis Set)

| | | | | | 11 to 17 | |
|---|---|---|---|---|---|---|
| Visit | | Ж | Result | 5 to 10 years (N=XX) | years<br>(N=XX) | Overall (N=XX) |
| XXX | Echocardiography performed? | Ė | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Ä | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Z | N/A | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Atherosclerosis and/or aortic valve | disease? | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Z | N/A | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Thickening of aortic valve leaflets | | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N | N/A | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Is this new? | 'Ā | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Z | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Is this progression of the condition | | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Z | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| <pre>N = the number of subject visit)*100]. Source: Listing 16.2.11.1</pre> | s in the analysis set. n | = the number of subjects meeting the criterion. (%) = $[(n/number\ who\ have\ a\ value\ at\ that$ | eting the criter | ion. (%) = [(n/ | number who have a | value at that |
| PROGRAM NAME: T_XXX_01.SAS | T_XXX_01.SAS DATE OF RUN:XXXXXXXX | XX TIME OF RUN: XX:XX:XX | | DATE OF EXTRACTION:XXXXXXXX | | |

NOTES: Repeat for all visits (Baseline, week 24, week 56, week 104).


Table 14.3.7.1 Summary of Echocardiography (Standard of Care) over Time (Safety Analysis Set)

| Visit | | Result | 5 to 10 years (N=XX) | 11 to 17<br>years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| Fusion of t | Fusion of the aortic valve leaflets | Yes | XX (XX.X) | XX (XX.X) | (X.XX) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N/A | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Is this | this new? | Yes | XX (XX.X) | (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Is this | Is this progression of the condition | Yes | XX (XX.X) | (XX.X) | (XXXX) |
| | | No | XX (XX.X) | XX (XX.X) | (X.XX) |
| Thickening | Thickening of the aortic root | Yes | XX (XX.X) | (XX.X) | (XXXX) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N/A | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Is this | new? | Yes | XX (XX.X) | (XX.X) | (XXXX) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Is this | Is this progression of the condition | Yes | XX (XX.X) | XX (XX.X) | (XXXX) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |

N = 1 the number of subjects in the analysis set. n = 1 the number of subjects meeting the criterion. (%) = [(n/number who have a value at that visit)\*100]. Source: Listing 16.2.11.1

PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX

NOTES: Repeat for all visits (Baseline, week 24, week 56, week 104).


Table 14.3.7.1 Summary of Echocardiography (Standard of Care) over Time (Safety Analysis Set)

| Visit | | Result | 5 to 10<br>years<br>(N=XX) | 11 to 17<br>years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| | Flow acceleration or turbulence over the aortic valve | Yes<br>No<br>N/A | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) |
| | Is this new? | Yes<br>No | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| | Is this progression of the condition | Yes.<br>No | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| | Regions present? | Supravalvular region<br>In the ascending aorta | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| | Aortic valve regurgitation? | Yes<br>No<br>N/A | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) |
| | Is this new? | Y e s<br>No | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| | Is this progression of the condition | Yes<br>No | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = [(n/number who have a value at that visit)\*100].Source: Listing 16.2.11.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX

NOTES: Repeat for all visits (Baseline, week 24, week 56, week 104).
Table 14.3.7.1 Summary of Echocardiography (Standard of Care) over Time (Safety Analysis Set)

| ;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;;; | | ,<br>,<br>, | 5 to 10 years | 11 to 17<br>years | Overall |
|---|---|---|---|---|---|
| ۵.<br>۲ | | IVESUIC | ( V.V.—NI ) | (114-72.7) | ( VVV — NT ) |
| | Coronary ostial narrowing or flow disturbances? | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N/A | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Is this new? | Yes | XX (XX.X) | (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Is this progression of the condition | Yes | XX (XX.X) | (XX.X) | (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Ventricular findings? | Yes | XX (XX.X) | (XX.X) | XX (XX.X) |
| | | No | (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N/A | XX (XX.X) | (X.XX) XX | XX (XX.X) |
| | Left ventricular hypertrophy? | Yes | XX (XX.X) | (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | N/A | XX (XX.X) | (X.XX) XX | (XX.X) |
| | Is this new? | Yes | XX (XX.X) | (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | (X.XX) XX | XX (XX.X) |
| | Is this progression of the condition | Yes | XX (XX.X) | (XX.X) | XX (XX.X) |
| | | 0 | (X, XX) XX | (XX, XX) | XX (XX.X) |

visit)\*100]. Source: Listing 16.2.11.1

NOTES: Repeat for all visits (Baseline, week 24, week 56, week 104).


TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.7.1 Summary of Echocardiography (Standard of Care) over Time (Safety Analysis Set)

| Visit | Result | 5 to 10 years (N=XX) | 11 to 17<br>years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Impairment of left ventricular function? | K es<br>No | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| | N/A | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Is this new? | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Is this progression of the condition | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| : | | | | |
| $N$ = the number of subjects in the analysis set. $n$ = the n visit) $\star 100].$ Source: Listing 16.2.11.1 | the number of subjects meeting the criterion. (%) = $[(n/number\ who\ have\ a\ value\ at\ that$ | criterion. (%) = $[(n/n)]$ | 'number who have | a value at that |
| PROGRAM NAME: T_XXX_01.SAS DATE OF RUN: XXXXXXXXX T | TIME OF RUN: XX:XX:XX DATE OF | DATE OF EXTRACTION:XXXXXXXX | | |

NOTES: Repeat for all visits (Baseline, week 24, week 56, week 104).

Table 14.3.7.2 Summary of Subjects with Worsening in Echocardiography over Time (Safety Analysis Set)

| 4 6 | 5 | 5 to 10 years | 11 to 17 years | Overall |
|---|---|---|---|---|
| Visit | | (N=XX) | (N=XX) | (N=XX) |
| Number of subjects with a worsening from | sening from | | | |
| baseline by: | | | | |
| Week 24 | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Week 56 | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| EOT / Week 104 | | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| N = the number of subjects in the analysis set. | =<br>u | e number of subjects meetir | the number of subjects meeting the criterion.<br>(\$) = [(n/N) $*100].$ | |
| source: Listing 10.2.11.1 | | | | |
| PROGRAM NAME: T_XXX_01.SAS | DATE OF RUN:XXXXXXXX | TIME OF RUN: XX:XX:XX | DATE OF EXTRACTION:XXXXXXXX | |

Table 14.3.8.1.1 Summary of Lipid Accumulation in the Liver over Time (Safety Analysis Set)

| liver fat | NMR Scan (N=XX) | tan<br>) | Ultraso<br>(N= | Ultrasound Scan<br>(N=XX) | |
|---|---|---|---|---|---|
| Total <pre> &lt; 10% liver fat &gt; 10% and \$ 20% liver fat &gt; 20% liver fat Total <pre></pre></pre> | 5 to 10 years 11 to 17 years (N=XX) (N=XX) | .1 to 17 years (N=XX) | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
| <pre>\$ 10% liver fat &gt; 10% and \$ 20% liver fat &gt; 20% liver fat Total \$ 10% liver fat &gt; 10% and \$ 20% liver fat &gt; 10% and \$ 20% liver fat</pre> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| > 10% and \$ 20% liver fat<br>> 20% liver fat<br>Total<br>\$ 10% liver fat<br>> 10% and \$ 20% liver fat | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| > 20% liver fat Total \$ 10% liver fat > 10% and \$ 20% liver fat | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total <pre> </pre> <pre> <pre> <pre> </pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre> <pre< td=""><td>XX (XX.X)</td><td>XX (XX.X)</td><td>XX (XX.X)</td><td>XX (XX.X)</td><td>XX (XX.X)</td></pre<></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre> | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| liver fat<br>and ≤ 20% liver fat | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| and < 20% liver fat | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1: | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| TIVEr IAU | (X.X.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = [(n/number who have a value at that visit)\*100].

Source: Listing 16.2.12.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits.

# Amryt Pharma study no: APH-19

### SQN Clinical study no: OCH19003

Table 14.3.8.1.2 Summary of Lipid Accumulation in the Liver over Time (Sensitivity Analysis - Excluding Site 12)

(Safety Analysis Set)

Excluding Site 12

Repeat of Table 14.3.8.1.1

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = [(n/number who have a value at that visit)\*100].

Source: Listing 16.2.12.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits. Exclude Site 12 data Repeat for Site 12 only


Table 14.3.8.2.1 Shift in Lipid Accumulation in the Liver over Time (Safety Analysis Set)

Age Group = XXX

| | | | | 0 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
|---|---|---|---|---|---|
| | | | >10% and < 20% | | |
| | | <pre>&lt; 10% liver fat</pre> | liver fat | >20% liver fat | Total |
| Visit | Result | n (%) | n (%) | n (%) | n (%) |
| XXX | <pre>&lt; 10% liver fat</pre> | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| | > 10% and < 20% liver fat | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | > 20% liver fat | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXX | <pre>&lt; 10% liver fat</pre> | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| | and ≤ | (X.XX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | > 20% liver fat | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = [(n/number who have a value at that visit)\*100].Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

visit)\*100]. Source: Listing 16.2.12.1 TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all post-baseline visits. Age group = 5 to 10 years; 11 to 17 years; Overall.

## Amryt Pharma study no: APH-19

#### SQN Clinical study no: OCH19003

Table 14.3.8.2.2 Shift in Lipid Accumulation in the Liver over Time (Sensitivity Analysis - Excluding Site 12)

(Safety Analysis Set)

Excluding Site 12 Age Group = XXX

Repeat of Table 14.3.8.2.

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4). N = 1 the number of subjects in the analysis set. N = 1 the number of subjects in the analysis set. N = 1 the number of subjects in the analysis set.

visit) \*100].

Source: Listing 16.2.12.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Repeat for all post-baseline visits. Age group = 5 to 10 years; 11 to 17 years; Overall. NOTES:

Exclude Site 12 data

Repeat for Site 12 only


Table 14.3.8.3.1 Summary of Lipid Accumulation in the Liver over Time (Safety Analysis Set)

| | | ιΩ | 5 to 10 years (N=XX) | Ñ | 11 | 11 to 17 years (N=XX) | rs | | Overall (N=XX) | |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | Observed | Change<br>from | % Change<br>from | Observed | Change<br>from | % Change<br>from | Observed | Change<br>from | % Change from |
| Visit | statistics | value | paseline | paseline | value | paseline | baseline | value | paseline | Daseline |
| XXX | n | XX | | | XX | | | × | | |
| | Mean | XX.XX | | | XX.X | | | XX.X | | |
| | SD | XX.XX | | | XX.XX | | | XX.XX | | |
| | Minimum | ×× | | | ×× | | | ×× | | |
| | Median | XX.XX | | | XX.X | | | XX.XX | | |
| | Maximum | ×× | | | ×× | | | ×× | | |
| | 25th percentile | XX.X | | | ×.×× | | | XX.X | | |
| | 75th percentile | XX.X | | | XX.X | | | XX.X | | |
| XXX | п | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.XX | XX.X | XX.X | XX.X | ×.×× | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | ×× | × | ×× | × | ×× | ×× | × | ×× | ×× |
| | Median | XX.X | XX.X | XX.XX | XX.X | XX.X | XX.X | ×.×× | XX.XX | XX.XX |
| | Maximum | ×× | × | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| | 25th percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | 75th percentile | ×. ×. | ×.× | ×. ×. | ×.× | ×. × | ×× | ×.×. | ×.× | ×.× |

Only NMR scan assessments are included.

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

At each time point, only subjects with a value at both baseline and that time point are included in the change from baseline column. N = the number of subjects in the analysis set who receive the respective treatment/dose. <math>n = the number of subjects with a measurement. Source: Listing 16.2.12.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits and parameters.


#### Amryt Pharma study no: APH-19

#### SQN Clinical study no: OCH19003

Table 14.3.8.3.2 Summary of Lipid Accumulation in the Liver over Time

(Safety Analysis Set)

Excluding Site 12

Repeat of Table 14.3.8.3.1

Only NMR scan assessments are included.

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

At each time point, only subjects with a value at both baseline and that time point are included in the change from baseline column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. Source: Listing 16.2.12.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits and parameters.

Exclude Site 12 data Repeat for Site 12 only


Table 14.3.8.4.1 Summary of Lipid Accumulation Increase over Time (Safety Analysis Set)

| Visit | | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| XXX | ∨<br>∾ | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | >10% | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | >15% | (X.XX) XX | XX (XX.X) | (XX.X) |
| | >20% | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXX | \<br>\<br>% | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | >10% | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | >15% | (X.XX) XX | XX (XX.X) | (XX.X) |
| | >20% | XX (XX,X) | XX (XX,X) | XX (XX,X) |

Only NMR scan assessments are included. N = 1 in the analysis set who receive the respective treatment/dose. n = 1 the number of subjects with a measurement. Source: Listing 16.2.12.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Repeat for each visit The increases will be presented cumulatively. NOTES:


#### Amryt Pharma study no: APH-19

#### SQN Clinical study no: OCH19003

Table 14.3.8.4.2 Summary of Lipid Accumulation Increase over Time

(Safety Analysis Set)

Excluding Site 12

Repeat of Table 14.3.8.4.1

Only NMR scan assessments are included. N = 1 in the analysis set who receive the respective treatment/dose. N = 1 the number of subjects with a measurement. Source: Listing 16.2.12.1

DATE OF EXTRACTION: XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

FOOTNOTE NOTES:

Present the maximum post-baseline change at the end. Exclude Site 12 data
Repeat for Site 12 only The increases will be presented cumulatively. Repeat for each visit

Table 14.3.9.1 Summary of Tanner Staging over Time (Safety Analysis Set)

| Visit | Result | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| XXX | Stage 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Stage 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Stage 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Stage 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Stage 5 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXX | Stage 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Stage 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Stage 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Stage 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Stage 5 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX,X) | XX (XX,X) | (XX,X) |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = [(n/number who have a value at that visit)\*100]. Source: Listing 16.2.12.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits.

Table 14.3.9.2 Summary of Sex Hormones in patients with Tanner Stage 2 2 over Time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | | 5 to 1 (N; | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | l7 years<br>=XX) | Ove<br>=N) | Overall (N=XX) |
|---|---|---|---|---|---|---|---|
| Visit | Statistics | Observed value | Change from baseline | Observed<br>value | Change from<br>baseline | Observed<br>value | Change from baseline |
| XXX | и | XX | | X | | ×× | |
| | Mean | XX.X | | XX.XX | | x.x. | |
| | SD | XX.XX | | XX.XX | | XX.XX | |
| | Minimum | XX | | ×× | | XX | |
| | Median | XX.XX | | x.xx | | x.xx | |
| | Maximum | XX | | XX | | XX | |
| | 25th percentile | XX.X | | XX.XX | | XX.X | |
| | 75th percentile | XX.XX | | XX.XX | | XX.X | |
| XXX | п | XX | XX | × | ×× | ×× | ×× |
| | Mean | XX.X | XX.X | XX.XX | XX.X | XX.X | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | XX.XX | XX.X | XX.XX | XX.XX | XX.X | XX.XX |
| | Maximum | XX | XX | XX | XX | XX | XX |
| | 25th percentile | XX.X | XX.X | XX.XX | XX.X | XX.X | XX.XX |
| | 75th percentile | XX.X | XX.X | XX.XX | XX.X | XX.X | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study

treatment in the Efficacy Phase (Visit 4).
At each time point, only subjects with a value at both baseline and that time point are included in the change from baseline column.

N = the number of subjects in the analysis set. n = the number of subjects with a measurement. Source: Listing 16.2.13.2

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits and parameters (serum testosterone, serum oestradiol).

Table 14.3.9.3 Shift in Tanner Staging Over Time (Safety Analysis Set)

Age Group = XXX

| | | | | Baseline I | Baseline Tanner Staging | | |
|---|---|---|---|---|---|---|---|
| Visit | Tanner Staging | 7 | 2 | 3 | 8 | 2 | Total |
| ××× | ₽ | XX (XX.X) | XX (XX.X) | (XX.X) | XX (XX.X) | XX (XX.X) | XX XXX |
| | 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XXXX) XX | XX (XX.X) |
| | ĸ | (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 4 | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Ŋ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | | (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) |
| XXX | Н | (XXXX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX.X) |
| | 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | E | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Ŋ | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Etc | | | | | | | |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = 1 the number of subjects in the analysis set. n = 1 the number of subjects with a measurement. (%) = [(n/number who have a value at that the number of subjects in the analysis set.Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

vvisit)\*100].
[-] denotes a zero count in the table.

[-] denotes a zero count in the t. Source: Listing 16.2.13.2

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits

Age group = 5 to 10 years; 11 to 17 years; Overall.

Please display '-' instead of '0' for zero counts and foornote to say that '-' represents a zero count in the table?

Table 14.3.10.1 Summary of Pulmonary Function Test (PFT) Parameters and Change from Baseline over Time

(Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | | 5 to 10 years (N=XX) | years<br><x)< th=""><th>11 to 17 <math>y</math> (N=XX)</th><th>11 to 17 years (N=XX)</th><th>Overal (N=XX)</th><th>Overall (N=XX)</th></x)<> | 11 to 17 $y$ (N=XX) | 11 to 17 years (N=XX) | Overal (N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|---|---|
| Visit | Statistics | Observed<br>value | Change from<br>baseline | Observed<br>value | Change from<br>baseline | Observed<br>value | Change from baseline |
| XXX | а | X | | XX | | XX | |
| | Mean | XX.XX | | XX.XX | | XX.X | |
| | SD | XX.XX | | XX.XX | | XX.XX | |
| | Minimum | XX | | ×× | | ×× | |
| | Median | XX.XX | | ×.×× | | XX.X | |
| | Maximum | XX | | XX | | XX | |
| | 25th percentile | XX.XX | | XX.XX | | XX.X | |
| | 75th percentile | XX.X | | XX.X | | XX.X | |
| XXX | ď | ×× | × | XX | ×× | ×× | ×× |
| | Mean | XX.XX | XX.XX | XX.XX | XX.X | XX.X | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | XX | × | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.XX | XX.X | XX.XX |
| | Maximum | XX | XX | × | XX | XX | XX |
| | 25th percentile | XX.XX | XX.XX | XX.XX | XX.XX | XX.X | XX.XX |
| | 75th percentile | x.xx | XX.X | ×.× | xx.x | x.x. | XX.X |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

At each visit time point, only subjects with a value at both baseline and that time point are included in the change from baseline column. N = the number of subjects in the analysis set who receive the respective treatment/dose. <math>n = the number of subjects with a measurement.Source: Listing 16.2.13.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits and parameters.

Table 14.3.11.1 Summary of Xanthoma Assessment over Time (Safety Analysis Set)

| Visit | | Result | 5 to 10 years<br>(N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| XXX | Pre-existing xanthomas | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | present | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | No | | XX (XX.X) | |
| | Pre-existing tendon | Total | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | xaiiciioillas preseiic | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Anatomical locations | Achilles tendon | (XX.X) | (X.X.X) | XX (XX.X) |
| | | Dorsum of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Pre-existing cutaneous | Total | XX (XX.X) | (XX.X) | XX (XX.X) |
| | xantinomas present | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Anatomical locations | Tuberous, elbow | (XXXX) | (XXXX) XX | XX (XX.X) |
| | (cucaiidous) | Tuberous, knee | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, palm of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, soles of the feet | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Intertriginous, fingers | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Xanthelasmas, eyelids | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| XXX | etc | | | | |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = [(n/number who have a value at that visit)\*100]. Source: Listing 16.2.17.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits (baseline, week 56, week 104).

Table 14.3.11.2 Changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | Visit | Result | 5 to 10 years (N=XX) | 11 to 17<br>years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| Pre-existing xanthomas present | | Yes | (xx.x) | (XX.X) | XX (XX.X) |
| Pre-existing xanthomas changed since previous visit | Week 4 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | Yes | (XXXXX) XX | XX (XX.X) | (X.XX) XX |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. (%) = [(n/number who have pre-existing xanthoma)\*100], unless otherwise stated. [\*] (%) = [n / N] Source: Listing 16.2.17.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.11.2 Changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | | | | 11 to 17 | |
|---|---|---|---|---|---|
| | Visit | Result | 5 to $10 \text{ years}$ (N=XX) | years (N=XX) | Overall (N=XX) |
| Xanthomas reduced in size | Week 4 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | Yes | XX (XX.X) | XX (XX.X) | (XX.XX) |
| | Week 12 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Yes | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| | Week 20 | Yes | XX (XX.X) | XX (XX.X) | (XXXXX) |
| | Week 24 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | Yes | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| | Week 32 | Yes | XX (XX.X) | XX (XX.X) | (XXXXX) |
| | Week 36 | Yes | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| | Week 40 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | Yes | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| | Week 48 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | Yes | (X, XX) XX | XX (XX.X) | (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = 1 the number of subjects in the analysis set who receive the respective treatment/dose. n = 1 the number of subjects with a measurement. (%) (n + 1) (n

[\*] (%) = [n / N]Source: Listing 16.2.17.1

n

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.11.2 Changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | | | 5 to 10 years | 11 to 17<br>years | Overall |
|---|---|---|---|---|---|
| | Visit | Result | (XX=N) | (N=XX) | (N=XX) |
| Xanthomas resolved | Week 4 | Yes | XX (XX.X) | XX (XX.X) | (XX.X) |
| | Week 8 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = 1 the number of subjects in the analysis set who receive the respective treatment/dose. n = 1 the number of subjects with a measurement. (%) (n + 1) (n

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

<sup>[\*]</sup> (%) = [n / N]Source: Listing 16.2.17.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF RUN:XXXXXXXX

Table 14.3.11.2 Changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | : | | 5 to 10 years | 11 to 17<br>years | Overall |
|---|---|---|---|---|---|
| | Visit | Kesult | (N=XX) | (N=XX) | (N=XX) |
| Xanthomas increased in size | Week 4 | Yes | XX (XX.X) | (XX.X) | XX (XX.X) |
| | Week 8 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | Yes | (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | Yes | XX (XX.X) | XX (XX.X) | (XX.X) |
| | Week 80 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | Yes | XX (XX.X) | XX (XX.X) | (XXXX) XX |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = 1 the number of subjects in the analysis set who receive the respective treatment/dose. n = 1 the number of subjects with a measurement. (%) n = 1 (n) number who have pre-existing xanthoma)\*100], unless otherwise stated.


<sup>[\*]</sup> (%) = [n / N]Source: Listing 16.2.17.1

PROGRAM NAME:T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX

Table 14.3.11.2 Changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | | | C 7 | 11 to 17 | |
|---|---|---|---|---|---|
| | Visit | Result | (N=XX) | Years<br>(N=XX) | (N=XX) |
| New xanthomas present* | Week 4 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | Yes | XX (XX.X) | XX (XX.X) | (XXXXX) |
| | Week 40 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column.

N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. (%)

= [(n/number who have pre-existing xanthoma)\*100], unless otherwise stated.

[\*] (%) = [n / N] Source: Listing 16.2.17.1

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

DATE OF EXTRACTION:XXXXXXXX

Table 14.3.11.3 Summary of new xanthomas over Time (Safety Analysis Set)

| | Visit | Result | 5 to 10<br>years<br>(N=XX) | 11 to 17<br>years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| Pre-existing xanthomas present | | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| New tendon xanthomas present* | Week 4 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. (%) = [(n/number who have pre-existing xanthoma)\*100], unless otherwise stated. [\*] (%) = [n / N] Source: Listing 16.2.17.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF RUN:XXXXXXXX

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX

Table 14.3.11.3 Summary of new xanthomas over Time (Safety Analysis Set)

| | | | 5 to 10 | 11 to 17 | |
|---|---|---|---|---|---|
| | Visit | Result | years<br>(N=XX) | years<br>(N=XX) | Overall (N=XX) |
| Anatomical locations (tendon)* | Week 4 | Achilles tendon | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Dorsum of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | Achilles tendon | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Dorsum of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | Achilles tendon | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Dorsum of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Achilles tendon | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Dorsum of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Etc | | | | |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. (%) =  $[(n/number\ who\ have\ pre-existing\ xanthoma)*100]$ , unless otherwise stated. [\*] (%) =  $[n\ N]$  Source: Listing 16.2.17.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.11.3 Summary of new xanthomas over Time (Safety Analysis Set)

| | | | 5 to 10 | 11 to 17 | - |
|---|---|---|---|---|---|
| | Visit | Result | Years<br>(N=XX) | years<br>(N=XX) | (N=XX) |
| New cutaneous xanthomas present* | Week 4 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = 1 the number of subjects in the analysis set who receive the respective treatment/dose. n = 1 the number of subjects with a measurement. (%) (n + 1) (n

<sup>[\*]</sup> (%) = [n / N]Source: Listing 16.2.17.1

PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX

Table 14.3.11.3 Summary of new xanthomas over Time (Safety Analysis Set)

| | Visit | Result | 5 to 10<br>years<br>(N=XX) | 11 to 17<br>years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| Anatomical locations (cutaneous)* | Week 4 | Tuberous, elbow | XX (XX.X) | (XXXX) | (XX.X) |
| | | Tuberous, knee | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, palm of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, soles of the feet | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Intertriginous, fingers | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Xanthelasmas, eyelids | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | Tuberous, elbow | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Tuberous, knee | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, palm of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, soles of the feet | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Intertriginous, fingers | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Xanthelasmas, eyelids | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | Tuberous, elbow | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Tuberous, knee | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, palm of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, soles of the feet | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Intertriginous, fingers | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Xanthelasmas, eyelids | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | Tuberous, elbow | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Tuberous, knee | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, palm of the hands | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Planar, soles of the feet | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Intertriginous, fingers | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Xanthelasmas, eyelids | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. (%) = [(n/number who have pre-existing xanthoma)\*100], unless otherwise stated. [\*] (%) = [n / N] Source: Listing 16.2.17.1

PROGRAM NAME: T\_XXX\_01.SAS

DATE OF RUN:XXXXXXXX

TIME OF RUN: XX:XX:XX

DATE OF EXTRACTION:XXXXXXXX


Table 14.3.11.4 Cumulative changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | Visit | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Pre-existing xanthomas present | | (X.XX) | XX (XX.X) | XX (XX.X) |
| Xanthomas reduced in size by: | Week 4 | XX (XX.X) | (XX.X) | XX (XX.X) |
| | Week 8 | (XXXXX) XX | (XXXXX) XX | XX (XX.X) |
| | Week 12 | (XXXX) XX | (XXXXX) XX | XX (XX.X) |
| | Week 16 | (XXXX) XX | (XXXX) XX | XX (XX.X) |
| | Week 20 | (XXXX) XX | (XXXX) XX | XX (XX.X) |
| | Week 24 | XX (XX.X) | (XXXXX) XX | XX (XX.X) |
| | Week 28 | (XXXX) XX | (XXXX) XX | XX (XX.X) |
| | Week 32 | XX (XX.X) | (XX.X) XX | XX (XX.X) |
| | Week 36 | (XXXX) XX | (XXXXX) XX | XX (XX.X) |
| | Week 40 | (XXXX) XX | (XXXXX) XX | XX (XX.X) |
| | Week 44 | (XXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 48 | (XXXX) XX | (XXXXX) XX | XX (XX.X) |
| | Week 52 | XX (XX.X) | (XX.X) XX | XX (XX.X) |
| | Week 56 | (XXXX) XX | (XXXXX) XX | XX (XX.X) |
| | Week 68 | (XXXX) XX | (XX.XX) | XX (XX.X) |
| | Week 80 | (XXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 92 | (XXXX) XX | (XX.XX) | XX (XX.X) |
| | EOT / Week 104 | XX (XX.X) | (XX.X) XX | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = 1 the number of subjects in the analysis set who receive the respective treatment/dose. n = 1 the number of subjects with a measurement. [\*] (%) = [n / N]Source: Listing 16.2.17.1

PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX

Table 14.3.11.4 Cumulative changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | : | 5 to 10 years | 11 to 17 years | Overall |
|---|---|---|---|---|
| | Visit | (N=XX) | (N=XX) | (XX=N) |
| Xanthomas resolved by: | Week 4 | XX (XX.X) | (XXXX) XX | XX (XX.X) |
| | Week 8 | (XXXX) XX | (XXXX) XX | XX (XX.X) |
| | Week 12 | (XXXX) XX | (XXXXX) XX | XX (XX.X) |
| | Week 16 | (XXXX) XX | (XXXX) XX | XX (XX.X) |
| | Week 20 | (XXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 24 | (XXXX) XX | (XXXX) XX | XX (XX.X) |
| | Week 28 | (XXXX) XX | (XXXX) XX | XX (XX.X) |
| | Week 32 | (XXXX) XX | (XXXXX) XX | XX (XX.X) |
| | Week 36 | (XXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 40 | (XXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 44 | (XXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 48 | (XXXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 52 | (XX.XX) | (XX.X) | XX (XX.X) |
| | Week 56 | (XXXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 68 | (XXXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 80 | (XXXX) XX | (XX.X) XX | XX (XX.X) |
| | Week 92 | (XXXXX) XX | (XX.X) XX | XX (XX.X) |
| | EOT / Week 104 | (XXXX) XX | (XXXXX) XX | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. [\*] (%) = [n / N] Source: Listing 16.2.17.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.11.4 Cumulative changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | Visit | 5 to 10 years (N=XX) | 11 to 17 years (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Xanthomas increased in size by: | Week 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| • | Week 8 | (X.XX) XX | | (X.XX) XX |
| | Week 12 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | XX (XX.X) | XX (XX.X) | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. [\*] (%) = [n / N] Source: Listing 16.2.17.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

Table 14.3.11.4 Cumulative changes to pre-existing Xanthoma over Time (Safety Analysis Set)

| | | 5 to 10 years | 11 to 17 years | Overall |
|---|---|---|---|---|
| | Visit | (N=XX) | (N=XX) | (N=XX) |
| New xanthomas present by: | Week 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | XX (XX.X) | (XXXX) XX | XX (XX.X) |
| | Week 20 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | (XX.XX) | (XX.XX) | XX (XX.X) |
| | Week 56 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 92 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | XX (XX.X) | XX (XX.X) | XX (XX.X) |

At each time point, only subjects with a value at both baseline and that time point are included in the column. N = 1 the number of subjects in the analysis set who receive the respective treatment/dose. n = 1 the number of subjects with a measurement. [\*] (%) = [n / N] Source: Listing 16.2.17.1

DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

Table 14.3.12.1 Carotid Intima-Media Thickness and Flow-mediated Dilation Summary and Percentage Change from Baseline over Time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | | 5 to 10 yes $(N=XX)$ | 5 to 10 years (N=XX) | 11 to 17 yes $(N=XX)$ | 11 to 17 years $(N=XX)$ | Overall (N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|---|---|---|
| | | Observed | % Change<br>from | Observed | % Change<br>from | Observed | % Change<br>from |
| Visit | Statistics | value | baseline | value | baseline | value | baseline |
| XXX | ជ | XX | | XX | | XX | |
| | Mean | XX.X | | XX.XX | | XX.X | |
| | SD | XX.XX | | XX.XX | | XX.XX | |
| | Minimum | XX | | X | | XX | |
| | Median | XX.X | | XX.XX | | XX.X | |
| | Maximum | XX | | X | | XX | |
| | 25th percentile | XX.XX | | XX.XX | | XX.XX | |
| | 75th percentile | XX.X | | XX.X | | XX.X | |
| XXX | и | XX | XX | XX | × | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.X | XX.XX | ××.× |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX | ×× | ×× | ×× | ×× | ×× |
| | Median | x.xx | XX.X | XX.X | XX.X | XX.XX | ××.× |
| | Maximum | XX | ×× | ×× | ×× | ×× | ×× |
| | 25th percentile | XX.XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X |
| | 75th percentile | XX.X | XX.X | XX.X | XX.X | XX.XX | ××.× |

Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

At each time point, only subjects with a value at both baseline and that time point are included in the change from baseline column.

N = the number of subjects in the analysis set who receive the respective treatment/dose. n = the number of subjects with a measurement. Source: Listing 16.2.17.2 and 16.2.17.3

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits and parameters (right CIMT, left CIMT, FWD baseline diameter, FWD maximum diameter, %FMD).


Table 14.3.13.1 Summary of Palatability over Time (Safety Analysis Set)

| | | | 5 to 10 | 11 to 17 | |
|---|---|---|---|---|---|
| Visit | | Result | years<br>(N=XX) | years<br>(N=XX) | Overall (N=XX) |
| XXX | Able to swallow capsule? | Z<br>O<br>S | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Missing | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Total | (XX.X) | XX (XX.X) | XX (XX.X) |
| | If no, food media used? | Mashed banana | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Apple Sauce | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Missing | (XX.X) | XX (XX.X) | XX (XX.X) |
| | First occasion subject used this food media? | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | No | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Missing | (XX.X) | XX (XX.X) | XX (XX.X) |
| | If yes, palatability rate? | Super bad | (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Bad | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Maybe Good or Maybe | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | Bad | | | |
| | | Good | XX (XX.X) | XX (XX.X) | (X.XX) XX |
| | | Super Good | XX (XX.X) | XX (XX.X) | (XXXX) |
| | | Missing | XX (XX.X) | XX (XX.X) | (XXXX) |

N = the number of Source: Listing 16.2.17.4

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS

NOTES: Repeat for all visits.


Table 14.3.13.1 Summary of Palatability over Time (Safety Analysis Set)

| Visit | | Result | 5 to 10<br>years<br>(N=XX) | 11 to 17<br>years<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| | Parent/Guardian interpretation of child's reaction / | Pleasant | (X.XX) | (XX.X) | (X.XX) XX |
| | racial expression | Unpleasant<br>Not sure | XX (XX.X)<br>XX (XX.X) | xx (xx.x) xx x | XX (XX.X)<br>XX (XX.X) |
| | Parent/Guardian Question: Do you sometimes have problems giving the medication to your child because he/she refuses to take it or throws up immediately after taking | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | it? | No<br>Missing | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| | Parent/Guardian Question: Do you sometimes have problems in giving the dietary supplement to your child because he/she refuses to take it or throws up immediately after | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | taking it? | No<br>Missing | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| XXX | etc | | | | |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100. Source: Listing 16.2.17.4

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01. SAS

NOTES: Repeat for all visits.

Table 14.3.14.1 Summary of Diet Compliance over Time (Safety Analysis Set)

| | 1 | o to in years | TI CO II Years | OVCERTE |
|---|---|---|---|---|
| | Visit | (N=XX) | (N=XX) | (X=XX) |
| Subjects compliant with low-fat diet, n(%) | Baseline | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 36 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 44 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 56 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | XX (XX.X) | (XX.X) XX | XX (XX.X) |
| | Week 92 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | XX (XX.X) | XX (XX.X) | (XX.X) |
| Subjects compliant with their low-fat diet [1] | Efficacy phase | XX (XX.X) | (XXXX) XX | XX (XX.X) |
| | Safety phase (up to Week 56): | (X.XX) XX | (X.XX) XX | XX (XX.X) |
| | Safety phase (up to Week 104): | XX (XX.X) | XX (XX.X) | XX (XX.X) |

N = the number of subjects in the analysis set. n = the number of subjects meeting the criterion. (%) = n/N\*100. [1] Compliance is defined as at least 80% of compliance with the low-fat diet during the respective study phase. Source: Listing 16.2.19.1

DATE OF EXTRACTION:XXXXXXXX

TIME OF RUN: XX:XX:XX

DATE OF RUN:XXXXXXXX

PROGRAM NAME: T XXX 01.SAS

Table 14.3.14.1 Summary of Diet Compliance over Time (Safety Analysis Set)

| | | 5 to 10 years | 11 to 17 years | Overall |
|---|---|---|---|---|
| | Visit | (N=XX) | (N=XX) | (N=XX) |
| Subjects compliant with dietary supplement regimen, n(%) | Baseline | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 8 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 12 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 16 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 20 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 24 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 28 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 32 | XX (XX.X) | XX (XX.X) | (XX.X) |
| | Week 36 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 40 | XX (XX.X) | XX (XX.X) | (XX.X) |
| | Week 44 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 48 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 52 | XX (XX.X) | XX (XX.X) | (XXXX) XX |
| | Week 56 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 68 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 80 | XX (XX.X) | XX (XX.X) | (XX.X) |
| | Week 92 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | EOT / Week 104 | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Subjects compliant with their dietary supplement regimen | Efficacy phase | (X.XX) XX | (X.XX) XX | (XX.X) |
| 7 + 1 | Safety phase (up to | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Week 104): | XX (XX.X) | XX (XX.X) | XX (XX.X) |

N= the number of subjects in the analysis set. n= the number of subjects meeting the criterion. (%) = n/N\*100. [1] Compliance is defined as at least 80% of compliance with the low-fat diet during the respective study phase. Source: Listing 16.2.19.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: T\_XXX\_01.SAS


Listing 16.2.1.1 Subject Completions and Withdrawals (Enrolled Set)

<sup>[1]</sup> Study day is relative to the date of first administration of study drug (Day 0).

[2] Study duration is the number of days between first visit and the date of completion/withdrawal, derived as: (date of completion/withdrawal - date of first visit + 1).

[3] Treatment duration is the number of days between first administration of study treatment in period 1 and the date of completion/withdrawal, derived as: (date of completion/withdrawal - date of first administration of study treatment in period 1 + 1).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Listing 16.2.2.1 Eligibility (Enrolled Set)

| toerdus/etts | | Were all<br>inclusion/exclusion | Toclesion/Exclusion | Informed | 80<br>80<br>40 | Protogol |
|---|---|---|---|---|---|---|
| number | Age group | criteria met? | criteria not met | given? | given? | Version |
| XXX/XXX | 5 to 10 years | Y @ S | | Yes/No | Yes/No | XXX |
| XXX/XXX | 11 to 17 years | No | IXXX, EXXX | Yes/No | Yes/No | XXX |
| XXX/XXX | 5 to 10 years | Yes | | Yes/No | Yes/No | XXX |

Criterion numbers prefixed by I are inclusion criteria, those prefixed by E are exclusion criteria.

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS
Listing 16.2.2. Protocol Deviations (Safety Analysis Set)

| Site/Subject<br>number | Age Group | Major/Minor<br>[2] | Start date (Study day [1]) | En<br>(S) | End date<br>(Study day<br>[1]) | | Deviation category (I/II/III) | Deviation details | Action<br>Taken |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 5 to 10 years | Major /<br>Minor | DDMONYYYY (XX) DDMONYYYY (XX) | MX) DD | () XXXXNOW | | XXXXXXXX<br>XXXXXXXX | ××××××××× | XXXXXXXXX |
| XXX/XXX | 11 to 17 years | Major /<br>Minor | DDMONYYYY (XX) | | DDMONYYYY (XX) | | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | XXXXXXXX | XXXXXXXXX |
| XXX/XXX | 11 to 17 years | Major /<br>Minor | DDMONYYYY (XX) | | DDMONYYYY (XX) | (XX | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXXX | XXXXXXXXX | XXXXXXXXX |

[1] Study day is relative to the date of first administration of study drug (Day 0).
[2] Major protocol deviations are a subset of protocol deviations that may significantly impact the completeness, accuracy and/or reliability of the study data or that may significantly affect a subject's rights, safety or well-being.

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME:L XXX 01.SAS Repeat protocol deviation listing for all protocol deviations regarding visits and assessments due to the COVID-19 pandemic. Add subheader accordingly to identify the PDs regarding the COVID-19 pandemic. NOTES:

SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Listing 16.2.2.3 COVID-19 Protocol Deviations (Safety Analysis Set)

Repeat of Listing 16.2.2.2

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as per Listing 16.2.2.2

Listing 16.2.3.1 Analysis Sets (Enrolled Set)

| +20-412/0+12 | | | | Fligible 1 | Eligible for analysis set? | ٠ | Beason for |
|---|---|---|---|---|---|---|---|
| number | Age group | Age/Sex/Race | Safety [1] | FAS [2] | CAS [3] | PPS [4] | exclusion |
| XXX/XXX | 5 to 10 years | XX/Female/White | Yes/No | Yes/No | Yes/No | Yes/No | XXXXXXXXX |
| XXX/XXX | 11 to 17 years | XX/Female/White | Yes/No | Yes/No | Yes/No | Yes/No | XXXXXXXXXX |
| XXX/XXX | 11 to 17 years | XX/Female/White | Yes/No | Yes/No | Yes/No | Yes/No | XXXXXXXXXX |

[1] The Safety Analysis Set includes all subjects who are treated with at least one dose of the IMP.
[2] The Full Analysis Set includes all subjects who receive at least one dose of the IMP and who have a baseline and at least one postbaseline measurement of LDL-C.

[3] The Completers Analysis Set includes all subjects from the FAS who have not discontinued the Efficacy Phase (up to Week 24) of the study

[4] The Per Protocol Set includes all patients from the FAS who reasonably adhere to all protocol conditions (i.e. who have met the eligibility criteria and receive planned study medication without important protocol deviations considered to have a serious impact on the efficacy results within the Efficacy Phase of the trial). early irrespective of the reason for discontinuation.

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L XXX 01.SAS

Listing 16.2.4.1 Demography (Safety Analysis Set)

| Site/Subject<br>number | Age group | Age<br>(years) | Age<br>(months) | ν<br>κ<br>κ | Race | Ethnicity | Height (cm) | Weight<br>(kg) | Body mass<br>index<br>(kg/m^2)<br>[1] |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 5 to 10 years | XXX | ××× | Male | XXXXXXXXX | XXXXXXXXX | XXX | XX.X | XX.X |
| XXX/XXX | 11 to 17 | XXX | XXX | Female | XXXXXXXXXX | XXXXXXXXXX | XXX | x.x | XX.X |
| | years | | | | | | | | |

Height and weight recorded at Screening. [1] Body mass index (BMI) is calculated as (weight (kg)/height (m)^2). [2] BSA (m^2) =  $\sqrt{\{\text{height}(cm) \ x \ weight(kg)\}}$  / 3600] [Mosteller formula] [3] z scores and percentiles calculated using the WHO growth reference indicators for children aged 5 to 19 years.

DATE OF EXTRACTION:XXXXXXXX

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Listing 16.2.4.1 Demography (Safety Analysis Set)

| Site/Subject | Body surface area | Height z score | | BMI z score | |
|---|---|---|---|---|---|
| number | [2] | [3] | Height percentile [3] | [3] | BMI percentile [3] |
| XXX/XXX | XX.X | XX.X | XX.X | XX.X | XX.X |
| XXX/XXX | ×.×.× | XX.X | XX.X | XX.X | xx.x |
| Height and weight recorded at Screening. [1] Body mass index (BMI) is calculated as (weight (kg)/height (m)^2). [2] BSA (m^2) = $\sqrt[\Lambda]{\text{height(cm) x weight(kg)}}$ / 3600] [Mosteller formula] [3] z scores and percentiles calculated using the WHO growth reference indi | t Screening. calculated as (weight ( m) x weight(kg)} / 3600] calculated using the WH | kg)/height (m)^2).<br>[Mosteller form<br>O growth reference | tht and weight recorded at Screening. Body mass index (BMI) is calculated as (weight (kg)/height (m)^2). BSA (m^2) = $\sqrt{\{\text{height}(cm) \times \text{weight}(kg)\}}$ / 3600] [Mosteller formula] z scores and percentiles calculated using the WHO growth reference indicators for children aged 5 to 19 years. | ged 5 to 19 years. | |
| PROGRAM NAME:L_XXX_01.SAS | DATE OF RUN:XXXXXXXX | TIME OF RUN: XX:XX:XX | X:XX:XX DATE OF EXTRACTION:XXXXXXXX | XXXXXXXXX | |

Listing 16.2.4.2 Diagnosis of HoFH (Safety Analysis Set)

| Site/Subject<br>number | Age/Sex/Race | Age group | Duration<br>of<br>diagnosis<br>(months) | Genetic<br>confirmation<br>of 2 mutant<br>alleles? | Type of<br>mutant<br>allele | LDL-C<br>receptor<br>function | Untreated LDL- C>500mg/dL or treated LDL- C≥300mg/dL? | Cutaneous<br>or tendon<br>xanthoma<br>before age<br>10 years? | Untreated<br>LDL-C level<br>consistent<br>with HoFH<br>on both<br>parents? |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | XX/Female/White | 5 to 10 | XX.X | Yes/No | XXXXXXXXX | XXXXX | Yes/No | Yes/No | Yes/No |
| XXX/XXX | XX/Female/White | years<br>11 to 17<br>Years | × | Yes/No | XXXXXXXXX | XXXXX | Yes/No | Yes/No | Yes/No |

Duration of diagnosis (months) = 12\*[(date of baseline - date of HoFH diagnosis)+1]/365.25

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS 

Listing 16.2.4.3 Medical History (Safety Analysis Set)

| | | | Reported term | | |
|---|---|---|---|---|---|
| Site/Subject | | | System organ class | | |
| number | Age/Sex/Race | Age Group | Preferred term | Start date | Stop date |
| XXX/XXX | XX/Female/White | 5 to 10 years | XXXXXXXX | DDMONYYYY | DDMONYYYY |
| | | | XXXXXXXX | | |
| | | | XXXXXXXX | | |
| XXX/XXX | XX/Female/White | 11 to 17 years | XXXXXXXX | DDMONYYYY | Ongoing |
| | | | XXXXXXXX | | |
| | | | XXXXXXXX | | |

Only subjects with medical history are listed. Medical history events were coded using the MedDRA Dictionary, version  $xx.\,x.\,x$ 

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Listing 16.2.4.4 Cardiovascular Medical History (Safety Analysis Set)

Repeat of Listing 16.2.4.3

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as per Listing 16.2.4.3 (as applicable)


Listing 16.2.4.5 Prior/Run-in/Concomitant Medications (Safety Analysis Set)

| Site/Subject<br>number | Age Group | Age/Sex/Race | Timing | Reported name Medication class Standardised medication name | Do<br>Se | Dose<br>unit | Frequency | Route |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 11 to 17 | XX/Female/White | P/R/C | XXXXXXX | XXX | XXX | XXX | XXX |
| | years | | | XXXXXXXX | | | | |
| xxx/xxx | 5 to 10 | XX/Female/White | | XXXXXXXX | XXX | XXX | XXX | XXX |
| | 7 | | | XXXXXXXX | | | | |

Only subjects who have recorded any medications during the study are listed.

Medications were coded using WHO Drug Dictionary, version xxx.

[1] Timing of Medication: P = Prior; R = 'Run-in'; C = Concomitant

[2] Study day is relative to the date of first administration of study drug (Day 0).

Prior medications / procedures are defined as those that started and ended prior to the enrolment date visit (visit 2) (i.e. start of the 'run-in period').

Concomitant medications / procedures are defined as those that are ongoing at the time of first administration of study treatment or started on or after the time of first administration of study treatment or started prior to the end / last dose of study treatment. If medication / procedure dates are incomplete and it is not clear whether the medication / procedure was concomitant, it will be assumed to be concomitant. Run-in period' medications / procedures are defined as those that are ongoing at the time of starting the 'run-in' period (i.e. Visit 2) or started after the start of the 'run-in' period, but before the time of first administration of study treatment.

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

If a medication is defined as prior medication only then timing = P. If a medication is defined as run-in medication then timing = R. If a medication is defined as concomitant medication then timing = C. NOTES:

If a medication is taken during run-in and concomitantly then timing = C.

Listing 16.2.4.5 Prior/Run-in/Concomitant Medications (Safety Analysis Set)

| | | | | Reported name<br>Medication class | Date (Stud | ly day [2]) | |
|---|---|---|---|---|---|---|---|
| Site/Subject<br>number | Age Group | Age/Sex/Race | Timing | Standardised medication name | Start of End of medication | Start of End of medication Indication | Indication |
| XXX/XXX | 11 to 17 | XX/Female/White | P/R/C | XXXXXXX | DDMONYYYY | DDMONYYYY | XXXXXXXXX |
| | years | | | XXXXXXXX | (XX) | (XX) | |
| XXX/XXX | 5 to 10 years | XX/Female/White | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY (XX) | Ongoing | XXXXXXXXX |
| | | | | AAAAAAAA | | | |

Only subjects who have recorded any medications during the study are listed.

Medications were coded using WHO Drug Dictionary, version xxx.

Prior medications / procedures are defined as those that started and ended prior to the enrolment date visit (visit 2) (i.e. start of the [1] Timing of Medication: P = Prior; R = 'Run-in'; C = Concomitant [2] Study day is relative to the date of first administration of study drug (Day 0).

Run-in period' medications / procedures are defined as those that are ongoing at the time of starting the 'run-in' period (i.e. Visit 2) or 'run-in period').

Concomitant medications / procedures are defined as those that are ongoing at the time of first administration of study treatment or started procedure dates are incomplete and it is not clear whether the medication / procedure was concomitant, it will be assumed to be concomitant. on or after the time of first administration of study treatment or started prior to the end / last dose of study treatment. If medication / started after the start of the 'run-in' period, but before the time of first administration of study treatment.

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L XXX 01.SAS

If a medication is taken during run-in and concomitantly then timing = C. If a medication is defined as concomitant medication then timing = C. If a medication is defined as prior medication only then timing = P. If a medication is defined as run-in medication then timing = R. NOTES:


Listing 16.2.4.6 Lipid-lowering-therapy (LLT) Medications (Safety Analysis Set)

Repeat of Listing 16.2.4.5

Only subjects who have recorded any medications during the study are listed. Medications were coded using WHO Drug Dictionary, version xxx. Procedures were coded using the MedDRA Dictionary, version xx.x.

[1] <LLTMDEF> [2] Study day is relative to the date of first administration of study drug (Day 0).

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as per Listing 16.2.4.5 (as applicable)

Listing 16.2.4.7 Prior/Run-in/Concomitant Procedures (Safety Analysis Set)

| | | | | | Reported name | | Date (Stud | y day [2]) |
|---|---|---|---|---|---|---|---|---|
| Site/Subject<br>number | Age Group | Age/Sex/Race | Study<br>Phase | Timing | Procedure Category<br>Indication | Frequency | Start of End of procedure | End of<br>procedure |
| XXX/XXX | 5 to 10<br>years | XX/Female/White | Efficacy<br>/ Safety | P / R / C | XXXXXXXX | XXX | DDMONYYYY (XX) | DDMONYYYY<br>(XX) |
| xxx/xxx | 11 to 17<br>Years | XX/Female/White | | | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXX | ××× | DDMONYYYY<br>(XX) | Ongoing |

Only subjects who have recorded any procedures during the study are listed. Procedures were coded using the MedDRA Dictionary, version xx.x.

'run-in period').

[1] Timing of Procedure: P = Prior; R = 'Run-in'; C = Concomitant [2] Study day is relative to the date of first administration of study drug (Day 0).

Prior medications / procedures are defined as those that started and ended prior to the enrolment date visit (visit 2) (i.e. start of the

Concomitant medications / procedures are defined as those that are ongoing at the time of first administration of study treatment or started procedure dates are incomplete and it is not clear whether the medication / procedure was concomitant, it will be assumed to be concomitant. on or after the time of first administration of study treatment or started prior to the end / last dose of study treatment. If medication / Run-in period' medications / procedures are defined as those that are ongoing at the time of starting the 'run-in' period (i.e. Visit 2) or started after the start of the 'run-in' period, but before the time of first administration of study treatment.

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L XXX 01.SAS

Listing 16.2.5.1 IMP Administration (Safety Analysis Set)

| | | | | | | Daily Dose (Increase | |
|---|---|---|---|---|---|---|---|
| | | | | Date of | Strength and<br>Number of | (I),<br>Decrease | |
| | | | | Dispensing | | (D), | |
| Site/Subject | | | Study Drug | (Study day | Dispensed | Unchanged | Reason Dose |
| number | Age Group | Visit | Administration* | [1]) | [2] | (U)) (mg) ** | Increased/Decreased/Unchanged |
| XXX/XXX | 11 to 17 | XXX | Yes (F) | DDMONYYYY | XXXXXXXXXX | XXX | XXXXXXXXX |
| | years | | | (XX) | n=xx | | |
| XXX/XXX | 5 to 10 | XXX | Yes | DDMONYYYY | XXXXXXXXXX | XXX | XXXXXXXXX |
| | years | | | (XX) | u=xx | (I) (MID) | |
| | | | | | | (Maint) | |


Listing 16.2.5.1 IMP Administration (Safety Analysis Set)

| Site/Subject Age<br>number Grou | Age<br>Group | Visit | Were<br>Capsules<br>Visit Returned? | Strength and number of capsules returned | Has<br>subject<br>complied<br>with IMP<br>dosing as<br>per<br>protocol? | Has<br>subject<br>complied<br>with IMP<br>dosing as<br>per<br>protocol? Reason missed doses | Number missed | Number missed Consecutively or intermittently |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX<br>XXX/XXX | 11 to 17 XXX<br>years<br>5 to 10 XXX<br>years | X XX X | N N K | XXXXXXXXX<br>n=xx | Yes/No<br>Yes/No | ××××××××××××××××××××××××××××××××××××××× | × | XXXXXXXXX |

[1] Study day is relative to the date of first administration of study drug (Day 0).
[2] Capsules are dispensed as 2mg, 5mg, 10mg and 20mg
[3] Derived total number of weeks exposure to study medication = [(date of last dose - date of first dose)+1]/7
[4] Derived total exposure (mg/day) to study medication = ([number of doses received\*treatment dose(mg)] / number of days exposed
[5] Derived total number of weeks of exposure to maintenance dose = [(date of last dose - date when maintenance dose is reached)+1]/7.
\*F denotes date of first dose (i.e. date of first study drug administration)

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Listing 16.2.5.1 IMP Administration (Safety Analysis Set)

| | | | | | Date (Study Day [1]) | ly Day [1]) | Derived | | Derived | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | total | Derived<br>total | total<br>number of | | |
| | | | | | | | weeks | exposure | weeks | Time | Time |
| | | | Was the | | | | exposure | (mg/day) | exposure | (weeks) | (weeks) to |
| Site/Subjec Age | Age | | treatment | Reason for | Start of | End of | to study | to study | to | to dose | dose |
| 4 | Grou | Visi | Visi interrupted | interruptio | interruptio | interruptio | medicatio | medicatio | maintenanc | reductio | interruptio |
| number | Q | t | ٠. | и | и | и | n [3] | n [4] | e dose [5] | п | и |
| XXX/XXX | 11 | XXX | | | | | XXX | XXX | XXX | XXX | XXX |
| | to | | | | | | | | | | |
| | 7 ( | | | | | | | | | | |
| | / T | | | | | | | | | | |
| | year | | | | | | | | | | |
| | Ø | | | | | | | | | | |
| XXX/XXX | 5<br>to | XXX | Yes/No | XXXXXXXXXX | DDMONYYYY | DDMONYYYY | XXX | XXX | XXX | XXX | XXX |
| | 10 | | | | (XX) | (XX) | | | | | |
| | Vear | | | | | | | | | | |
| | 1<br>5<br>7<br>8 | | | | | | | | | | |
| | 0 | | | | | | | | | | |

DATE OF EXTRACTION: XXXXXXXX

<sup>[1]</sup> Study day is relative to the date of first administration of study drug (Day 0).

[2] Capsules are dispensed as 2mg, 5mg, 10mg and 20mg

[3] Derived total number of weeks exposure to study medication = [(date of last dose - date of first dose)+1]/7

[4] Derived total exposure (mg/day) to study medication = ([number of doses received\*treatment dose(mg)] / number of days exposed

[5] Derived total number of weeks of exposure to maintenance dose = [(date of last dose - date when maintenance dose is reached)+1]/7.

\*F denotes date of first dose (i.e. date of first study drug administration)

TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L XXX 01.SAS

Listing 16.2.6.1 Lipoprotein Apheresis (LA) History (Safety Analysis Set)

| Site/Subject Age<br>number Grou | Age<br>Group | Age/Sex/Race | Receiving / Received (i.e.previous 60 days) LA treatment? | Date LA<br>started [1] | Receive LA during run-in<br>period and through Week<br>24? | Planned frequency<br>of LA treatments |
|---|---|---|---|---|---|---|
| XXX/XXX | 11 to 17 | XX/Female/White | Yes/No | DDMONYYYY | Yes/No | XXXXXXXXXX |
| XXX/XXX | years<br>5 to 10<br>years | XX/Female/White | Yes/No | (XX)<br>DDMONYYYY<br>(XX) | Yes/No | Other: XXXXXXXXXX |

<sup>[1]</sup> Study day is relative to the date of first administration of study drug (Day 0).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Listing 16.2.6.2 Lipoprotein Apheresis (LA) Treatment (Safety Analysis Set)

| Days to<br>next LDL-C<br>assessment | ×× |
|---|---|
| Fasting<br>lipid<br>panel<br>local lab<br>sample<br>taken<br>before<br>scheduled<br>LA? | Yes/No |
| Fast lipi pane loce samg take Change befor to ConMeds? LA? | Yes/No |
| Days<br>since<br>previous<br>LA | × × |
| Scheduled /<br>Unscheduled | Scheduled / XX Unscheduled XX |
| Date of<br>LA [1] | DDMONYYYY (XX) |
| Received<br>LA<br>treatment<br>since<br>last<br>visit? | Yes/No |
| Visit | XXX<br>Run-in<br>weighted<br>average* |
| Study<br>Phase | Efficacy<br>/ Safety |
| Age/Sex/Race | XX/Female/White Efficacy / Safety |
| Age<br>Group | 11 to<br>17<br>years |
| Site/Subject Age<br>number Grou | XXX/XXX |

<sup>[1]</sup> Study day is relative to the date of first administration of study drug (Day 0).  $\star$  Weighted averaged regimen during run-in.

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES:

Repeat for all visits. Study Phase: Efficacy - up to (and including) Week 24; Safety - up to (and including) Week 104. After run-in, add Run-in weighted average.

Listing 16.2.7.1 Adverse Events (Enrolled Set)

| | | | | t + | Date (Study | Date (Study day [2]) Time [3] | Time | |
|---|---|---|---|---|---|---|---|---|
| | | | | reported term<br>System organ<br>class | | | onset | Duration |
| Site/Subject | | | TE? | Preferred | | | [5] | [2] |
| number | Age Group | Age/Sex/Race | [1] | term | Start | End | (days) | (d:hh:mm) |
| XXX/XXX | 5 to 10 | XX/Female/White | Yes/No | XXXXXXX | DDMONYYYY (XX) | DDMONYYYY (XX) | XXX | d:hh:mm |
| | years | | | XXXXXXXX<br>XXXXXXXX G | нн:мм | нн:мм | | |
| XXX/XXX | 11 to 17 | XX/Female/White | Yes/No | XXXXXXXX | DDMONYYYY (XX) | Ongoing | XXX | UK |
| | 7 (25) | | | ×××××××× | 1 | | | |

G = Gastrointestinal event, H = Hepatic event.

Only subjects with any adverse event are listed.

Adverse events were coded using the MedDRA Dictionary, version xx.x.

[1] TE = Treatment-emergent adverse event defined as an adverse event that started after administration of study drug. [2] Study day is relative to the date of first administration of study drug (Day 0).
[3] 24-hour clock (HH:MM).
[4] Time from date of first administration of study drug to onset of adverse event.
[5] For missing or partial dates and times, not calculated and is reported as unknown (UK).

DATE OF RUN: XXXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Listing can go over multiple pages. Data for a given subject will appear on the consecutive page

Listing 16.2.7.1 Adverse Events (Enrolled Set)

| Site/Subject<br>number | | Age Group Age/Sex/Race | TE?<br>[1] | Reported term<br>System<br>organ class<br>Preferred term | Reported term System organ class Was adverse Preferred term event serious? | Serious<br>Criteria | Adverse Event of Special<br>Interest? If yes, reason | Severity |
|---|---|---|---|---|---|---|---|---|
| xxx/xxx | 5 to 10<br>years | XX/Female/White Yes/No | Yes/No | XXXXXXXX | S<br>O | XXXXXXXXX | Yes, XXXXXXXXX | XXX |
| xxx/xxx | 11 to 17<br>years | XX/Female/White | Yes/No | XXXXXXXX | ON | XXXXXXXXX | ON | XXX |

Only subjects with any adverse event are listed.

Adverse events were coded using the MedDRA Dictionary, version xx.x.

[1] TE = Treatment-emergent adverse event defined as an adverse event that started after administration of study drug (Day 0).

[2] Study day is relative to the date of first administration of study drug (Day 0).

[3] 24-hour clock (HH:MM).

[4] Time from date of first administration of study drug to onset of adverse event.

[5] For missing or partial dates and times, not calculated and is reported as unknown (UK).

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS Listing can go over multiple pages. Data for a given subject will appear on the consecutive page NOTES:


Listing 16.2.7.1 Adverse Events (Enrolled Set)

| | | | | Reported<br>term | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | System<br>ordan class | Relations. | Action | | | |
| | | | | | to | with | Other | Was a concomitant | |
| Site/Subject Age | Age | | TE? | Preferred | study | study | action | treatment given for this | |
| number | Group | Age/Sex/Race | [1] | term | treatment | treatment | taken | adverse event? | Outcome |
| XXX/XXX | 5 to 10<br>years | XX/Female/White | Yes/No | XXXXXXX | ××× | XXX | ××× | K es | XXX |
| XXX/XXX | 11 to<br>17 | XX/Female/White | Yes/No | XXXXXXXX<br>XXXXXXXX | ××× | XXX | XXX | No | XXX |
| | years | | | XXXXXXX | | | | | |

Only subjects with any adverse event are listed.

Adverse events were coded using the MedDRA Dictionary, version xx.x.

[1] TE = Treatment-emergent adverse event defined as an adverse event that started after administration of study drug.

[2] Study day is relative to the date of first administration of study drug (Day 0).

[3] 24-hour clock (HH:MM).

[4] Time from date of first administration of study drug to onset of adverse event.

[5] For missing or partial dates and times, not calculated and is reported as unknown (UK).

PROGRAM NAME: L\_XXX\_01.SAS

DATE OF RUN:XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX

NOTES: Listing can go over multiple pages. Data for a given subject will appear on the consecutive page

SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Listing 16.2.7.2 Serious Adverse Events (Enrolled Set)

Repeat of Listing 16.2.7.1 but just for Serious AEs

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as Listing 16.2.7.1 (as appropriate)


Listing 16.2.8.1 Serum Clinical Chemistry (Fasting Lipid Panel) Values

(Safety Analysis Set)

Central lab Sex

Unit

Local lab

| Normal range | Normal range |
|---|---|
| Sex | × |
| Age range | Age range |
| Unit | Unit |
| Normal range | Normal range |
| Sex | × oo |
| Age range | Age range |
| Site | in the state of th |
| Unit Site | Onit |
| Parameter | Parameter |

DATE OF EXTRACTION: XXXXXXXX

TIME OF RUN: XX:XX:XX

DATE OF RUN: XXXXXXXXX

PROGRAM NAME: L\_XXX\_01.SAS

Listing 16.2.8.1 Serum Clinical Chemistry (Fasting Lipid Panel) Values (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| Local Lab | % Change from baseline | UCS H |
|-----------|-------------------------------|--------------------------------|
| | Observed | XX.X B NCS H |
| | Time<br>[2] | HH: MM |
| Date of | collection<br>(Study day [1]) | DDMONYYYY (XX) |
| | Lomitapide Dose (mg) | 2 / 5 / 10 / 20 / 30 / 40 / 60 |
| | Visit | ××× |
| | Age/Sex/Race | XX/Female/White |
| | Age Group | 5 to 10 years |
| | Site/Subject<br>number | XXX/XXX |

CS = clinically significant, NCS = not clinically significant. H = High, L = Low. \* = Maximum post-baseline value. B = Paseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject

receiving study treatment in the Efficacy Phase (Visit 4). [1] Study day is relative to the date of first administration of study drug (Day 0). [2] 24-hour clock (HH:MM).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Unscheduled assessments will be included in the listing and flagged as such in the visit column. NOTES:

The listing may go over multiple pages to capture all data. Repeat for all visits and all parameters (i.e. LDL-C, Non-HDL-C, TC, VLDL-C, apo B, TG, Lp(a) in this order).

Listing 16.2.8.1 Serum Clinical Chemistry (Fasting Lipid Panel) Values (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| İ | | | |
|---|---|---|---|
| Central Lab | % Change<br>from<br>baseline | | XX. X |
| Centr | Change<br>from<br>baseline | | ×. ×× |
| Central<br>lab | Observed | HH:MM XX.X B NCS | ×. ×. |
| | Time<br>[2] | HH: MM | нн:мм |
| Date of | ion<br>lay | DDMONYYYY (XX) | DDMONYYYY (XX) |
| | .t Lomitapide Dose (mg) | 2 / 5 / 10 / 20 / 40 / | 60<br>2 / 5 / 10 / 20 / 40 /<br>60 |
| | Visit | XXX | ××× |
| | Age/Sex/Race | XX/Female/White | |
| | Age Group | 5 to 10 | Years |
| | Site/Subject<br>number | XXX/XXX | |

CS = clinically significant, NCS = not clinically significant.

B = baseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

[1] Study day is relative to the date of first administration of study drug (Day 0). [2] 24-hour clock (HH:MM).

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Unscheduled assessments will be included in the listing and flagged as such in the visit column. NOTES:

The listing may go over multiple pages to capture all data. Repeat for all visits and all parameters (i.e. LDL-C, Non-HDL-C, TC, VLDL-C, apo B, TG, Lp(a) in this order).

## Amryt Pharma study no: APH-19

## SQN Clinical study no: OCH19003

Listing 16.2.8.2 Serum Clinical Chemistry (Metabolic Panel) Values

(Safety Analysis Set)

Local lab

| | Normal range |
|-----------|--------------|
| | Sex |
| LOCAL LAD | Age range |
| | Site |
| | Unit |
| | Parameter |

DATE OF EXTRACTION: XXXXXXXX

TIME OF RUN: XX:XX:XX

DATE OF RUN: XXXXXXXXX

PROGRAM NAME: L\_XXX\_01.SAS

Listing 16.2.8.2 Serum Clinical Chemistry (Metabolic Panel) Values (Safety Analysis Set)

Parameter: <Parameter (Unit)>

% Change baseline ××. from Local Lab baseline Change ××× XX.X B NCS H Observed ×××× HH: MM HH: MM Time [2] collection (Study day DDMONYYYY (XX) Date of [11] 2 / 5 / 10 / 20 / 40 / 60 Visit Lomitapide Dose (mg) XX/Female/White XXX Age/Sex/Race Age Group 11 to 17 years Site/Subject XXX/XXX number

CS = clinically significant, NCS = not clinically significant.

H = High, L = Low.

B = baseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

[1] Study day is relative to the date of first administration of study drug (Day 0). [2] 24-hour clock (HH:MM).

PROGRAM NAME: L\_XXX\_01.SAS

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXXX

Unscheduled assessments will be included in the listing and flagged as such in the visit column. The listing may go over multiple pages to capture all data. Repeat for all visits and all parameters. NOTES:

#### Amryt Pharma study no: APH-19

## SQN Clinical study no: OCH19003

Listing 16.2.8.3 Serum Clinical Chemistry (Liver Function Tests) Values

(Safety Analysis Set)

Parameter: <Parameter (Unit)>

Repeat of Listing 16.2.8.2

PROGRAM NAME: L\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX

NOTES:

Footnotes as per Listing 16.2.8.2 (as applicable) Add \*, ^, +, ! flags with footnote: [\*] = > 3 x ULN (ALP and AST) or > 1.5 x ULN (ALP and TBL). [^] = > 5 x ULN (ALT and AST) or > 2 x ULN (TBL). [+] = > 10 x ULN (ALT and AST). [!] = > 20 x ULN (ALT and AST).

## SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Listing 16.2.8.4 Serum Clinical Chemistry (Essential Fatty Acids) Values

(Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | Ì |
|-------------|--------------|
| | Normal range |
| Central lab | Sex |
| | Age range |
| | Unit |
| | Parameter |

DATE OF RUN:XXXXXXXXXX IIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Columns for site, age range and sex will be included in the final listing output if required.


Listing 16.2.8.4 Serum Clinical Chemistry (Essential Fatty Acids) Values (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| | | | | | Date of | | | Central Lab | |
|---|---|---|---|---|---|---|---|---|---|
| Site/Subject | | | | | collection (Study day | Time | | Change<br>from | % Change<br>from |
| number | Age Group | Age/Sex/Race | Visit | Lomitapide Dose (mg) | [1]) | [2] | Observed | baseline | baseline |
| XXX/XXX | 11 to 17<br>years | XX/Female/White | ×× | 2 / 5 / 10 / 20 / 40<br>/ 60 | DDMONYYYY<br>(XX) | HH: MM | HH:MM XX.X B NCS | | |
| | ı | | | | | HH:MM | xx.x | xx.x | ××.× |

CS = clinically significant, NCS = not clinically significant.

H = High, L = Low.

B = baseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).
[1] Study day is relative to the date of first administration of study drug (Day 0).
[2] 24-hour clock (HH:MM).

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Unscheduled assessments will be included in the listing and flagged as such in the visit column. The listing may go over multiple pages to capture all data. Repeat for all visits and all parameters. NOTES:


## SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Listing 16.2.8.5 Serum Clinical Chemistry (Fat Soluble Vitamin Levels) Values (Safety Analysis Set)

Parameter: <Parameter (Unit)>

Repeat of Listing 16.2.8.4

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as per Listing 16.2.8.4 (as applicable)


## SQN Clinical study no: OCH19003

Listing 16.2.8.6 Serum Clinical Chemistry (Hormones) Values

Amryt Pharma study no: APH-19

(Safety Analysis Set)

Parameter: <Parameter (Unit)>

Repeat of Listing 16.2.8.2

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

PROGRAM NAME: L\_XXX\_01.SAS DATE OF RUN: XXXXXXXXX

NOTES: Footnotes as per Listing 16.2.8.2 (as applicable)


## SQN Clinical study no: OCH19003

Amryt Pharma study no: APH-19

Listing 16.2.8.7 Serum Clinical Chemistry (Sex Hormones) Values

(Safety Analysis Set)

Parameter: <Parameter (Unit)>

Repeat of Listing 16.2.8.2

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as per Listing 16.2.8.2 (as applicable)


## SQN Clinical study no: OCH19003

Listing 16.2.8.8 Serum Clinical Chemistry (Serum Lipase) Values

Amryt Pharma study no: APH-19

(Safety Analysis Set)

Parameter: <Parameter (Unit)>

Repeat of Listing 16.2.8.2

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as per Listing 16.2.8.2 (as applicable)


## SQN Clinical study no: OCH19003

Listing 16.2.8.9 Serum Haematology Values

(Safety Analysis Set)

Amryt Pharma study no: APH-19

Parameter: <Parameter (Unit)>

Repeat of Listing 16.2.8.2

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as per Listing 16.2.8.2 (as applicable)


## SQN Clinical study no: OCH19003

Listing 16.2.8.10 Urinalysis Values (Safety Analysis Set)

Amryt Pharma study no: APH-19

Parameter: <Parameter (Unit)>

Repeat of Listing 16.2.8.2

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Footnotes as per Listing 16.2.8.2 (as applicable)


Listing 16.2.9.1 Vital Signs (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| Site/Subject<br>number | Age Group | Age/Sex/Race | Visit | Date of collection (Study day [1]) | Observed | Change from baseline | % Change from baseline |
|---|---|---|---|---|---|---|---|
| *XXX/XXX | 11 to 17 years | XX/Female/White | × ×<br>× × | DDMONYYYY (XX)<br>DDMONYYYY (XX) | XX.X B<br>XX.X Min | XX.X | XX.X |

 $<sup>\</sup>star$  = Subject just met inclusion criterion #3 of having a body weight  $\geq 15~\mathrm{kg}$ .

# Unscheduled assessments should be included in the listing and flagged as such in the visit column. NOTES:

Repeat for all visits. Parameters (i.e. weight, height, BMI, BSA, heart rate, respiration rate, SBP, DBP, body temp, BMI, height & The listing may go over multiple pages to capture all data. weight percentile, BMI, height & weight Z score).

B = baseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).

Min = Minimum Post Baseline Value, Max=Maximum Post Baseline Value, Last=Last Post Baseline Value (for height and weight parameters only). [1] Study day is relative to the date of first administration of study drug (Day 0)

DATE OF EXTRACTION: XXXXXXXX DATE OF RUN: XXXXXXXXX TIME OF RUN: XX:XX:XX PROGRAM NAME: L XXX 01.SAS
Listing 16.2.10.1 ECG Results (Safety Analysis Set)

| Site/Subject | | | Date of assessment | |
|---|---|---|---|---|
| number | Age Group | Visit | (Study day [1]) | Overall interpretation |
| XXX/XXX | 11 to 17 years | XXX | DDMONYYYY (XX) | Normal |
| XXX/XXX | 5 to 10 years | XXX | DDMONYYYY (XX) | Abnormal, NCS |
| XXX/XXX | 11 to 17 years | XXX | DDMONYYYY (XX) | Abnormal, CS |

CS = clinically significant, NCS = not clinically significant. [1] Study day is relative to the date of first administration of study drug (Day 0).

DATE OF RUN:XXXXXXXX

PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Unscheduled assessments will be included in the listing and flagged as such in the visit column.

DATE OF EXTRACTION:XXXXXXXX

TIME OF RUN: XX:XX:XX


Listing 16.2.11.1 Echocardiography Results (Safety Analysis Set)

| Site/Subject<br>number | Age<br>Group | Visit | Scan<br>Visit performed? | Date of assessment (Study day [1]) | Atherosclerosis and/or<br>aortic valve disease? | Thickening aortic valve leaflets New (N): Progression (P): | Thickening aortic Fusion of aortic valve leaflets valve leaflets New (N): Progression (P): Progression (P): | Thickening of aortic root New (N): Progression (P): |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 5 to 10 XXX<br>years | ×× | Yes/No | DDMONYYYY<br>(XX) | Yes / No / N/A | Yes / No / N/A<br>N: Yes/No<br>P: Yes/No | Yes / No / N/A<br>N: Yes/No<br>P: Yes/No | Yes / No / N/A<br>N: Yes/No<br>P: Yes/No |

[1] Study day is relative to the date of first administration of study drug (Day 0).

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Unscheduled assessments will be included in the listing and flagged as such in the visit column.

Listing 16.2.11.1 Echocardiography Results (Safety Analysis Set)

| aortic valve N): ession (P): n (Re): No / N/A s/No upravalvular / ascending | | | | | Flow acceleration / turbulence | | |
|---|---|---|---|---|---|---|---|
| New (N): Scan Progression (P): Age Group Visit performed? Region (Re): 5 to 10 XXX Yes/No Yes/No N: Yes/No P: Yes/No P: Yes/No P: Yes/No P: Yes/No P: Yes/No P: Yes/No P: Supravalvular / ascending | | | | | over aortic valve | Aortic valve | Coronary ostial narrowing / |
| Scan Progression (P): Age Group Visit performed? Region (Re): 5 to 10 XXX Yes/No Yes/No N: Yes/No P: Yes | | | | | New (N): | regurgitation | flow disturbances |
| Age Group Visit performed? Region (Re): 5 to 10 XXX Yes/No Yes/No N: Yes/No P: Yes/No Re: Supravalvular / ascending | Site/Subject | | | Scan | Progression (P): | New (N): | New (N): |
| 5 to 10 XXX Yes/No Yes / No / N/A years N: Yes/No P: Yes/No Re: Supravalvular / ascending | number | Age Group | Visit | performed? | Region (Re): | Progression (P): | Progression (P): |
| 5 to 10 XXX Yes/No Yes / No / N/A years N: Yes/No P: Yes/No Re: Supravalvular / ascending | | | | | | | |
| N: Yes/No<br>P: Yes/No<br>Re: Supravalvular / ascending | XXX/XXX | 5 to 10 | XXX | Yes/No | Yes / No / N/A | Yes / No / N/A | Yes / No / N/A |
| P:<br>valvular / ascending | | years | | | N: Yes/No | N: Yes/No | N: Yes/No |
| Re: Supravalvular / ascending | | | | | P: Yes/No | P: Yes/No | P: Yes/No |
| « طبحات<br>م | | | | | Re: Supravalvular / ascending | | |
| 53435 | | | | | aorta | | |

[1] Study day is relative to the date of first administration of study drug (Day 0).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Unscheduled assessments will be included in the listing and flagged as such in the visit column.


Listing 16.2.11.1 Echocardiography Results (Safety Analysis Set)

| Other relevant<br>findings | Yes/No<br>Yes: XXXXXXXXX |
|---|---|
| <pre>Impairment of left ventricular function New (N): Progression (P):</pre> | Yes / No / N/A<br>N: Yes/No<br>P: Yes/No |
| Left ventricular hypertrophy New (N): Progression (P): | Yes / No / N/A<br>N: Yes/No<br>P: Yes/No |
| Ventricular<br>findings | Yes / No / N/A |
| Scan<br>Visit performed? | Yes/No |
| Visit | ××× |
| Age Group | 5 to 10<br>years |
| Site/Subject<br>number | XXX/XXX |

[1] Study day is relative to the date of first administration of study drug (Day 0).

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Unscheduled assessments will be included in the listing and flagged as such in the visit column. NOTES:

Listing 16.2.12.1 Lipid Accumulation in the Liver Results (Safety Analysis Set)

| Site/Subject Age<br>number Grou | Age<br>Group | Visit | Age NMR Scan<br>Group Visit performed? | Reason not<br>performed? | Date of scan (Study day [1]) | Ultrasound<br>Scan<br>performed? | Reason not<br>performed? | Date of scan (Study day [1]) | Result | Change<br>from<br>Result baseline | % Change<br>from<br>baseline |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 11 to<br>17 | ××× | Yes/No | | DDMONYYYY (XX) | Yes/No | | DDMONYYYY (XX) | XXX | XXX | XXX |
| XXX/XXX | years<br>5 to<br>10<br>years | × | Yes/No | XXXXXXXXX | DDMONYYYY<br>(XX) | Yes/No | XXXXXXXX | | | | |

[1] Study day is relative to the date of first administration of study drug (Day 0).

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Unscheduled assessments will be included in the listing and flagged as such in the visit column.

Listing 16.2.13.1 Physical Examination (Safety Analysis Set)

| Date of examination (Study day Body Physical Examination [1]) System Findings Comments | DDMONYYYY XXXXXXXXXX Normal / Abnormal / Not XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|
| Date of examinati. Reason not (Study da performed? [1]) | DDMONYYYY (XX) XXXXXXXXXX DDMONYYYY (XX) |
| | М - П - |
| Assessment<br>Visit performed? | X Yes/No<br>X Yes/No |
| Age Group Vi: | 5 to 10 XXX<br>years<br>11 to 17 XXX<br>years |
| Site/Subject<br>number | XXX/XXX |

[1] Study day is relative to the date of first administration of study drug (Day 0).

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Repeat for all visits recorded

Listing 16.2.13.2 Tanner Staging (Safety Analysis Set)

| Site/Subject<br>number | Age Group | Age/Sex/Race | Visit | Date (Study Day [1]) | Was assessment<br>performed? | Reason not<br>performed? | Tanner<br>Stage |
|---|---|---|---|---|---|---|---|
| XXX/XXX | 11 to 17 | XX/Female/White | XXX | DDMMMYYYY (XX) | X | | XXX |
| XXX/XXX | years<br>5 to 10 years | XX/Female/White | XXX | DDMMMYYYY (XX) | N | XXXXXXXXXX | |

B = baseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).
[1] Study day is relative to the date of first administration of study drug (Day 0).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS Unscheduled assessments should be included in the listing and flagged as such in the visit column. The listing may go over multiple pages to capture all data. NOTES:

Listing 16.2.14.1 Pulmonary Function Test (Safety Analysis Set)

Parameter: <Parameter (Unit)>

| Site/Subject<br>number | Age Group | Age/Sex/Race | Visit | Was assessment<br>Visit performed? | Reason not<br>performed? | Date of<br>assessment<br>(Study day<br>[1]) | Observed | Change<br>from<br>baseline |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 5 to 10<br>vears | XX/Female/White | XXX | Yes | | DDMONYYYY (XX) XX.X B | XX.X B | |
| | 1 | | XXX | Yes | | DDMONYYYY (XX) | x.xx | ××.× |
| | | | XXX | No | XXXXXXXXX | | | |

B = baseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).
[1] Study day is relative to the date of first administration of study drug (Day 0)

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS NOTES: Unscheduled assessments should be included in the listing and flagged as such in the visit column.

Listing 16.2.15.1 Pregnancy Test (Safety Analysis Set)

| Site/Subject<br>number | Age Group | Visit | Was a pregnancy<br>test performed? | If No, reason pregnancy<br>test not performed | <pre>If Yes, date of pregnancy test (Study day [1])</pre> | Result |
|---|---|---|---|---|---|---|
| XXX/XXX<br>XXX/XXX | 5 to 10 years<br>11 to 17 years<br>11 to 17 years | XXX<br>XXX<br>XXX | Yes/No<br>Yes/No<br>Yes/No | Subject is premenarchal<br>Subject is male | DDMONYYYY (XX) | Negative/Positive |

Pregnancy test data was collected at Screening.  $\[1]$  Study day is relative to the date of first administration of study drug (Day 0).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Listing 16.2.16.1 Visit Dates (Enrolled Set)

| 40010110101 | | | Baseline | Week 4 | Week 8 | Week 12 | Week 16 | Week 20 | Week 24 |
|---|---|---|---|---|---|---|---|---|---|
| number | Age Group | Screening 1) | (Study Day | (Study Day<br>28) | (Study Day<br>56) | (Study Day<br>84) | (Study Day<br>112) | (Stusy Day<br>140) | (Study Day<br>168) |
| XXX/XXX | 5 to 10<br>years | DDMONYYY | DDMONYYYY DDMONYYYY (1) | DDMONYYYY<br>(XX) | DDMONYYYY (XX) | DDMONYYYY<br>(XX) | DDMONYYYY<br>(XX) | DDMONYYYY<br>(XX) | DDMONYYYY (XX) |
| Study Day in | relation to B | aseline visi | t date (Study | Day 1) present | Study Day in relation to Baseline visit date (Study Day 1) presented in brackets | • | | | |
| PROGRAM NAME:L XXX 01.SAS | L XXX 01.SAS | DATE OF | DATE OF RUN:XXXXXXXX | | TIME OF RUN: XX:XX:XX | DATE OF EXTRACTION:XXXXXXXX | ION: XXXXXXXXX | | |


Listing 16.2.16.1 Visit Dates (Enrolled Set)

| Site/Subject<br>number | Week (Studian Studian Age Group 196) | 28<br>y Day | Week 32<br>(Study Day<br>224) | Week 36<br>(Study Day<br>252) | Week 40<br>(Study Day<br>280) | Week 44<br>(Study Day<br>308) | Week 48<br>(Study Day<br>336) | Week 52<br>(Study Day<br>364) | Week 56<br>(Study Day<br>392) |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 5 to 10<br>years | DDMONYYYY<br>(XX) | DDMONYYYY<br>(XX) | DDMONYYYY<br>(XX) | DDMONYYYY<br>(XX) | DDMONYYYY<br>(XX) | DDMONYYYY<br>(XX) | DDMONYYYY<br>(XX) | DDMONYYYY (XX) |
| Study Day in | relation to E | Study Day in relation to Baseline visit date (Study | | Day 1) presented in brackets. | in brackets. | | | | |
| PROGRAM NAME: L_XXX_01.SAS | XXX_01.SAS | | DATE OF RUN:XXXXXXXX | TIME OF RUN: | OF RUN: XX:XX:XX DAT | DATE OF EXTRACTION:XXXXXXXX | N:XXXXXXXX | | |

Listing 16.2.16.1 Visit Dates (Enrolled Set)

| Site/Subject<br>number | Age Group | Week 68<br>(Study Day 476) | Week 80<br>(Study Day 560) | Week 92<br>(Study Day 644) | Week 104<br>(Study Day 728) | Week 108<br>(Study Day 756) |
|---|---|---|---|---|---|---|
| XXX/XXX | 5 to 10 years | rs DDMONYYYY (XX) | DDMONYYY (XX) | DDMONYYYY (XX) | DDMONYYYY (XX) | DDMONYYYY (XX) |
| Study Day in re | elation to Base | Study Day in relation to Baseline visit date (Study Day 1) presented in brackets. | y 1) presented in brack | ets. | | |
| PROGRAM NAME:L_XXX_01.SAS | _XXX_01.SAS | DATE OF RUN:XXXXXXXX | TIME OF RUN: XX:XX:XX | C DATE OF EXTRACTION:XXXXXXXXX | N:XXXXXXXX | |


Listing 16.2.17.1 Xanthoma Examination (Safety Analysis Set)

| | F | | Was | | Date of assessment | Were there<br>pre-existing | Were there pre-existing tendon | | Pre-existing cutaneous | |
|---|---|---|---|---|---|---|---|---|---|---|
| number Grou | Group | Visit | Visit performed? | performed? | (Study day<br>[1]) | present? | ranchomas<br>present? | Anacomicai<br>location | present | Anacomicai<br>location |
| XXX/XXX | 5 to<br>10 | XXX | × | | DDMONYYYY<br>(XX) | Yes/No | Yes/No | XXXXXXXXX | Yes/No | XXXXXXXXX |
| xxx/xxx | years<br>11 to<br>17 | XXX | Z | ××××××××××××××××××××××××××××××××××××××× | DDMONYYYY<br>(XX) | Yes/No | Yes/No | Other:<br>XXXXXXXXX | Yes/No | Other:<br>XXXXXXXXX |
| | years | | | | | | | | | |

[1] Study day is relative to the date of first administration of study drug (Day 0).

DATE OF RUN:XXXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Repeat for all visits recorded

Listing 16.2.17.1 Xanthoma Examination (Safety Analysis Set)

| | | | Pre- | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | existing | If yes, | | | | | | | |
| | | | xanthomas | have | Have they | | | Were new | | Were new | |
| | | | changed | they | resolved? | Have they | Were new | tendon | | cutaneous | |
| Site/Subject | Age | | since last | | (Date of | increased | xanthomas | xanthomas | Anatomical | xanthomas | Anatomical |
| number Group | Group | Visit | | in size? | resolution) | in size? | present? | present? | location | present? | location |
| XXX/XXX | 5 to | XXX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | XXXXXXXXXX | Yes/No | XXXXXXXXXX |
| | 10 | | | | | | | | | | |
| | years | | | | | | | | | | |
| XXX/XXX | 11 to | XXX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Other: | Yes/No | Other: |
| | 17 | | | | (DDMONYYYY) | | | | XXXXXXXXXX | | XXXXXXXXXX |
| | years | | | | | | | | | | |

[1] Study day is relative to the date of first administration of study drug (Day 0).

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Repeat for all visits recorded

Listing 16.2.17.2 Carotid Intima-Media Thickness (CIMT) (Safety Analysis Set)

| Site/Subject Age<br>number Grou | Age<br>Group | Age/Sex/Race | Visit | Was CIMT<br>assessment<br>performed? | Reason not<br>performed? | Date of collection (Study day [1]) | Parameter | Unit | Parameter Unit Observed | Change<br>from<br>baseline | % Change<br>from<br>baseline |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 11 to<br>17 | XX/Female/White | XX | X | | DDMONYYYY (XX) | XXX | XXX | XX.X B | | |
| | years | | × | Z | XXXXXXXXX | DDMONYYYY (XX) | XXX | XXX | XX.X | X. XX | ×. ×. |

B = baseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).
[1] Study day is relative to the date of first administration of study drug (Day 0)

DATE OF RUN:XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

Unscheduled assessments should be included in the listing and flagged as such in the visit column. The listing may go over multiple pages to capture all data. Repeat for all visits. NOTES:

Listing 16.2.17.3 Flow-mediated Dilation (FMD) (Safety Analysis Set)

| Site/Subject Age<br>number Grou | Age<br>Group | Age/Sex/Race | Visit | Was FMD<br>assessment<br>performed? | Reason not<br>performed? | Date of collection (Study day [1]) | Parameter | Unit | Parameter Unit Observed | Change<br>from<br>baseline | % Change<br>from<br>baseline |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 5 to<br>10 | XX/Female/White | XXX | X | | DDMONYYYY (XX) | XXX | XXX | XX.X B | | |
| | years | | XXX | Z | XXXXXXXXXX | DDMONYYYY (XX) | XXX | XXX | ×.×× | × ×. | ×. ×. |

B = baseline value. Baseline is defined as the last non-missing value (including scheduled and unscheduled assessments) prior to the subject receiving study treatment in the Efficacy Phase (Visit 4).
[1] Study day is relative to the date of first administration of study drug (Day 0)

PROGRAM NAME: L\_XXX\_01.SAS

DATE OF RUN:XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXXX

Unscheduled assessments should be included in the listing and flagged as such in the visit column. The listing may go over multiple pages to capture all data. Repeat for all visits. NOTES:

Listing 16.2.17.4 Palatability (Safety Analysis Set)

| Site/Subject Age<br>number Group | Age<br>Group | Visit | Was<br>assessment<br>Visit performed? | Reason not<br>performed? | Date of assessment (Study day [1]) | Able to<br>swallow<br>capsule? | If no, food<br>media used? | First occasion used this food media | If yes, rate<br>palatability |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 11 to<br>17 | ××× | X | | DDMONYYYY (XX) | Yes/No | | | |
| XXX/XXX | years<br>5 to 10<br>years | XXX | Z | XXXXXXXXX | DDMONYYYY<br>(XX) | Yes/No | XXXXXXXXX | Yes/No | XXXXXXXXX |

[1] Study day is relative to the date of first administration of study drug (Day 0).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Repeat for all visits recorded


Listing 16.2.17.4 Palatability (Safety Analysis Set)

| Site/Subject Age<br>number Grou | Age<br>Group | Visit | Was<br>assessment<br>Visit performed? | Parent / guardian<br>interpretation of child's<br>reaction / facial<br>expression | Problems giving medication to child as refuses to take or throws up immediately after? | Problems giving dietary supplements to child as refuses to take or throws up immediately after? |
|---|---|---|---|---|---|---|
| XXX/XXX | 11 to<br>17 | ××× | X | XXXXXXXXX | Yes/No | Yes/No |
| xxx/xxx | years<br>5 to 10<br>Years | XXX | N | XXXXXXXXX | Yes/No | Yes/No |

[1] Study day is relative to the date of first administration of study drug (Day 0).

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: L\_XXX\_01.SAS

NOTES: Repeat for all visits recorded

Listing 16.2.19.1 Diet and Dietary Supplement Compliance (Safety Analysis Set)

| Site/Subject Age<br>number Grou | Age<br>Group | Visit | Were 2-day diet<br>records<br>Visit completed? | Were 2-day<br>diet records<br>checked? | Dietary<br>discussion took<br>place? | Subject compliant with low fat diet? | Dietary<br>supplements<br>dispensed? | Subject compliant with dietary supplement regimen? |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 11 to<br>17 | XXX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| xxx/xxx | years<br>5 to 10<br>years | XXX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| PROGRAM NAME:L_XXX_01.SAS | _XXX_01.S | 1.5 | DATE OF RUN:XXXXXXX | XXX | TIME OF RUN: XX:XX:XX DP | DATE OF EXTRACTION:XXXXXXXX | XXXXXXX | |

NOTES: Repeat for all study visits

Figure 14.1.5.1 Kaplan-Meier Plot of Time to Dose Reduction (Safety Analysis Set)

## Kaplan-Meier plot of time to dose reduction

Time to dose reduction is defined as the time (weeks) from the date of the start of the safety phase to the time of first dose reduction, if any. Subjects who do not enter the safety phase will be censored at time 0. If a patient discontinues study drug they will be conneed as an event at the time of study discontinuation. If a patient has not had a dose reduction and is still on study drug, they will be censored at their last visit assessment date.

 $\ensuremath{\mathrm{N}} = \ensuremath{\mathrm{the}}$  number of subjects in the analysis set. Source: Listing 16.2.5.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Treatment group N counts should be presented in the legend.


Figure 14.1.5.2 Kaplan-Meier Plot of Time to Dose Interruption (Safety Analysis Set)

# Kaplan-Meier plot of time to dose interruption

Time to dose interruption is defined as the time (weeks) from the date of the start of the safety phase to the time of first dose interruption, if any. Subjects who do not enter the safety phase will be censored at time 0. If a patient discontinues study drug they will be counted as an event at the time of study discontinuation. If a patient has not had a dose interruption and is still on study drug, they will be censored at their last visit assessment date.

N= the number of subjects in the analysis set. Source: Listing 16.2.5.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Treatment group N counts should be presented in the legend.


## SQN Clinical study no: OCH19003

Figure 14.2.1.1 Waterfall Plot of Percentage Change (%) from Baseline in Fasting Lipid Panel at Week 24 by age group (Full Analysis Set)

Parameter: <Parameter (Unit)>

y-axis: percentage change from baseline at Week 24.

x-axis: subject.

Use 3 colours for the blocks representing the respective age group for the subject and overall.

Source: Listing 16.2.8.1, Table 14.2.1.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES:

Please present LDL-C first and then same order as specified in SAP rather than alphabetically.

Update table source according to parameter Table 14.2.1.1 (LDL-C), Table 14.2.2.1 (Non-HDL-C), Table 14.2.3.1 (TC), Table 14.2.4.1

(VLDL-C), Table 14.2.5.1 (Apo B), Table 14.2.6.1 (TG), Table 14.2.7.1 (Lp(a) Include reference line at 0. Repeat for all parameters.

## SQN Clinical study no: OCH19003

Figure 14.2.1.2 Forest Plot of Sub-group analysis for primary end point (percentage change at week 24) (Full Analysis Set)

Analysis Study Visit

Point estimate and 95% confidence interval. Point estimate will be estimated as the mean percentage change and corresponding 95% CI y-axis: Overall estimate and Sub-group analysis references (i.e. SG1 to SG7). x-axis: Mean difference in percentage change at week 24. calculated from the ANCOVA model. Source: Listing 16.2.8.1, Table 14.2.1.4 (SG1), Table 14.2.1.5 (SG2), Table 14.2.1.6 (SG3), Table 14.2.1.7 (SG4), Table 14.2.1.8 (SG5), Table 14.2.1.10 (SG7) SG3: Established CVD history (defined as aortic valve disease and/or coronary atherosclerosis) vs no established CVD history (as defined SG4: Taken concomitant LLT medications vs not taken concomitant LLT medications (pooled across age groups). SG2: Documented CVD vs no documented CVD history at screening (pooled across age groups). SG5: No dose reductions vs at least one dose reduction (pooled across age groups). SG6: Reached MTD for age group vs did not reach MTD for age group. previously) at screening (pooled across age groups). SG7: Male vs Female (pooled across age groups). SG1: Age cohorts i.e. 2 age groups).

DATE OF EXTRACTION:XXXXXXXX

TIME OF RUN: XX:XX:XX

DATE OF RUN:XXXXXXXX

PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Repeat for Nominal Study Visit. Include reference line at 0.

Figure 14.2.1.3 Profile Plot of LSMeans percentage change from baseline over time in Fasting Lipid Panel

(Full Analysis Set)

Parameter: <Parameter (Unit)>

y-axis: dynamic based on the parameter <Parameter (Unit)>. Point estimate and corresponding error bar. LS mean percentage change at time point with corresponding standard error. The mean and median x-axis: time (weeks) relative to baseline.

Source: Listing 16.2.8.1, Table 14.2.9.1

dose at each timepoint will be added.

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F XXX 01.SAS

Please present Week 104 as EOT / Week 104 (as we do in the tables)

Update table source according to parameter Table 14.2.9.1 (LDL-C), Table 14.2.9.2 (Non-HDL-C), Table 14.2.9.3 (TC), Table 14.2.9.4 (VLDL-C), Table 14.2.9.8 (TC/HDL-C) and Table 14.2.12.2 (HDL-C), Table 14.2.9.5 (Apo B), Table 14.2.9.6 (TG), Table 14.2.9.7 (Lp(a)), Table 14.2.9.8 (TC/HDL-C) and Table 14.2.12.2 (HDL-C) C) Use analysis study visit data. Include reference line at 0. Repeat for all parameters. NOTES:

## SQN Clinical study no: OCH19003

Figure 14.2.1.4 Forest Plot of Sub-group analysis for key secondary endpoint: Non-HDL-C (percentage change at week 24) (Full Analysis Set)

Analysis Study Visit

Repeat of Figure 14.2.1.2 for NON-HDL-C

Source: Listing 16.2.8.1, Table 14.2.2.4 (SG1), Table 14.2.2.5 (SG2), Table 14.2.2.6 (SG3), Table 14.2.2.7 (SG4), Table 14.2.2.8 (SG5), Table 14.2.2.9 (SG6), Table 14.2.2.10 (SG7)

SG1: Age cohorts i.e. 2 age groups).

SG2: Documented CVD vs no documented CVD history at screening (pooled across age groups).
SG3: Established CVD history (defined as aortic valve disease and/or coronary atherosclerosis) vs no established CVD history (as defined previously) at screening (pooled across age groups).

SG4: Taken concomitant LLT medications vs not taken concomitant LLT medications (pooled across age groups). SG5: No dose reductions vs at least one dose reduction (pooled across age groups).

SG6: Reached MTD for age group vs did not reach MTD for age group

SG7: Male vs Female (pooled across age groups).

DATE OF RUN:XXXXXXXX

PROGRAM NAME: F XXX 01.SAS

DATE OF EXTRACTION: XXXXXXXXX

TIME OF RUN: XX:XX:XX

NOTES:

Repeat for Nominal Study Visit. Include reference line at 0.


## SQN Clinical study no: OCH19003

Figure 14.2.1.5 Forest Plot of Sub-group analysis for key secondary endpoint: TC (percentage change at week 24)

(Full Analysis Set)

Analysis Study Visit

Repeat of Figure 14.2.1.2 for TC

Source: Listing 16.2.8.1, Table 14.2.3.4 (SG1), Table 14.2.3.5 (SG2), Table 14.2.3.6 (SG3), Table 14.2.3.7 (SG4), Table 14.2.3.8 (SG5), Table

14.2.3.9 (SG6), Table 14.2.3.10 (SG7) SG1: Age cohorts i.e. 2 age groups).

SG2: Documented CVD vs no documented CVD history at screening (pooled across age groups).
SG3: Established CVD history (defined as aortic valve disease and/or coronary atherosclerosis) vs no established CVD history (as defined previously) at screening (pooled across age groups).

SG4: Taken concomitant LLT medications vs not taken concomitant LLT medications (pooled across age groups). SG5: No dose reductions vs at least one dose reduction (pooled across age groups).

SG6: Reached MTD for age group vs did not reach MTD for age group

SG7: Male vs Female (pooled across age groups).

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F XXX 01.SAS

Repeat for Nominal Study Visit. Include reference line at 0. NOTES:

## SQN Clinical study no: OCH19003

Figure 14.2.1.6 Forest Plot of Sub-group analysis for key secondary endpoint: VLDL-C (percentage change at week 24) (Full Analysis Set)

Analysis Study Visit

Repeat of Figure 14.2.1.2 for VLDL-C

Source: Listing 16.2.8.1, Table 14.2.4.4 (SG1), Table 14.2.4.5 (SG2), Table 14.2.4.6 (SG3), Table 14.2.4.7 (SG4), Table 14.2.4.8 (SG5), Table

14.2.4.9 (SG6), Table 14.2.4.10 (SG7)

SG1: Age cohorts i.e. 2 age groups).

SG2: Documented CVD vs no documented CVD history at screening (pooled across age groups). SG3: Established CVD history (defined as aortic valve disease and/or coronary atherosclerosis) vs no established CVD history (as defined

previously) at screening (pooled across age groups).

SG4: Taken concomitant LLT medications vs not taken concomitant LLT medications (pooled across age groups). SG5: No dose reductions vs at least one dose reduction (pooled across age groups).

 $SG6\colon$  Reached MTD for age group vs did not reach MTD for age group  $SG7\colon$  Male vs Female (pooled across age groups).

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F XXX 01.SAS

NOTES: Repeat for Nominal Study Visit.

: Repeat for Nominal Study Visit Include reference line at 0.


## SQN Clinical study no: OCH19003

Figure 14.2.1.7 Forest Plot of Sub-group analysis for key secondary endpoint: Apo B (percentage change at week 24) (Full Analysis Set)

Analysis Study Visit

Repeat of Figure 14.2.1.2 for Apo B

Source: Listing 16.2.8.1, Table 14.2.5.4 (SG1), Table 14.2.5.5 (SG2), Table 14.2.5.6 (SG3), Table 14.2.5.7 (SG4), Table 14.2.5.8 (SG5), Table 14.2.5.9 (SG6), Table 14.2.5.10 (SG7)

SG1: Age cohorts i.e. 2 age groups).

SG2: Documented CVD vs no documented CVD history at screening (pooled across age groups).
SG3: Established CVD history (defined as aortic valve disease and/or coronary atherosclerosis) vs no established CVD history (as defined

SG4: Taken concomitant LLT medications vs not taken concomitant LLT medications (pooled across age groups). SG5: No dose reductions vs at least one dose reduction (pooled across age groups). previously) at screening (pooled across age groups).

SG6: Reached MTD for age group vs did not reach MTD for age group SG7: Male vs Female (pooled across age groups).

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F XXX 01.SAS

NOTES:

Repeat for Nominal Study Visit. Include reference line at 0.

## SQN Clinical study no: OCH19003

Figure 14.2.1.8 Forest Plot of Sub-group analysis for key secondary endpoint: TG (percentage change at week 24)

(Full Analysis Set)

Analysis Study Visit

Repeat of Figure 14.2.1.2 for TG

Source: Listing 16.2.8.1, Table 14.2.6.4 (SG1), Table 14.2.6.5 (SG2), Table 14.2.6.6 (SG3), Table 14.2.6.7 (SG4), Table 14.2.6.8 (SG5), Table

14.2.6.9 (SG6), Table 14.2.6.10 (SG7) SG1: Age cohorts i.e. 2 age groups).

SG2: Documented CVD vs no documented CVD history at screening (pooled across age groups). SG3: Established CVD history (defined as aortic valve disease and/or coronary atherosclerosis) vs no established CVD history (as defined

previously) at screening (pooled across age groups).

SG4: Taken concomitant LLT medications vs not taken concomitant LLT medications (pooled across age groups). SG5: No dose reductions vs at least one dose reduction (pooled across age groups).

SG6: Reached MTD for age group vs did not reach MTD for age group SG7: Male vs Female (pooled across age groups).

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F XXX 01.SAS

NOTES:

Repeat for Nominal Study Visit. Include reference line at 0.


## SQN Clinical study no: OCH19003

Figure 14.2.1.9 Forest Plot of Sub-group analysis for key secondary endpoint: Lp(a) (percentage change at week 24)

(Full Analysis Set)

Analysis Study Visit

Repeat of Figure 14.2.1.2 for Lp(a)

Source: Listing 16.2.8.1, Table 14.2.7.4 (SG1), Table 14.2.7.5 (SG2), Table 14.2.7.6 (SG3), Table 14.2.7.7 (SG4), Table 14.2.7.8 (SG5), Table 14.2.7.9 (SG6), Table 14.2.7.10 (SG7)

SG1: Age cohorts i.e. 2 age groups).

SG2: Documented CVD vs no documented CVD history at screening (pooled across age groups). SG3: Established CVD history (defined as aortic valve disease and/or coronary atherosclerosis) vs no established CVD history (as defined

SG4: Taken concomitant LLT medications vs not taken concomitant LLT medications (pooled across age groups). previously) at screening (pooled across age groups).

SG5: No dose reductions vs at least one dose reduction (pooled across age groups). SG6: Reached MTD for age group vs did not reach MTD for age group

SG7: Male vs Female (pooled across age groups).

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXX PROGRAM NAME: F XXX 01.SAS

Repeat for Nominal Study Visit. NOTES:

Include reference line at 0.

## SQN Clinical study no: OCH19003

Figure 14.2.1.10 Profile Plot of percentage change from baseline over time in Fasting Lipid Panel

(Full Analysis Set)

Parameter: <Parameter (Unit)>

Percentage change at time point. The mean and median dose at each timepoint will be added.  $y\mbox{-}\mathrm{axis}\colon$  dynamic based on the parameter <Parameter (Unit)>. x-axis: time (weeks) relative to baseline.

Source: Listing 16.2.8.1, Table 14.2.8.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES:

Use analysis study visit data.

Include reference line at 0.

Please present Week 104 as EOT / Week 104 (as we do in the tables)

Update table source according to parameter Table 14.2.8.1 (LDL-C), Table 14.2.8.2 (Non-HDL-C), Table 14.2.8.3 (TC), Table 14.2.8.4 (VLDL-C), Table 14.2.8.5 (Apo B), Table 14.2.8.6 (TG), Table 14.2.8.7 (Lp(a)), Table 14.2.8.8 (TC/HDL-C) and Table 14.2.12.1 (HDL-Include reference line at 0. Repeat for all parameters.

Figure 14.3.2.1 Cumulative distribution function (CDF) plot of LDL-C at Week 24 (Full Analysis Set)

The cumulative distribution function for LDL-C at week 24 will be plotted with a reference line at 135 mg/dL. Use 3 different coloured lines to represent each of the 2 age groups and overall. x-axis: LDL-C (mg/dL) at Week 24. y-axis: cumulative percentage.

Source: Listing 16.2.8.1, Table 14.2.8.1

DATE OF EXTRACTION: XXXXXXXXX

TIME OF RUN: XX:XX:XX

DATE OF RUN:XXXXXXXX

PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Include reference line at 135. Use analysis study visit Week 24. Date: 28JUN2024 Version: Final 5.0


Figure 14.3.2.2 Cumulative distribution function (CDF) plot of LDL-C over time (Full Analysis Set)

The cumulative distribution function for LDL-C at Week X will be plotted with a reference line at 135 mg/dL. Use 3 different coloured lines to represent each of the 2 age groups and overall. x-axis: LDL-C (mg/dL) at Week X. Y-axis: cumulative percentage.

Source: Listing 16.2.8.1, Table 14.2.11.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for each analysis study visit within the efficacy and safety phase (except week 24). Replace Week X with corresponding analysis study visit for each run, NOTES:

 Date: 28JUN2024

Version: Final 5.0

## SQN Clinical study no: OCH19003

Figure 14.3.2.3 Cumulative distribution function (CDF) plot of percentage change in LDL-C at Week 24 (Full Analysis Set)

x-axis: percentage change in LDL-C (%) at Week 24. y-axis: cumulative percentage.

The cumulative distribution function for percentage change in LDL-C at week 24 will be plotted with a reference line at -15, -25 and -50%. Use 3 different coloured lines to represent each of the 2 age groups and overall.

Source: Listing 16.2.8.1, Table 14.2.8.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

Include reference line at -15, -25 and -50. Use analysis study visit Week 24. NOTES:

## SQN Clinical study no: OCH19003

Figure 14.3.2.4 Cumulative distribution function (CDF) plot of lowest percentage change in LDL-C from Week (Full Analysis Set)

x-axis: lowest percentage change in LDL-C (%) from Week 8. y-axis: cumulative percentage. The cumulative distribution function for percentage change in LDL-C from Week 8 will be plotted with a reference line at -15, -25 and -

Use 3 different coloured lines to represent each of the 2 age groups and overall.

Source: Listing 16.2.8.1, Table 14.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

Include reference line at -15, -25 and -50. NOTES:

#### SQN Clinical study no: OCH19003

Figure 14.3.1.1 Subject profile for distribution of Treatment-Emergent adverse events and dose at time of event

(Safety Analysis Set)

All subjects

For each subject bar, the colour of the bar would change over time, with each colour representing the dose of the drug the subject was on Any periods the subject was unable to take any dose should be clearly marked in a grey or white colour (for example). Overlayed on each subject bar will be a symbol to represent the TEAE PT (e.g. vomiting, abdominal pain, diarrhoea, etc). The symbol will be placed at the relevant timepoint the TEAE began and an arrow added to represent the duration of the TEAE. The colour of the arrow for each TEAE will correspond to the TEAE being related / unrelated to lomitapide. Each subject would have a horizontal bar. The length of the bar would represent the time on the study. Note: Time (weeks) should correspond with visits and days used for TEAE onset and recovery. The line style of the arrow for each TEAE will correspond to the TEAE severity. Each TEAE experienced by the subject will be represented in a similar manner. Y-axis = subject number. X-axis = Time (weeks).

Source: Listing 16.2.7.1, Table 14.3.1.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN: XXXXXXXX PROGRAM NAME: F XXX 01.SAS

Repeat for: Non-compliant with diet - All subjects; Non- compliant with diet - All subjects aged 5 to 10 years; Non-compliant with diet - All subjects aged 11 to 17 years. Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Repeat for: Compliant with diet - All subjects; Compliant with diet - All subjects aged 5 to 10 years; Compliant with diet - All subjects aged 11 to 17 years. NOTES:

#### SQN Clinical study no: OCH19003

Figure 14.3.1.2 Age profile for distribution of Treatment-Emergent adverse events and MTD

(Safety Analysis Set)

Overall - All subjects

Each subject would have a vertical bar.

The length of the bar would represent the time on study.

Under the x-axis, rather than the subject number being displayed the subject's age will be displayed on the graphic. The patients will be ordered by age starting with the youngest age closest to the y-axis and moving in an ascending order of age. For each patient bar, the colour of bar would represent the MTD the subject achieved, with each colour representing the MTD the subject achieved.

Y-axis = Time (weeks).

X-axis = Subject.

Note: Time (weeks) should correspond with visits.

Overlayed on each patient bar will be a symbol to represent the TEAE PT (e.g. vomiting, abdominal pain, diarrhoea, etc). The symbol will be placed at the relevant timepoint the TEAE began. Each TEAE experienced by the subject will be represented in a similar manner.

Source: Listing 16.2.7.1, Table 14.3.1.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXXX PROGRAM NAME: F XXX 01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Repeat for: Related TEAEs - All subjects; Related TEAEs - All subjects aged 5 to 10 years; Related TEAEs - All subjects aged 11 to NOTES:

17 years.

## SQN Clinical study no: OCH19003

Figure 14.3.1.3 Histogram of Time to First Gastrointestinal Treatment-Emergent Adverse Event (Safety Analysis Set)

Overall

Histogram showing the time (days) of onset from the first dose to the first gastrointestinal TEAE

Source: Listing 16.2.7.1, Table 14.3.1.13

DATE OF EXTRACTION: XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Repeat for: Subjects aged 5 to 10 years; Subjects aged 11 to 17 years.


## SQN Clinical study no: OCH19003

Figure 14.3.1.4 Histogram of Time to First Hepatic Treatment-Emergent Adverse Event (Safety Analysis Set)

Overall

Histogram showing the time of onset from the first dose to the first hepatic TEAE

Source: Listing 16.2.7.1, Table 14.3.1.14

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Repeat for: Subjects aged 5 to 10 years; Subjects aged 11 to 17 years.

## SQN Clinical study no: OCH19003

Figure 14.3.3.1 Individual subject profiles of liver function data (Safety Analysis Set)

Subject XXXX

Each line will be colour coordinated by the liver function test (e.g. AST, ALT, GGT, Alk Phos, Total bilirubin, serum albumin). A line joining all plotted values will be added to show the patient profile of the liver function test over time. A separate line will be generated for each liver function test profile over time. For each patient, at each time point the corresponding liver function tests value will be plotted. Heptic fat will also be added with a second y-axis with the hepatic fat scale. Patient's dose of drug included under the x-axis at each of the analysis study weeks. Each patient would have their own plot to show all liver function tests on one page. Y-axis = liver function scale. X-axis = Analysis Study Week. Y-axis2 = hepatic fat scale.

Source: Listing 16.2.8.3, Table 14.3.3.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F XXX 01.SAS

Time (week) on x-axis will use the analysis study week window for statistical analyses as defined in the SAP to determine study Screening will be defined at week -12. week for the time axis. NOTES:

Include unscheduled visits in figure (as approporiate).

#### SQN Clinical study no: OCH19003

Figure 14.3.3.2 AST profiles over time, by subject age (Safety Analysis Set)

Overall - All subjects

A line joining all plotted values will be added to show the patient profile of the liver function test over time. For each patient, at each time point the corresponding AST liver function tests value will be plotted. Each line will be colour coordinated by patient's age. Y-axis = AST liver function scale. X-axis = time (weeks).

Source: Listing 16.2.8.3, Table 14.3.3.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Screening will be defined at week -12. NOTES:

Time (week) on x-axis will use the study say window for statistical analyses as defined in the SAP to determine study week for the

Include unscheduled visits in figure (as approporiate).


#### SQN Clinical study no: OCH19003

Figure 14.3.3.3 ALT profiles over time, by subject age (Safety Analysis Set)

Subject XXXX

A line joining all plotted values will be added to show the patient profile of the liver function test over time. For each patient, at each time point the corresponding ALT liver function tests value will be plotted. Each line will be colour coordinated by patient's age. Y-axis = ALT liver function scale. X-axis = time (weeks).

Source: Listing 16.2.8.3, Table 14.3.3.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Screening will be defined at week -12. NOTES:

Time (week) on x-axis will use the study say window for statistical analyses as defined in the SAP to determine study week for the

Include unscheduled visits in figure (as approporiate).

#### SQN Clinical study no: OCH19003

Figure 14.3.3.4 AST profiles over time, by subject MTD (Safety Analysis Set)

Overall - All subjects

A line joining all plotted values will be added to show the patient profile of the liver function test over time. For each patient, at each time point the corresponding AST liver function tests value will be plotted. Each line will be colour coordinated by patient's MTD. Y-axis = AST liver function scale.

X-axis = time (weeks).

Source: Listing 16.2.8.3, Table 14.3.3.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Screening will be defined at week -12. NOTES:

Time (week) on x-axis will use the study say window for statistical analyses as defined in the SAP to determine study week for the

Include unscheduled visits in figure (as approporiate).

#### SQN Clinical study no: OCH19003

Figure 14.3.3.5 ALT profiles over time, by subject MTD (Safety Analysis Set)

Overall - All subjects

A line joining all plotted values will be added to show the patient profile of the liver function test over time. For each patient, at each time point the corresponding ALT liver function tests value will be plotted. Each line will be colour coordinated by patient's MTD. Y-axis = ALT liver function scale. X-axis = time (weeks).

Source: Listing 16.2.8.3, Table 14.3.3.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Screening will be defined at week -12. NOTES:

Time (week) on x-axis will use the study say window for statistical analyses as defined in the SAP to determine study week for the

Include unscheduled visits in figure (as approporiate).


#### SQN Clinical study no: OCH19003

Figure 14.3.3.6 Individual subject profiles of LDL-C data (Safety Analysis Set)

Subject XXXX

Markers will be added to each LDL-C profile line to denote the treatment dose the patient was on at that time point. Any periods the subject was unable to take any dose should also be clearly marked using a different marker. Dose adjustments will be identified with a different marker and lipoprotein apheresis with a vertical line. A line joining all plotted values will be added to show the patient profile of the LDL-C over time. For each patient, at each time point the corresponding LDL-C value will be plotted. Each patient would have their own plot to show their LDL-C profile. A horizontal line denoting an LDL-C of 110 mg/dL will be added. Y-axis = LDL-C scale. X-axis = time (weeks)

Source: Listing 16.2.8.1, Table 14.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F XXX 01.SAS

Time (week) on x-axis will use the study say window for statistical analyses as defined in the SAP to determine study week for the Repeat for: Overall – All subjects aged 5 to 10 years; Overall – All subjects aged 11 to 17 years. Screening will be defined at week -12. Add a reference line at  $y=110~{\rm mg/dL}$ . time axis. NOTES:

Include unscheduled visits in figure (as approporiate).


#### SQN Clinical study no: OCH19003

Figure 14.3.3.7 LDL-C profiles over time, by subject age (Safety Analysis Set)

Overall - All subjects

A line joining all plotted values will be added to show the patient profile of the LDL-C over time. Each line will be colour coordinated by patient's age. For each patient, at each time point the corresponding LDL-C value will be plotted. Y-axis = LDL-C scale. X-axis = time (weeks)

Source: Listing 16.2.8.1, Table 14.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F XXX 01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Screening will be defined at week -12. NOTES:

Time (week) on x-axis will use the analysis study week window for statistical analyses as defined in the SAP to determine study week for the time axis.

Patients who discontinue early and use EOT/Week 104, please use the calculated study day the EOT was completed to assign the subject to the relevant analysis study week window (e.g. patients 01-02 and 01-03). Include unscheduled visits in figure (as approporiate).

#### SQN Clinical study no: OCH19003

Figure 14.3.3.8 LDL-C profiles over time, by subject MTD (Safety Analysis Set)

Overall - All subjects

A line joining all plotted values will be added to show the patient profile of the LDL-C over time. Each line will be colour coordinated by patient's MTD. For each patient, at each time point the corresponding LDL-C value will be plotted. Y-axis = LDL-C scale. X-axis = time (weeks)

Source: Listing 16.2.8.1, Table 14.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Screening will be defined at week -12. NOTES:

Time (week) on x-axis will use the study say window for statistical analyses as defined in the SAP to determine study week for the

Include unscheduled visits in figure (as approporiate).

## SQN Clinical study no: OCH19003

Figure 14.3.3.9 Spaghetti plot of lipid profiles over time (Safety Analysis Set)

Parameter: <Parameter (Unit)>

Overall - All subjects

For each patient, at each time point the corresponding lipid value will be plotted. A separate line will be generated for each patient to show their individual parameter value over time. Y-axis = Lipid value. X-axis = time (weeks).

Source: Listing 16.2.8.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Inlcude assessments from Run-in up to Week  $104/{\rm EoT.}$ NOTES:

## SQN Clinical study no: OCH19003

Figure 14.3.3.10 eDISH plot of Maximum Post-Baseline ALT by Maximum Post-Baseline Total Bilirubin

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

Plot maximum post baseline ALT by maximum post baseline TBL for each patient. Use log scale for both sets of axes. y-axis: Maximum post-baseline TBL (x ULN) x-axis: Maximum post-baseline ALT (x ULN)

Label the 4 quadrants created by the reference lines: Top left = Hyperbilirubinemia; Top right = Hy's Law range; Bottom right = Temple's Include the following reference lines: x-axis (vertical line) = 3, y-axis (horizontal line) = 2. Include reference lines also where x = y = 1 (will create a 'box' in the lower left of the plot). Corollary range; Bottom left: Normal Range (inside 'box' created by x = y = 1 reference lines)

ALT = Alanine Aminotransaminase, TBL = Total Bilirubin, ULN = Upper Limit of Normal. Source: Listing 16.2.8.3

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX Different coulour/symbol for each age group DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS NOTES:

Include any abnormal observation (scheduled or unscheduled) Repeat for each study phase 

## SQN Clinical study no: OCH19003

Figure 14.3.3.11 eDISH plot of Maximum Post-Baseline AST by Maximum Post-Baseline Total Bilirubin

(Safety Analysis Set)

Overall / Efficacy Phase / Safety Phase / Follow-up

Repeat Figure 14.3.3.9 for AST

 ${\tt AST = Aspartate Aminotransferase, TBL = Total Bilirubin, ULN = Upper Limit of Normal. Source: Listing 16.2.8.3}$ 

DATE OF RUN:XXXXXXXX

PROGRAM NAME: F\_XXX\_01.SAS

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX

Different coulour/symbol for each age group Include any abnormal observation (scheduled or unscheduled) NOTES:

Repeat for each study phase

#### SQN Clinical study no: OCH19003

Figure 14.3.3.12 Subject profile for distribution of Liver Function Test Abnormalities and dose at time of event (Safety Analysis Set)

All subjects

Each subject experiencing an LFT abnormality will be identified with a bar starting at LFT elevation start and ending at the date when the Each subject would have a horizontal bar.

LFT abnormality ends.

Dose taken will be marked in the plot. Any periods the subject was unable to take any dose should be clearly marked.

Overlayed on each subject bar will be a symbol to represent the Hepatic TEAE PT (e.g. vomiting, abdominal pain, diarrhoea, etc).

The symbol will be placed at the relevant timepoint the TEAE began and an arrow added to represent the duration of the TEAE.

Each Hepatic TEAE experienced by the subject will be represented in a similar manner.

Y-axis = subject number. X-axis = Time (weeks). Source: Listing 16.2.5.1, Listing 16.2.7.1, Listing 16.2.8.3

DATE OF EXTRACTION:XXXXXXXX DATE OF RUN: XXXXXXXXX TIME OF RUN: XX:XX:XX PROGRAM NAME: F\_XXX\_01.SAS NOTES: Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years.

## SQN Clinical study no: OCH19003

Figure 14.3.5.1 Boxplot of Observed Vital Signs over Time (Safety Analysis Set)

|L|Parameter: <Parameter (Unit)>

x-axis: Time (weeks)

x-axis: IIme (weeks) y-axis: Observed value Boxplot of the observed value for the respective parameter over time. A boxplot will be displayed for each age group at each side of the tick mark, Use a different colour for each age group.

Source: Listing 16.2.9.1, Table 14.3.5.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Different coulour/symbol for each age group

# DocuSign Envelope ID: A18FEEF9-59CA-4D21-B668-F2E37C0A9EAE

## SQN Clinical study no: OCH19003

Figure 14.3.5.2 Boxplot of Change from Baseline Vital Signs over Time

(Safety Analysis Set)

Amryt Pharma study no: APH-19

|L|Parameter: <Parameter (Unit)>

Repeat Figure 14.3.5.1 for change from baseline

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION: XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Different coulour/symbol for each age group


#### SQN Clinical study no: OCH19003

Figure 14.3.5.3 Waterfall plot of change in BMI at Week 24, 56 and 104, by patient sex

(Safety Analysis Set)

Week 24 Overall - All subjects Each patient will be represented by a vertical bar, where the length of the bar represents the change in BMI (baseline to the respective Order the vertical bars in decreasing order of size of change in BMI. For each patient bar, the colour of the bar will represent the sex of the patient. Y-axis = change in BMI. week, as applicable).

Source: Listing 16.2.9.1, Table 14.3.5.1

X-axis = subject.

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years.

#### SQN Clinical study no: OCH19003

Figure 14.3.8.1 Scatter plot of change in hepatic fat up with change in BMI Z score up to week 56 and 104, by subject age

(Safety Analysis Set)

Overall - All subjects Week 56

Each patient will be represented with a mark on the graphic displaying their change in BMI Z score and corresponding change in hepatic

Each symbol will be colour coded to represent the patient's age in years. Y-axis = change in hepatic fat. X-axis = change in BMI Z score.

Only NMR scan assessments are included. Source: Listing 16.2.12.1, Table 14.3.8.1.1, Table 14.1.2.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Repeat for Week 104 NOTES:

#### SQN Clinical study no: OCH19003

Figure 14.3.8.2 Scatter plot of change in hepatic fat with change in BMI Z score up to week 56 and 104, by subject MTD

(Safety Analysis Set)

Week 56 Overall - All subjects Each patient will be represented with a mark on the graphic displaying their change in BMI Z score and corresponding change in hepatic

Each symbol will be colour coded to represent the patient's MTD they achieved. Y-axis = change in hepatic fat.

Y-axis = change in hepatic fat. X-axis = change in BMI Z score.

Only NMR scan assessments are included. Source: Listing 16.2.12.1, Table 14.3.8.1.1, Table 14.1.2.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Repeat for week 104 NOTES:


#### SQN Clinical study no: OCH19003

Figure 14.3.8.3 Scatter plot of change in hepatic fat up to week 56 and 104 and time fom Lomitapide administration, by subject age

(Safety Analysis Set)

Week 56

Overall - All subjects

Each patient will be represented with a mark on the graphic displaying their time from lomitapide administration and corresponding change in hepatic fat up to week 56.

Each symbol will be colour coded to represent the patient's age in years.

Y-axis = change in hepatic fat. X-axis = time from lomitapide administration.

Only NMR scan assessments are included. Source: Listing 16.2.12.1, Table 14.3.8.1.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Repeat for week 104 NOTES:

#### SQN Clinical study no: OCH19003

Figure 14.3.8.4 Scatter plot of change in hepatic fat up to week 56 and 104 and time from Lomitapide administration, by subject MTD

(Safety Analysis Set)

Week 56 Overall - All subjects

Each patient will be represented with a mark on the graphic displaying their time from lomitapide administration and corresponding change in hepatic fat up to week 56.

Each symbol will be colour coded to represent the patient's MTD they achieved.

Y-axis = change in hepatic fat.

X-axis = time from lomitapide administration.

Only NMR scan assessments are included. Source: Listing 16.2.12.1, Table 14.3.8.1.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Repeat for Week 104 NOTES:


## SQN Clinical study no: OCH19003

Figure 14.3.8.5 Cumulative distribution function (CDF) plot of percentage change in hepatic fat over time

(Safety Analysis Set)

Analysis Study Week XX

 $x\hbox{-}axis.$  Percentage change from baseline in hepatic fat. y-axis: cumulative percentage.

The cumulative distribution function for percentage change in hepatic fat will be plotted with a reference line at 5, 10, 15 and 20%. Use 3 different coloured lines to represent each of the 2 age groups and overall.

Only NMR scan assessments are included. Source: Listing 16.2.12.1, Table 14.3.8.3.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

Include reference line at 5, 10, 15 and 20%. Repeat for each analysis study week. NOTES:


#### SQN Clinical study no: OCH19003

Figure 14.3.8.6 Scatter plot of ALT vs hepatic fat over time (Safety Analysis Set)

Imaging technology: NMR
All subjects

y-axis: Observed ALT (in x ULN) Scatter plot of ALT vs hepatic fat will be plotted at baseline, Week 24, Week 56 and Week 104/EOT. Use different colour to represent each age group. Use different symbols for each time point. Add Pearson's correlation coefficient (NMR) or Spearman's Rank correlation coefficient (Ultrasound) x-axis: Hepatic fat

Source: Listing 16.2.8.3, Listing 16.2.12.1, Table 14.3.8.3.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

Repeat for each age group and for ultrasound scan Present ALT as x times ULN. NOTES:

# DocuSign Envelope ID: A18FEEF9-59CA-4D21-B668-F2E37C0A9EAE

## SQN Clinical study no: OCH19003

Figure 14.3.8.7 Scatter plot of AST vs hepatic fat over time

Amryt Pharma study no: APH-19

(Safety Analysis Set)

Imaging technology: NMR
All subjects

Repeat of Figure 14.3.8.6

Source: Listing 16.2.8.3, Listing 16.2.12.1, Table 14.3.8.3.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Repeat for each age group and for ultrasound scan Present AST as x times ULN.


#### SQN Clinical study no: OCH19003

Figure 14.3.9.1 Waterfall plot of change in BMI Z score at Week 24, 56 and 104, by patient age

(Safety Analysis Set)

Week XX

Overall - All subjects

Each patient will be represented by a vertical bar, where the length of the bar represents the change in BMI Z score (baseline to week 24, 56 or 104).

Order the vertical bars in decreasing order of size of change in BMI  ${\tt Z}$  score. For each patient bar, the colour of the bar will represent the age (years) of the patient.

Y-axis = change in BMI Z score.

X-axis = subject.

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Present for Weeks 24, 56 and 104. NOTES:


#### SQN Clinical study no: OCH19003

Figure 14.3.9.2 Waterfall plot of change in BMI Z score at Week 24, 56 and 104, by patient sex

(Safety Analysis Set)

Week XX

Overall - All subjects

Each patient will be represented by a vertical bar, where the length of the bar represents the change in BMI Z score (baseline to week 24, 56 or 104).

Order the vertical bars in decreasing order of size of change in BMI  ${\tt Z}$  score. For each patient bar, the colour of the bar will represent the age (years) of the patient.

Y-axis = change in BMI Z score.

X-axis = subject.

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Present for Week 24, 56 and 104. NOTES:

#### SQN Clinical study no: OCH19003

Figure 14.3.9.3 Spaghetti plot of BMI Z score over time, by patient age and sex (Safety Analysis Set)

Overall - All subjects

For each patient, at each time point the corresponding BMI Z score will be plotted. A separate line will be generated for each patient to show their individual BMI Z score profile over time. The symbol used for the patient to generate their profile spaghetti line will represent the patient's sex. Y-axis = BMI Z score value. Each line will be colour co-ordinated by the patient's age. X-axis = time (weeks).

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS NOTES: Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years.

Date: 28JUN2024


#### SQN Clinical study no: OCH19003

Figure 14.3.9.4 Spaghetti plot of BMI absolute value over time, by patient age and sex (Safety Analysis Set)

Overall - All subjects

For each patient, at each time point the corresponding BMI absolute value will be plotted. A separate line will be generated for each patient to show their individual BMI absolute value profile over time. The symbol used for the patient to generate their profile spaghetti line will represent the patient's sex. Y-axis = BMI absolute value. Each line will be colour co-ordinated by the patient's age. X-axis = time (weeks).

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS NOTES: Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years.


#### SQN Clinical study no: OCH19003

Figure 14.3.9.5 Spaghetti plot of weight absolute value over time, by patient age and sex (Safety Analysis Set)

Overall - All subjects

For each patient, at each time point the corresponding weight absolute value will be plotted. A separate line will be generated for each patient to show their individual weight absolute value profile over time. The symbol used for the patient to generate their profile spaghetti line will represent the patient's sex. Y-axis = weight absolute value. X-axis = time (weeks). Each line will be colour co-ordinated by the patient's age.

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS NOTES: Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years.

## SQN Clinical study no: OCH19003

Figure 14.3.9.6 Spaghetti plot of sexual maturation development over time (Full Analysis Set)

Age Group = 5 to 10 years; Sex = Male/Female

x-axis: time (weeks) relative to baseline. y-axis: tanner staging category (1 to 5). Separate line for each subject plotting tanner stage category over time. Generate 4 different plots for each age group and sex.

Source: Listing 16.2.13.2, Table 14.3.9.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS


## SQN Clinical study no: OCH19003

Figure 14.3.9.7 Spaghetti plot of growth development over time (Full Analysis Set)

Age Group = 5 to 10 years; Sex = Male/Female

x-axis: time (weeks) relative to baseline. y-axis: BMI percentile (scale 1 to 100). Separate line for each subject plotting BMI percentile over time. Generate 4 different plots for each age group and sex.

Source: Listing 16.2.9.1, Table 14.3.5.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS 

#### SQN Clinical study no: OCH19003

Figure 14.3.9.8 Waterfall plot of change in BMI Z-score at Week 24, 56 and 104, by baseline BMI for Age Z-score

(Safety Analysis Set)

Overall - All subjects

Each patient will be represented by a vertical bar, where the length of the bar represents the change in BMI Z score (baseline to week 24, 56 or 104).

Order the vertical bars in decreasing order of size of change in BMI Z-score. For each patient bar, the colour of the bar will represent the baseline BMI for Age Z-score of the patient.

Y-axis = change in BMI Z-score.

X-axis = subject.

BMI for Age Z-score cut-points are lower than -2.0 (wasted), between -2.0 and 1.0 (normal), between 1.0 and 2.0 (risk of overweight), between 2.0 and 3.0 (overweight) and more than 3.0 (obese).

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Group baseline BMI for Age Z score in the following categories: <-2.0 (wasted); >= -2.0 and <= 1.0 (normal); > 1.0 and <= 2.0 (risk of overweight); > 2.0 and <= 3.0 (overweight); > 3.0 (obese). Present for weeks 24, 56 and 104. NOTES:


#### SQN Clinical study no: OCH19003

Figure 14.3.9.9 Spaghetti plot of BMI Z-score over time, by baseline BMI for Age Z-score

(Safety Analysis Set)

Overall - All subjects

Each line will be colour co-ordinated by the patient's baseline BMI for Age Z-score (<-2, -2 <= x <= 1, 1 < x <= 2, 2 < x <= 3 and > 3). A separate line will be generated for each patient to show their individual BMI Z-score profile over time. The symbol used for the patient to generate their profile spaghetti line will represent the patient's sex. For each patient, at each time point the corresponding BMI Z-score will be plotted. Y-axis = BMI Z-score value. X-axis = time (weeks). BMI for Age Z-score cut-points are lower than -2.0 (wasted), between -2.0 and 1.0 (normal), between 1.0 and 2.0 (risk of overweight), between 2.0 and 3.0 (overweight) and more than 3.0 (obese). Source: Listing 16.2.9.1, Table 14.3.5.1

TIME OF RUN: XX:XX:XX DATE OF EXTRACTION:XXXXXXXX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. Group baseline BMI for Age Z-score in the following categories: <-2.0 (wasted); >= -2.0 and <= 1.0 (normal); > 1.0 and <= 2.0 (risk of overweight); > 2.0 and <= 3.0 (overweight); > 3.0 (obese). NOTES:


## SQN Clinical study no: OCH19003

Figure 14.3.9.10 Individual spaghetti plot of weight and Z scores over time (Safety Analysis Set)

Subject XXX

For each patient, at each time point the corresponding Weight and Z scores will be plotted. There will be one Y axis for Z-scores and a second Y-axis for absolute weight. A separate line will be generated for each parameter over time.

Y-axis = Height, Weight and BMI Z scores values. Y2-axis = absolute weight. X-axis = time (weeks).

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS 

#### SQN Clinical study no: OCH19003

Figure 14.3.9.11 Waterfall plot of change from baseline to maximum weight loss (Safety Analysis Set)

Overall - All subjects

Each patient will be represented by a vertical bar, where the length of the bar represents the change form basleline to the minimum post-baseline weight (baseline to the respective week, as applicable).

Order the vertical bars in decreasing order of size of change in weight. For each patient bar, the colour of the bar will represent the sex of the patient.

Y-axis = change in BMI.

X-axis = subject.

Source: Listing 16.2.9.1, Table 14.3.5.1

DATE OF EXTRACTION: XXXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS

NOTES: Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years.


#### SQN Clinical study no: OCH19003

Figure 14.3.9.12 Waterfall plot of change from baseline to minimum BMI z-score change

(Safety Analysis Set)

Overall - All subjects

Each patient will be represented by a vertical bar, where the length of the bar represents the change form baseline to the minimum BMI z-For each patient bar, the colour of the bar will represent the sex of the patient. Y-axis = Change from baseline to minimum  $BMI\ Z$ -score. Order the vertical bars in decreasing order of size of change in z-score. score change (baseline to the respective week, as applicable).

Source: Listing 16.2.9.1, Table 14.3.5.1

X-axis = subject.

DATE OF EXTRACTION:XXXXXXXX TIME OF RUN: XX:XX:XX DATE OF RUN:XXXXXXXX PROGRAM NAME: F\_XXX\_01.SAS Repeat for: Overall - All subjects aged 5 to 10 years; Overall - All subjects aged 11 to 17 years. NOTES:

